CLINICAL TRIAL: NCT01336621
Title: A Multicentre, Open-Label, Long-Term, Safety and Tolerability Study of Retigabine Immediate Release (IR) in Adults With Partial-Onset Seizures (Extension of Study RGB113905)
Brief Title: Long-Term Safety Study of Retigabine Immediate Release (IR) as Adjunctive Therapy in the Treatment of Adults With Partial-Onset Seizures (POS)
Acronym: IR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 113413; 2010-022777-34 (EudraCT Number)
Record Dates: First submitted 2011-03-10; First posted 2011-04-18 (Estimated); Results first posted 2018-02-26 (Actual); Last update posted 2020-03-11 (Actual); Status verified 2020-03

CONDITIONS: Epilepsy
Keywords: Partial-onset seizures; retigabine IR; Open Label Extension; GW582892; Epilepsy
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Retigabine IR (Experimental): Open label flexible dose between 300 mg/day (Minimum) and 1200 mg/day (maximum).
  Interventions: Drug: Retigabine IR

INTERVENTIONS:
Drug: Retigabine IR — Flexible dose between 300 mg/day (minimum) and 1200 mg/day (maximum)

SUMMARY:
The purpose of this Phase III study is to assess the long-term safety, tolerability and efficacy of flexibly dosed retigabine Immediate Release (IR) as adjunctive therapy in adult subjects with partial-onset seizures. In addition, those subjects who successfully completed 20 weeks of adjunctive treatment with retigabine IR in the parent study, RGB113905, and who were thought to have benefitted from treatment will be provided continued access to retigabine IR.

DETAILED DESCRIPTION:
RTG113413 is an open-label, multicentre extension study of RGB113905. This study will enroll adult subjects with partial-onset seizures (POS) who successfully completed 20 weeks of adjunctive treatment with retigabine IR (4-weeks Titration Phase and 16-weeks Flexible Dose Evaluation Phase) in the parent study, RGB113905 and who were thought to have benefitted from the treatment.

The Screening Visit (Visit 1) will be performed on the same day as the final visit of the parent study (Visit 7/Week 20). Subjects entering the extension study will initially receive the same dose of retigabine IR and concurrent antiepileptic drug (AED) as they were receiving on the final visit of the parent study. After the first week of the extension study, the subject's retigabine dose can be adjusted based on efficacy and tolerability. The overall daily dose of retigabine IR must be maintained between 300 mg/day (minimum) and 1200 mg/day (maximum). In addition, the dose and the number of concurrent AEDs can be adjusted to meet the individual needs of the subject. Retigabine IR monotherapy is not permitted. If concurrent AED therapy is removed, the subject must be withdrawn from the study.

Subjects in this study will be eligible to receive retigabine IR treatment until one of the following criteria have been met: 1) regulatory approval and commercial availability of retigabine IR or 2) retigabine IR is not approved by the regulatory authorities or 3) the study is terminated by the sponsor for reasons including, but not limited to, safety issues or 4) subject is withdrawn or withdraws consent or 5) subject has received retigabine IR treatment for a total of 3 years and options i-iv have not been met. After the Screening Visit, subjects will be required to attend 4 further clinic visits at Weeks 13, 26, 39, and 52 in the first year of the study and a total of 3 clinic visits at approximately 4-monthly intervals during each of the second and third year of study. Upon completion or early withdrawal, subjects will begin a 3-week taper period and then return for a follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* The subject has successfully completed the 20-weeks (4-weeks Titration and 16-weeks of Flexible Dose Evaluation Phases) of treatment with retigabine IR as adjunctive therapy to one of the pre-specified AEDs in the parent study RGB113905.
* The investigator and the subject, or caregiver, if applicable, should consider it beneficial for the subject to receive continued retigabine IR therapy.
* The subject is able and willing to maintain an accurate and complete daily written Seizure Calendar or has a caregiver who is able and willing to maintain an accurate and complete daily written Seizure Calendar for the entire duration of the study.
* The subject has given written informed consent, or has a legally authorized representative who has given written informed consent, prior to the performance of any study assessments.
* A female subject is eligible to enter and participate in the study if she is of non-childbearing potential (i.e., physiologically incapable of becoming pregnant, including any female who is pre- menarcheal or post menopausal).
* A female subject is eligible to enter and participate in the study if she is child-bearing potential and has a negative pregnancy test at Screening, and agrees to use one of the contraceptive methods listed in Appendix 3 of the protocol.
* A female subject is eligible to enter and participate in the study if she not pregnant or lactating or planning to become pregnant during the study.
* French subjects only: In France, a subject will be eligible for inclusion in this study only if either affiliated to or a beneficiary of a social security category.

Exclusion Criteria:

* Has met any of the withdrawal criteria in the previous RGB113905 study or has clinically significant abnormal clinical laboratory or ECG findings not resolved prior to entry to the open-label extension study.
* Is suffering from acute or progressive neurological disease, severe psychiatric disease, or severe mental abnormalities that are likely to interfere with the study objectives.
* Has any medical condition that, in the investigator's judgment, is considered to be clinically significant and could potentially affect subject safety or study outcome, including but not limited to: clinically significant cardiac, renal, hepatic condition, or a condition that affects the absorption, distribution, metabolism or excretion of drugs.
* Has any abnormality on 12-lead ECG at Screening which is clinically significant in the opinion of the investigator, or has QTc (either QTcB Bazett's correction or QTcF Fridericia's correction) >500 msec or >530 msec for subjects with Bundle Branch Block or an increase in QTc of >60 msec from Baseline in the parent study.
* Is unwilling or inability to follow the study procedures or reporting of AEs.
* Is planning on following a ketogenic diet or planning surgery or implantation of a Vagus Nerve Stimulator (VNS) to control seizures during the study. Note: Subjects who already have a VNS implanted which is functional may be permitted to enter the study.
* Has active suicidal plan/intent or has had active suicidal thoughts in the past 6 months. Has history of suicide attempt in the last 2 years or more than 1 lifetime suicide attempt.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2011-02-21 (Actual); Primary Completion 2016-12-14 (Actual); Study Completion 2017-09-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (28):
- GSK Investigational Site, Ghent, Belgium
- Bulgaria (2):
  - GSK Investigational Site, Plovdiv
  - GSK Investigational Site, Sofia
- France (2):
  - GSK Investigational Site, Limoges
  - GSK Investigational Site, Strasbourg
- GSK Investigational Site, Bielefeld, North Rhine-Westphalia, Germany
- Italy (6):
  - GSK Investigational Site, Foggia, Apulia
  - GSK Investigational Site, Bologna, Emilia-Romagna
  - GSK Investigational Site, Rome, Lazio
  - GSK Investigational Site, Genoa, Liguria
  - GSK Investigational Site, Torrette Di Ancona, The Marches
  - GSK Investigational Site, Pisa, Tuscany
- GSK Investigational Site, Heemstede, Netherlands
- GSK Investigational Site, Warsaw, Poland
- Russia (7):
  - GSK Investigational Site, Belgorod
  - GSK Investigational Site, Kazan'
  - GSK Investigational Site, Krasnodar
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Saint Petersburg
  - GSK Investigational Site, Samara
  - GSK Investigational Site, Smolensk
- Thailand (2):
  - GSK Investigational Site, Bangkok
  - GSK Investigational Site, Khon Kaen
- Ukraine (5):
  - GSK Investigational Site, Dnipro
  - GSK Investigational Site, Luhansk
  - GSK Investigational Site, Odesa
  - GSK Investigational Site, Oleksandrivka Village, Odesa
  - GSK Investigational Site, Poltava

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com/Posting.aspx?ID=20279

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with partial-onset seizures (POS) who successfully completed the 20 weeks of treatment in parent study NCT01336621 were recruited in this open-label extension (OLE) study. The study was conducted in two periods, a primary treatment phase and a safety follow-up continuation phase (SFUCP).
Pre-assignment Details: Screening was performed on the same day as the final visit of the parent study NCT01336621. A total of 98 participants completed the parent study and opted to enter into this study. All participants received at least one dose of retigabine immediate release (IR) tablets.
Groups:
- Retigabine IR: Eligible participants continued on the same maintenance dose of retigabine IR and the concurrent anti-epileptic drugs (AEDs) as they were taking at Visit 7 (Week 20) in the parent study NCT01336621. After the first week of the study, the dose of retigabine IR could be increased or decreased by 50-150 milligrams per day (mg/day) on a weekly basis. The overall daily dose of retigabine IR was to be maintained between 300 mg/day (minimum) and 1200 mg/day (maximum).
Period: Primary Reporting Phase (Upto 5.8 Years)
Arm/Group | Retigabine IR
Started | 98
Completed | 0
Not Completed | 98
Not completed — Adverse Event | 11
Not completed — Lack of Efficacy | 2
Not completed — Protocol Violation | 12
Not completed — Withdrawal by Subject | 27
Not completed — Other: study terminated | 11
Not completed — Physician Decision | 2
Not completed — Other: Reached stopping criteria | 22
Not completed — Other: lost to follow up | 2
Not completed — Other: Continued in SFUCP | 9
Period: SFUCP (up to 2.6 Years)
Arm/Group | Retigabine IR
Started | 9
Completed | 0
Not Completed | 9
Not completed — Other: Reached stopping criteria | 1
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 3
Not completed — Physician Decision | 1
Not completed — Other: Study closed/terminated | 3

BASELINE CHARACTERISTICS:
Arm/Group | Retigabine IR
Number analyzed (Participants) | 98
Age, Continuous [Mean (Standard Deviation); unit: Years] | 39.2 (13.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48
  Male | 50
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race customized: Asian: South East Asian Heritage | 8
  Race customized: White- White/Caucasian/ European Heritage | 90

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Serious AEs (TESAEs): Safety Population
Description: An AE is any untoward medical occurrence in a clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. SAE is defined as any untoward medical occurrence that, at any dose results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability, is a congenital anomaly/ birth defect or is associated with liver injury or impaired liver function. TEAE refers to an AE for which the onset was on or after the date of the first retigabine dose in this study and on or before 30 days after the last retigabine dose date. AEs that started in the parent study that increased in severity during this study were also considered treatment-emergent. The analysis was performed on Safety Population, which included participants who took at least one dose of study medication after they had enrolled into this OLE study.
Time Frame: Up to 5.8 years
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | Retigabine IR
Number analyzed (Participants) | 98
Participants
  Any TEAE | 38
  Any TESAE | 4

2. Primary Outcome: Number of Participants With AEs and SAEs: All SFUCP Subjects
Description: An AE is any untoward medical occurrence in a clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. SAE is defined as any untoward medical occurrence that, at any dose results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability, is a congenital anomaly/ birth defect or is associated with liver injury or impaired liver function. The following AEs were collected in the SFUCP: AEs related to the finding(s) of pigmentation/, discoloration of the eye/skin, AEs related to unexplained vision loss, SAEs, Deaths and Pregnancies. SFUCP collected AEs are those for which onset was 31 days or more after the last dose of retigabine. The analysis was performed on the All SFUCP Subjects population which comprised of all subjects who enter the SFUCP.
Time Frame: Up to 2.6 years
Population: All SFUCP subjects
Measure: Number; unit: Participants
Groups:
- Retigabine IR in SFUCP: Participants who withdrew from the Open-Label Treatment Phase and who had retinal pigmentation or unexplained vision loss, pigmentation of non-retinal ocular tissue or abnormal discoloration of nails, lips, skin or mucosa were followed-up in SFUCP after discontinuation of RTG. This is the final reporting phase of the study. During SFUCP, participants underwent six monthly comprehensive eye examinations and/or dermatological assessments. Participants were followed-up until the discoloration /pigmentation either resolves or stabilizes, as defined by no change over two consecutive six monthly assessments over at least 12 months after discontinuation of RTG IR .
Arm/Group | Retigabine IR in SFUCP
Number analyzed (Participants) | 9
Participants
  Any AE | 3
  Any SAE | 1

3. Primary Outcome: Number of Participants Withdrawn Due to TEAEs
Description: An AE is any untoward medical occurrence in a clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. SAE is any untoward medical occurrence that, at any dose results in death, is life-threatening, requires hospitalization or prolonged existing hospitalization, results in disability, is a congenital anomaly/birth defect or is associated with liver injury or impaired liver function. TEAE refers to an AE for which the onset was on or after the date of the first retigabine dose and on or before 30 days after the last retigabine dose date.
Time Frame: Up to 5.8 years
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | Retigabine IR
Number analyzed (Participants) | 98
Participants | 16

4. Primary Outcome: Number of Participants With Retinal Pigmentary Abnormalities
Description: Number of participants with abnormal findings after eye examination were evaluated. Only retinal pigmentary abnormalities detected on-treatment with retigabine were presented. Retinal pigmentary abnormalities included abnormalities in the macula, peripheral retina and unspecified location.
Time Frame: Up to 5.8 years
Population: Safety Population. Only those participants with >=1 ophthalmology exam on or before last dose of RTG are presented.
Measure: Number; unit: Participants
Arm/Group | Retigabine IR
Number analyzed (Participants) | 53
Participants | 8

5. Primary Outcome: Number of Participants With Pigmentation of Non-retinal Ocular Tissue(s)
Description: Number of participants with abnormal findings after eye examination were evaluated. Pigmentation of non-retinal ocular tissue (s) detected on-treatment with retigabine were presented. Non-retinal pigmentary abnormalities included abnormalities in the sclera and/ or conjunctiva, cornea, iris and lens.
Time Frame: Up to 5.8 years
Population: Safety Population. Only those participants with >=1 ophthalmology exam on or before last dose of RTG are presented.
Measure: Number; unit: Participants
Arm/Group | Retigabine IR
Number analyzed (Participants) | 53
Participants | 15

6. Primary Outcome: Number of Participants With Abnormal Discoloration of Skin
Description: Number of participants with Dermatologist-Confirmed abnormal discoloration of skin including skin around the eyes and eyelids, lips, nails, or mucosa were evaluated. Only abnormalities occurring on-treatment with retigabine were presented.
Time Frame: Up to 5.8 years
Population: Safety Population. Only those participants who had at least one skin exam by the investigator or dermatologist on or before the last dose of RTG or dermatologist-confirmed discoloration with start date on or before the date of last dose of RTG are presented.
Measure: Number; unit: Participants
Arm/Group | Retigabine IR
Number analyzed (Participants) | 58
Participants
  Any abnormal discoloration | 11
  Discoloration of skin | 5
  Discoloration of lips | 3
  Discoloration of nails | 10
  Discoloration of mucosa | 9

7. Primary Outcome: Number of Participants With a Clinically Significant Decrease in Visual Acuity From Initial Examination
Description: Number of participants with a clinically significant decrease in visual acuity from initial examination were evaluated. Only abnormalities occurring on-treatment with retigabine were presented.
Time Frame: Up to 5.8 years
Population: Safety Population. Only those participants with both initial and at least 1 follow-up exam while on RTG treatment are presented.
Measure: Number; unit: Participants
Arm/Group | Retigabine IR
Number analyzed (Participants) | 48
Participants | 3

8. Primary Outcome: Number of Participants With Decrease in Confrontational Visual Field From Initial Examination
Description: Number of participants with a clinically significant decrease in confrontational visual field from initial examination were evaluated. Only abnormalities occurring on-treatment with retigabine were presented.
Time Frame: Up to 5.8 years
Population: Safety Population. Only those subjects with both initial and at least 1 follow-up exam while on RTG treatment are presented.
Measure: Number; unit: Participants
Arm/Group | Retigabine IR
Number analyzed (Participants) | 48
Participants | 1

9. Primary Outcome: Number of Participants With Potential Clinical Concern (PCC) Values of Change From Baseline in Vital Signs and Weight
Description: Vital signs including systolic blood pressure (SBP), diastolic blood pressure (DBP) and heart rate (HR) were measured after at least 5 minutes of rest. Body weight was measured without shoes and wearing light clothing. Baseline assessments in this OLE study were defined by and taken directly from the Baseline assessments in the parent study NCT01336621. Change from Baseline was calculated by subtracting the Baseline value from the post-baseline value. Increase or decrease of >=20 in SBP, increase or decrease of >=15 in DBP and HR were considered as PCC values. Number of participants with PCC values of vital signs for any visit post-Baseline are presented.
Time Frame: Up to 5.8 years
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | Retigabine IR
Number analyzed (Participants) | 98
Participants
  DBP; decrease of >=15 | 15
  DBP; increase of >=15 | 7
  HR; decrease of >=15 | 15
  HR; increase of >=15 | 18
  SBP; decrease of >=20 | 18
  SBP; increase of >=20 | 8
  Weight; decrease of >=7 percent | 10
  Weight; increase of >=7 percent | 32

10. Primary Outcome: Change From Baseline in Electrocardiogram (ECG) Parameter Including HR
Description: Single measurements of 12-lead ECG were obtained in supine position after at least 10 minutes of rest using an ECG machine to measure HR. Baseline was defined by and taken directly from the Baseline assessments in the parent study NCT01336621. Change from Baseline was defined as post-Baseline value minus Baseline value. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Time Frame: Baseline and up to 5.8 years
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Beats per minute (bpm)
Arm/Group | Retigabine IR
Number analyzed (Participants) | 98
Beats per minute (bpm)
  Visit 1 (Screening); n= 89: number analyzed (Participants) | 89
  Visit 1 (Screening); n= 89 | -2.2 (10.54)
  Visit 2 (Week 13); n= 90: number analyzed (Participants) | 90
  Visit 2 (Week 13); n= 90 | -0.6 (9.77)
  Visit 3 (Week 26); n= 80: number analyzed (Participants) | 80
  Visit 3 (Week 26); n= 80 | -1.5 (9.21)
  Visit 4 (Week 39); n= 71: number analyzed (Participants) | 71
  Visit 4 (Week 39); n= 71 | -1.7 (8.72)
  Visit 5 (Week 52); n= 67: number analyzed (Participants) | 67
  Visit 5 (Week 52); n= 67 | -0.6 (10.30)
  Visit 6 (Week 69); n= 63: number analyzed (Participants) | 63
  Visit 6 (Week 69); n= 63 | -0.2 (9.96)
  Visit 7 (Week 86); n= 56: number analyzed (Participants) | 56
  Visit 7 (Week 86); n= 56 | 1.6 (8.89)
  Visit 8 (Week 104); n= 42: number analyzed (Participants) | 42
  Visit 8 (Week 104); n= 42 | -1.8 (10.30)
  Visit 9 (Week 121); n= 38: number analyzed (Participants) | 38
  Visit 9 (Week 121); n= 38 | 1.7 (11.01)
  Visit 10 (Week 138); n= 37: number analyzed (Participants) | 37
  Visit 10 (Week 138); n= 37 | 1.6 (12.17)
  Visit 11 (Week 156); n= 30: number analyzed (Participants) | 30
  Visit 11 (Week 156); n= 30 | 1.1 (10.23)
  Visit 12 (Week 173); n= 24: number analyzed (Participants) | 24
  Visit 12 (Week 173); n= 24 | -0.8 (13.43)
  Visit 13 (Week 190); n= 19: number analyzed (Participants) | 19
  Visit 13 (Week 190); n= 19 | 2.7 (11.29)
  Visit 14 (Week 208); n= 10: number analyzed (Participants) | 10
  Visit 14 (Week 208); n= 10 | 5.6 (10.41)
  Visit 15 (Week 225); n= 5: number analyzed (Participants) | 5
  Visit 15 (Week 225); n= 5 | -0.2 (8.04)
  Visit 16 (Week 242); n= 4: number analyzed (Participants) | 4
  Visit 16 (Week 242); n= 4 | -4.3 (13.30)
  Visit 17 (Week 260); n= 4: number analyzed (Participants) | 4
  Visit 17 (Week 260); n= 4 | -7.3 (6.95)
  Visit 18 (Week 277); n= 2: number analyzed (Participants) | 2
  Visit 18 (Week 277); n= 2 | 2.5 (9.19)
  Withdrawal visit; n= 83: number analyzed (Participants) | 83
  Withdrawal visit; n= 83 | -1.8 (11.49)
  Follow up visit; n= 59: number analyzed (Participants) | 59
  Follow up visit; n= 59 | -1.1 (11.95)

11. Primary Outcome: Change From Baseline in ECG Parameter Including PR Interval, QRS Duration, Uncorrected QT Interval, Corrected QT by Bazett's Formula (QTcB), Corrected QT by Fridericia's Formula (QTcF) and RR Interval
Description: Single measurements of 12-lead ECG were obtained in supine position after at least 10 minutes of rest using an ECG machine to measure parameters including PR interval, QRS duration, uncorrected QT interval, QTcB, QTcF and RR interval. Baseline was defined by and taken directly from the Baseline assessments in the parent study NCT01336621. Change from Baseline was defined as post-Baseline value minus Baseline value. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Time Frame: Baseline and up to 5.8 years
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Milliseconds (msec)
Arm/Group | Retigabine IR
Number analyzed (Participants) | 98
Milliseconds (msec)
  PR interval; Visit 1 (Screening); n= 86: number analyzed (Participants) | 86
  PR interval; Visit 1 (Screening); n= 86 | 2.4 (13.11)
  PR interval; Visit 2 (Week 13); n= 88: number analyzed (Participants) | 88
  PR interval; Visit 2 (Week 13); n= 88 | 1.3 (15.42)
  PR interval; Visit 3 (Week 26); n= 78: number analyzed (Participants) | 78
  PR interval; Visit 3 (Week 26); n= 78 | 3.2 (12.99)
  PR interval; Visit 4 (Week 39); n= 70: number analyzed (Participants) | 70
  PR interval; Visit 4 (Week 39); n= 70 | 1.2 (13.25)
  PR interval; visit 5 (Week 52); n= 66: number analyzed (Participants) | 66
  PR interval; visit 5 (Week 52); n= 66 | -0.2 (13.17)
  PR interval; Visit 6 (Week 69); n= 62: number analyzed (Participants) | 62
  PR interval; Visit 6 (Week 69); n= 62 | 1.3 (13.93)
  PR interval; Visit 7 (Week 86); n= 54: number analyzed (Participants) | 54
  PR interval; Visit 7 (Week 86); n= 54 | -0.7 (12.58)
  PR interval; Visit 8 (Week 104); n= 42: number analyzed (Participants) | 42
  PR interval; Visit 8 (Week 104); n= 42 | 3.1 (10.85)
  PR interval; Visit 9 (Week 121); n= 38: number analyzed (Participants) | 38
  PR interval; Visit 9 (Week 121); n= 38 | -1.1 (12.79)
  PR interval; Visit 10 (Week 138); n= 37: number analyzed (Participants) | 37
  PR interval; Visit 10 (Week 138); n= 37 | 1.2 (15.13)
  PR interval; Visit 11 (Week 156); n= 30: number analyzed (Participants) | 30
  PR interval; Visit 11 (Week 156); n= 30 | -0.5 (13.50)
  PR interval; Visit 12 (Week 173); n= 24: number analyzed (Participants) | 24
  PR interval; Visit 12 (Week 173); n= 24 | 4.8 (11.89)
  PR interval; Visit 13 (week 190); n= 19: number analyzed (Participants) | 19
  PR interval; Visit 13 (week 190); n= 19 | -2.1 (10.19)
  PR interval; Visit 14 (Week 208); n= 10: number analyzed (Participants) | 10
  PR interval; Visit 14 (Week 208); n= 10 | 7.8 (15.03)
  PR interval; Visit 15 (Week 225); n= 5: number analyzed (Participants) | 5
  PR interval; Visit 15 (Week 225); n= 5 | 8.4 (7.23)
  PR interval; Visit 16 (Week 242); n= 4: number analyzed (Participants) | 4
  PR interval; Visit 16 (Week 242); n= 4 | -3.0 (8.04)
  PR interval; Visit 17 (Week 260); n= 4: number analyzed (Participants) | 4
  PR interval; Visit 17 (Week 260); n= 4 | 9.3 (11.09)
  PR interval; Visit 18 (Week 277); n= 2: number analyzed (Participants) | 2
  PR interval; Visit 18 (Week 277); n= 2 | -5.5 (7.78)
  PR interval; Withdrawal visit; n= 81: number analyzed (Participants) | 81
  PR interval; Withdrawal visit; n= 81 | 3.6 (13.86)
  PR interval; follow up visit; n= 57: number analyzed (Participants) | 57
  PR interval; follow up visit; n= 57 | 3.7 (12.43)
  QRS duration; Visit 1 (Screening); n= 88: number analyzed (Participants) | 88
  QRS duration; Visit 1 (Screening); n= 88 | -0.1 (6.37)
  QRS duration; Visit 2 (Week 13); n= 89: number analyzed (Participants) | 89
  QRS duration; Visit 2 (Week 13); n= 89 | 0.2 (6.99)
  QRS duration; Visit 3 (Week 26); n= 80: number analyzed (Participants) | 80
  QRS duration; Visit 3 (Week 26); n= 80 | 1.1 (8.77)
  QRS duration; Visit 4 (Week 39); n= 71: number analyzed (Participants) | 71
  QRS duration; Visit 4 (Week 39); n= 71 | 1.1 (7.10)
  QRS duration; Visit 5 (Week 52); n= 67: number analyzed (Participants) | 67
  QRS duration; Visit 5 (Week 52); n= 67 | 0.9 (9.81)
  QRS duration; Visit 6 (Week 69); n= 63: number analyzed (Participants) | 63
  QRS duration; Visit 6 (Week 69); n= 63 | 1.9 (8.56)
  QRS duration; Visit 7 (Week 86); n= 55: number analyzed (Participants) | 55
  QRS duration; Visit 7 (Week 86); n= 55 | -0.4 (7.20)
  QRS duration; Visit 8 (Week 104); n= 42: number analyzed (Participants) | 42
  QRS duration; Visit 8 (Week 104); n= 42 | 0.1 (6.40)
  QRS duration; Visit 9 (Week 121); n= 38: number analyzed (Participants) | 38
  QRS duration; Visit 9 (Week 121); n= 38 | -0.7 (7.79)
  QRS duration; Visit 10 (Week 138); n= 37: number analyzed (Participants) | 37
  QRS duration; Visit 10 (Week 138); n= 37 | -2.0 (7.85)
  QRS duration; Visit 11 (Week 156); n= 30: number analyzed (Participants) | 30
  QRS duration; Visit 11 (Week 156); n= 30 | -3.3 (9.54)
  QRS duration; Visit 12 (Week 173); n= 24: number analyzed (Participants) | 24
  QRS duration; Visit 12 (Week 173); n= 24 | -1.3 (9.04)
  QRS duration; Visit 13 (Week 190); n= 19: number analyzed (Participants) | 19
  QRS duration; Visit 13 (Week 190); n= 19 | -4.9 (8.80)
  QRS duration; Visit 14 (Week 208); n= 10: number analyzed (Participants) | 10
  QRS duration; Visit 14 (Week 208); n= 10 | -6.1 (6.34)
  QRS duration; Visit 15 (Week 225); n= 5: number analyzed (Participants) | 5
  QRS duration; Visit 15 (Week 225); n= 5 | -2.9 (3.44)
  QRS duration; Visit 16 (Week 242); n= 4: number analyzed (Participants) | 4
  QRS duration; Visit 16 (Week 242); n= 4 | -5.9 (9.58)
  QRS duration; Visit 17 (Week 260); n= 4: number analyzed (Participants) | 4
  QRS duration; Visit 17 (Week 260); n= 4 | -7.8 (5.19)
  QRS duration; Visit 18 (Week 277); n= 2: number analyzed (Participants) | 2
  QRS duration; Visit 18 (Week 277); n= 2 | -4.5 (2.12)
  QRS duration; withdrawal visit; n= 82: number analyzed (Participants) | 82
  QRS duration; withdrawal visit; n= 82 | -2.5 (9.49)
  QRS duration; follow up visit; n= 59: number analyzed (Participants) | 59
  QRS duration; follow up visit; n= 59 | 0.0 (11.90)
  Uncorrected QT interval;Visit 1 (Screening); n= 85: number analyzed (Participants) | 85
  Uncorrected QT interval;Visit 1 (Screening); n= 85 | 10.1 (26.19)
  Uncorrected QT interval; Visit 2 (Week 13); n= 88: number analyzed (Participants) | 88
  Uncorrected QT interval; Visit 2 (Week 13); n= 88 | 4.9 (23.43)
  Uncorrected QT interval; Visit 3 (Week 26); n= 78: number analyzed (Participants) | 78
  Uncorrected QT interval; Visit 3 (Week 26); n= 78 | 7.9 (23.44)
  Uncorrected QT interval; Visit 4 (Week 39); n= 69: number analyzed (Participants) | 69
  Uncorrected QT interval; Visit 4 (Week 39); n= 69 | 9.3 (23.77)
  Uncorrected QT interval; Visit 5 (Week 52); n= 65: number analyzed (Participants) | 65
  Uncorrected QT interval; Visit 5 (Week 52); n= 65 | 6.6 (25.18)
  Uncorrected QT interval; Visit 6 (Week 69); n= 61: number analyzed (Participants) | 61
  Uncorrected QT interval; Visit 6 (Week 69); n= 61 | 7.4 (26.39)
  Uncorrected QT interval; Visit 7 (Week 86); n= 53: number analyzed (Participants) | 53
  Uncorrected QT interval; Visit 7 (Week 86); n= 53 | -1.6 (23.81)
  Uncorrected QT interval; Visit 8 (Week 104); n= 41: number analyzed (Participants) | 41
  Uncorrected QT interval; Visit 8 (Week 104); n= 41 | 6.0 (26.77)
  Uncorrected QT interval; Visit 9 (Week 121); n= 37: number analyzed (Participants) | 37
  Uncorrected QT interval; Visit 9 (Week 121); n= 37 | -0.5 (24.52)
  Uncorrected QT interval; Visit 10 (Week 138);n= 36: number analyzed (Participants) | 36
  Uncorrected QT interval; Visit 10 (Week 138);n= 36 | -8.7 (33.60)
  Uncorrected QT interval; Visit 11 (Week 156);n= 29: number analyzed (Participants) | 29
  Uncorrected QT interval; Visit 11 (Week 156);n= 29 | -4.9 (33.01)
  Uncorrected QT interval; Visit 12 (Week 173);n= 23: number analyzed (Participants) | 23
  Uncorrected QT interval; Visit 12 (Week 173);n= 23 | 4.7 (25.06)
  Uncorrected QT interval; Visit 13 (Week 190);n= 19: number analyzed (Participants) | 19
  Uncorrected QT interval; Visit 13 (Week 190);n= 19 | -1.9 (26.01)
  Uncorrected QT interval; Visit 14 (Week 208);n= 10: number analyzed (Participants) | 10
  Uncorrected QT interval; Visit 14 (Week 208);n= 10 | -17.0 (27.93)
  Uncorrected QT interval; Visit 15 (Week 225);n= 5: number analyzed (Participants) | 5
  Uncorrected QT interval; Visit 15 (Week 225);n= 5 | -1.5 (5.68)
  Uncorrected QT interval; Visit 16 (Week 242);n= 4: number analyzed (Participants) | 4
  Uncorrected QT interval; Visit 16 (Week 242);n= 4 | 3.1 (26.90)
  Uncorrected QT interval; Visit 17 (Week 260);n= 4: number analyzed (Participants) | 4
  Uncorrected QT interval; Visit 17 (Week 260);n= 4 | 17.5 (36.08)
  Uncorrected QT interval; Visit 18 (Week 277);n= 2: number analyzed (Participants) | 2
  Uncorrected QT interval; Visit 18 (Week 277);n= 2 | -3.5 (36.06)
  Uncorrected QT interval; withdrawal visit; n= 80: number analyzed (Participants) | 80
  Uncorrected QT interval; withdrawal visit; n= 80 | 5.2 (29.01)
  Uncorrected QT interval; follow up visit; n= 56: number analyzed (Participants) | 56
  Uncorrected QT interval; follow up visit; n= 56 | 2.7 (28.41)
  QTcB; Visit 1 (Screening); n= 85: number analyzed (Participants) | 85
  QTcB; Visit 1 (Screening); n= 85 | 5.0 (17.35)
  QTcB; Visit 2 (Week 13); n= 88: number analyzed (Participants) | 88
  QTcB; Visit 2 (Week 13); n= 88 | 3.2 (18.52)
  QTcB; Visit 3 (Week 26); n= 78: number analyzed (Participants) | 78
  QTcB; Visit 3 (Week 26); n= 78 | 4.0 (16.48)
  QTcB; Visit 4 (Week 39); n= 69: number analyzed (Participants) | 69
  QTcB; Visit 4 (Week 39); n= 69 | 6.0 (17.27)
  QTcB; Visit 5 (Week 52); n= 65: number analyzed (Participants) | 65
  QTcB; Visit 5 (Week 52); n= 65 | 5.8 (17.14)
  QTcB; Visit 6 (Week 69); n= 61: number analyzed (Participants) | 61
  QTcB; Visit 6 (Week 69); n= 61 | 6.8 (15.01)
  QTcB; Visit 7 (Week 86); n= 53: number analyzed (Participants) | 53
  QTcB; Visit 7 (Week 86); n= 53 | 4.3 (15.71)
  QTcB; Visit 8 (Week 104); n= 41: number analyzed (Participants) | 41
  QTcB; Visit 8 (Week 104); n= 41 | 2.5 (20.70)
  QTcB; Visit 9 (Week 121); n= 37: number analyzed (Participants) | 37
  QTcB; Visit 9 (Week 121); n= 37 | 4.9 (16.01)
  QTcB; Visit 10 (Week 138); n= 36: number analyzed (Participants) | 36
  QTcB; Visit 10 (Week 138); n= 36 | -2.8 (16.46)
  QTcB; Visit 11 (Week 156); n= 29: number analyzed (Participants) | 29
  QTcB; Visit 11 (Week 156); n= 29 | -0.3 (19.63)
  QTcB; Visit 12 (Week 173); n= 23: number analyzed (Participants) | 23
  QTcB; Visit 12 (Week 173); n= 23 | 4.2 (24.12)
  QTcB; Visit 13 (Week 190); n= 19: number analyzed (Participants) | 19
  QTcB; Visit 13 (Week 190); n= 19 | 3.9 (20.16)
  QTcB; Visit 14 (Week 208); n= 10: number analyzed (Participants) | 10
  QTcB; Visit 14 (Week 208); n= 10 | -1.6 (14.91)
  QTcB; Visit 15 (Week 225); n= 5: number analyzed (Participants) | 5
  QTcB; Visit 15 (Week 225); n= 5 | -1.9 (18.26)
  QTcB; Visit 16 (Week 242); n= 4: number analyzed (Participants) | 4
  QTcB; Visit 16 (Week 242); n= 4 | -9.8 (15.09)
  QTcB; Visit 17 (Week 260); n= 4: number analyzed (Participants) | 4
  QTcB; Visit 17 (Week 260); n= 4 | -2.0 (27.12)
  QTcB; Visit 18 (Week 277); n= 2: number analyzed (Participants) | 2
  QTcB; Visit 18 (Week 277); n= 2 | 4.5 (17.68)
  QTcB; withdrawal visit; n= 80: number analyzed (Participants) | 80
  QTcB; withdrawal visit; n= 80 | -0.7 (20.78)
  QTcB; follow up visit; n= 56: number analyzed (Participants) | 56
  QTcB; follow up visit; n= 56 | -1.0 (17.84)
  QTcF; Visit 1 (Screening); n= 85: number analyzed (Participants) | 85
  QTcF; Visit 1 (Screening); n= 85 | 6.8 (16.11)
  QTcF; Visit 2 (Week 13); n= 88: number analyzed (Participants) | 88
  QTcF; Visit 2 (Week 13); n= 88 | 3.7 (15.74)
  QTcF; Visit 3 (Week 26); n= 78: number analyzed (Participants) | 78
  QTcF; Visit 3 (Week 26); n= 78 | 5.4 (15.01)
  QTcF; Visit 4 (Week 39); n= 69: number analyzed (Participants) | 69
  QTcF; Visit 4 (Week 39); n= 69 | 7.1 (16.58)
  QTcF; Visit 5 (Week 52); n= 65: number analyzed (Participants) | 65
  QTcF; Visit 5 (Week 52); n= 65 | 6.1 (14.92)
  QTcF; Visit 6 (Week 69); n= 61: number analyzed (Participants) | 61
  QTcF; Visit 6 (Week 69); n= 61 | 7.1 (14.47)
  QTcF; Visit 7 (Week 86); n= 53: number analyzed (Participants) | 53
  QTcF; Visit 7 (Week 86); n= 53 | 2.3 (16.04)
  QTcF; Visit 8 (Week 104); n= 41: number analyzed (Participants) | 41
  QTcF; Visit 8 (Week 104); n= 41 | 3.7 (19.31)
  QTcF; Visit 9 (Week 121); n= 37: number analyzed (Participants) | 37
  QTcF; Visit 9 (Week 121); n= 37 | 3.0 (12.90)
  QTcF; Visit 10 (Week 138); n= 36: number analyzed (Participants) | 36
  QTcF; Visit 10 (Week 138); n= 36 | -4.8 (18.22)
  QTcF; Visit 11 (Week 156); n= 29: number analyzed (Participants) | 29
  QTcF; Visit 11 (Week 156); n= 29 | -1.8 (21.86)
  QTcF; Visit 12 (Week 173); n= 23: number analyzed (Participants) | 23
  QTcF; Visit 12 (Week 173); n= 23 | 4.6 (17.51)
  QTcF; Visit 13 (Week 190); n= 19: number analyzed (Participants) | 19
  QTcF; Visit 13 (Week 190); n= 19 | 1.9 (17.47)
  QTcF; Visit 14 (Week 208); n= 10: number analyzed (Participants) | 10
  QTcF; Visit 14 (Week 208); n= 10 | -7.0 (14.99)
  QTcF; Visit 15 (Week 225); n= 5: number analyzed (Participants) | 5
  QTcF; Visit 15 (Week 225); n= 5 | -1.6 (10.53)
  QTcF; Visit 16 (Week 242); n= 4: number analyzed (Participants) | 4
  QTcF; Visit 16 (Week 242); n= 4 | -5.4 (8.96)
  QTcF; Visit 17 (Week 260); n= 4: number analyzed (Participants) | 4
  QTcF; Visit 17 (Week 260); n= 4 | 5.3 (29.75)
  QTcF; Visit 18 (Week 277); n= 2: number analyzed (Participants) | 2
  QTcF; Visit 18 (Week 277); n= 2 | 2.0 (24.04)
  QTcF; withdrawal visit; n= 80: number analyzed (Participants) | 80
  QTcF; withdrawal visit; n= 80 | 1.3 (18.24)
  QTcF; follow up visit; n= 56: number analyzed (Participants) | 56
  QTcF; follow up visit; n= 56 | 0.3 (15.49)
  RR interval; visit 1 (Screening); n= 89: number analyzed (Participants) | 89
  RR interval; visit 1 (Screening); n= 89 | 27.9 (120.57)
  RR interval; visit 2 (Week 13); n= 90: number analyzed (Participants) | 90
  RR interval; visit 2 (Week 13); n= 90 | 12.2 (115.82)
  RR interval; visit 3 (Week 26); n= 80: number analyzed (Participants) | 80
  RR interval; visit 3 (Week 26); n= 80 | 20.5 (110.48)
  RR interval; visit 4 (Week 39); n= 71: number analyzed (Participants) | 71
  RR interval; visit 4 (Week 39); n= 71 | 22.4 (107.77)
  RR interval; visit 5 (Week 52); n= 67: number analyzed (Participants) | 67
  RR interval; visit 5 (Week 52); n= 67 | 10.3 (128.05)
  RR interval; visit 6 (Week 69); n= 63: number analyzed (Participants) | 63
  RR interval; visit 6 (Week 69); n= 63 | 6.2 (127.01)
  RR interval; visit 7 (Week 86); n= 56: number analyzed (Participants) | 56
  RR interval; visit 7 (Week 86); n= 56 | -18.5 (102.45)
  RR interval; visit 8 (Week 104); n= 42: number analyzed (Participants) | 42
  RR interval; visit 8 (Week 104); n= 42 | 23.7 (121.17)
  RR interval; visit 9 (Week 121); n= 38: number analyzed (Participants) | 38
  RR interval; visit 9 (Week 121); n= 38 | -17.5 (134.18)
  RR interval; visit 10 (Week 138); n= 37: number analyzed (Participants) | 37
  RR interval; visit 10 (Week 138); n= 37 | -19.6 (145.64)
  RR interval; visit 11 (Week 156); n= 30: number analyzed (Participants) | 30
  RR interval; visit 11 (Week 156); n= 30 | -16.0 (120.50)
  RR interval; visit 12 (Week 173); n= 24: number analyzed (Participants) | 24
  RR interval; visit 12 (Week 173); n= 24 | 12.9 (163.66)
  RR interval; visit 13 (Week 190); n= 19: number analyzed (Participants) | 19
  RR interval; visit 13 (Week 190); n= 19 | -19.5 (138.03)
  RR interval; visit 14 (Week 208); n= 10: number analyzed (Participants) | 10
  RR interval; visit 14 (Week 208); n= 10 | -70.7 (130.51)
  RR interval; visit 15 (Week 225); n= 5: number analyzed (Participants) | 5
  RR interval; visit 15 (Week 225); n= 5 | -2.8 (108.30)
  RR interval; visit 16 (Week 242); n= 4: number analyzed (Participants) | 4
  RR interval; visit 16 (Week 242); n= 4 | 56.6 (165.75)
  RR interval; visit 17 (Week 260); n= 4: number analyzed (Participants) | 4
  RR interval; visit 17 (Week 260); n= 4 | 83.5 (91.72)
  RR interval; visit 18 (Week 277); n= 2: number analyzed (Participants) | 2
  RR interval; visit 18 (Week 277); n= 2 | -30.0 (86.27)
  RR interval; withdrawal visit; n= 83: number analyzed (Participants) | 83
  RR interval; withdrawal visit; n= 83 | 29.1 (152.19)
  RR interval; follow up visit; n= 59: number analyzed (Participants) | 59
  RR interval; follow up visit; n= 59 | 15.9 (150.13)

12. Primary Outcome: Number of Participants With Clinical Chemistry Parameters of PCC
Description: Number of participants with chemistry parameters of PCC at 'any visit post-Baseline' are presented. Chemistry parameters for which PCC values were identified were alanine aminotransferase (ALT) (if value >=3 * upper limit of normal [ULN]), alkaline phosphatase (alk.phosphatase) (if value >=3*ULN), aspartate aminotransferase (AST) (if value >=3*ULN), calcium (if value <=1.8962 or >=2.8692), carbon-di-oxide (CO2) (if value <=18 or >=36), chloride (if value <=92 or >=112), creatine kinase (if value >=3*ULN), direct bilirubin (if value >=1.5*ULN), glucose (if value <=2.7755 or >=11.102), lactate dehydrogenase (LD) (if value >=3*ULN), magnesium (if value <0.36 or >2.50), potassium (if value <=3.0 or >=6.0), sodium (if value <=127 or >=153), total bilirubin (if value >=1.5*ULN), total protein (if value <45 or >100), blood urea nitrogen (BUN) (if value >=14.28). Only those participants with data available at specific time points were analyzed (represented by n=X in the category titles).
Time Frame: Up to 5.8 years
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | Retigabine IR
Number analyzed (Participants) | 98
Participants
  ALT; high; n= 98 | 2
  Alk.phosphatase; high; n= 98 | 0
  AST; high; n= 98 | 1
  Calcium; high; n= 98 | 0
  Calcium; low; n= 98 | 0
  CO2 content/bicarbonate; high; n= 98 | 0
  CO2 content/bicrbonate; low; n= 98 | 10
  Chloride; high; n= 98 | 6
  Chloride; low; n= 98 | 2
  Creatine kinase; high; n= 98 | 6
  Creatinine; high; n= 98 | 0
  Direct bilirubin; high; n= 98 | 0
  Glucose; high; n= 98 | 3
  Glucose; low; n= 98 | 1
  LD ; high; n= 98 | 1
  Magnesium; high; n= 98 | 0
  Magnesium; low; n= 98 | 0
  Potassium; high; n= 98 | 1
  Potassium; low; n= 98 | 0
  Sodium; high; n= 91: number analyzed (Participants) | 91
  Sodium; high; n= 91 | 0
  Sodium; low; n= 91: number analyzed (Participants) | 91
  Sodium; low; n= 91 | 2
  Total bilirubin; high; n= 98 | 1
  Total protein; high; n= 98 | 0
  Total protein; low; n= 98 | 0
  BUN; high; n= 91: number analyzed (Participants) | 91
  BUN; high; n= 91 | 0

13. Primary Outcome: Number of Participants With Hematology Parameters of PCC
Description: Blood samples were collected from participants to evaluate hematology parameters. Number of participants with clinical hematology parameters of PCC at 'any visit post-Baseline' are presented. Hematology parameters for which PCC values were identified were eosinophils (if value is >0.8), hematocrit (if value is <=0.32 for males and <=0.28 for females), platelet count (if value is <=100 or >=550), total neutrophils (if value is <=1.8), white blood cells (WBC) (if value is <=2.8 or >=16). Only those participants with data available at specific time points were analyzed (represented by n=X in the category titles).
Time Frame: Up to 5.8 years
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | Retigabine IR
Number analyzed (Participants) | 98
Participants
  Eosinophils; high; n= 98 | 7
  Hematocrit; low; n= 98 | 4
  Hemoglobin; low; n= 98 | 3
  Platelet count; high; n= 98 | 1
  Platelet count; low; n= 98 | 4
  Total neutrophils; low; n= 98 | 20
  WBC; high; n= 91: number analyzed (Participants) | 91
  WBC; high; n= 91 | 2
  WBC; low; n= 91: number analyzed (Participants) | 91
  WBC; low; n= 91 | 3

14. Primary Outcome: Number of Participants With Urinalysis Parameters of PCC
Description: Urine samples were collected from participants at specific time points. Number of participants with urinalysis parameters of PCC at 'any visit post-Baseline' are presented. Urinalysis parameters for which PCC values were identified were albumin/creatinine ratio (if value is >11.3), red blood cells (RBC) (if value is 3-5 or higher), WBC (if value is 5-10 or higher for male and 10-15 or higher for females), specific gravity (if value is <1.001 or >1.035) and potential of hydrogen (pH) (if value is <4.6 or >8.0). Only those participants with data available at specific time points were analyzed (represented by n=X in the category titles).
Time Frame: Up to 5.8 years
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | Retigabine IR
Number analyzed (Participants) | 98
Participants
  Albumin/creatinine ratio; high; n= 96: number analyzed (Participants) | 96
  Albumin/creatinine ratio; high; n= 96 | 4
  RBC; high; n= 98 | 54
  WBC; high; n= 91: number analyzed (Participants) | 91
  WBC; high; n= 91 | 59
  Specific gravity; high; n= 91: number analyzed (Participants) | 91
  Specific gravity; high; n= 91 | 4
  Specific gravity; low; n= 91: number analyzed (Participants) | 91
  Specific gravity; low; n= 91 | 0
  pH; high; n= 98 | 1
  pH; low; n= 98 | 0

15. Primary Outcome: Change From Baseline in Albumin and Total Protein
Description: Blood samples were collected from participants for evaluation of change from Baseline in clinical chemistry parameters including albumin and total protein. Baseline was defined by and taken directly from the Baseline assessments in the parent study NCT01336621. Change from Baseline was defined as post-Baseline value minus Baseline value. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Time Frame: Baseline and up to 5.8 years
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Gram per liter (G/L)
Arm/Group | Retigabine IR
Number analyzed (Participants) | 98
Gram per liter (G/L)
  Albumin; visit 1 (Screening); n= 83: number analyzed (Participants) | 83
  Albumin; visit 1 (Screening); n= 83 | -1.6 (2.72)
  Albumin; visit 2 (Week 13); n= 87: number analyzed (Participants) | 87
  Albumin; visit 2 (Week 13); n= 87 | -0.9 (2.70)
  Albumin; visit 3 (Week 26); n= 75: number analyzed (Participants) | 75
  Albumin; visit 3 (Week 26); n= 75 | -0.8 (2.83)
  Albumin; visit 4 (Week 39); n= 70: number analyzed (Participants) | 70
  Albumin; visit 4 (Week 39); n= 70 | -0.7 (3.09)
  Albumin; visit 5 (Week 52); n= 65: number analyzed (Participants) | 65
  Albumin; visit 5 (Week 52); n= 65 | -1.5 (3.25)
  Albumin; visit 6 (Week 69); n= 62: number analyzed (Participants) | 62
  Albumin; visit 6 (Week 69); n= 62 | -1.1 (3.11)
  Albumin; visit 7 (Week 86); n= 54: number analyzed (Participants) | 54
  Albumin; visit 7 (Week 86); n= 54 | -1.0 (2.70)
  Albumin; visit 8 (Week 104); n= 42: number analyzed (Participants) | 42
  Albumin; visit 8 (Week 104); n= 42 | -1.6 (3.05)
  Albumin; visit 9 (Week 121); n= 39: number analyzed (Participants) | 39
  Albumin; visit 9 (Week 121); n= 39 | -2.1 (2.88)
  Albumin; visit 10 (Week 138); n= 36: number analyzed (Participants) | 36
  Albumin; visit 10 (Week 138); n= 36 | -2.2 (3.16)
  Albumin; visit 11 (Week 156); n= 30: number analyzed (Participants) | 30
  Albumin; visit 11 (Week 156); n= 30 | -3.0 (3.62)
  Albumin; visit 12 (Week 173); n= 23: number analyzed (Participants) | 23
  Albumin; visit 12 (Week 173); n= 23 | -1.7 (2.82)
  Albumin; visit 13 (Week 190); n= 19: number analyzed (Participants) | 19
  Albumin; visit 13 (Week 190); n= 19 | -2.9 (3.62)
  Albumin; visit14 (Week 208); n= 10: number analyzed (Participants) | 10
  Albumin; visit14 (Week 208); n= 10 | -3.9 (3.78)
  Albumin; visit 15 (Week 225); n= 5: number analyzed (Participants) | 5
  Albumin; visit 15 (Week 225); n= 5 | -3.4 (1.52)
  Albumin; visit 16 (Week242); n= 4: number analyzed (Participants) | 4
  Albumin; visit 16 (Week242); n= 4 | -4.3 (1.26)
  Albumin; visit 17 (Week 260); n= 4: number analyzed (Participants) | 4
  Albumin; visit 17 (Week 260); n= 4 | -4.0 (1.15)
  Albumin; visit 18 (Week 277); n= 2: number analyzed (Participants) | 2
  Albumin; visit 18 (Week 277); n= 2 | -4.5 (0.71)
  Albumin; withdrawal visit; n= 79: number analyzed (Participants) | 79
  Albumin; withdrawal visit; n= 79 | -1.8 (3.11)
  Albumin; follow up visit; n= 60: number analyzed (Participants) | 60
  Albumin; follow up visit; n= 60 | -2.3 (3.42)
  Total protein; visit 1 (Screening); n= 83: number analyzed (Participants) | 83
  Total protein; visit 1 (Screening); n= 83 | -2.0 (4.57)
  Total protein; visit 2 (Week 13); n= 87: number analyzed (Participants) | 87
  Total protein; visit 2 (Week 13); n= 87 | -1.0 (4.59)
  Total protein; visit 3 (Week 26); n= 75: number analyzed (Participants) | 75
  Total protein; visit 3 (Week 26); n= 75 | -1.5 (5.15)
  Total protein; visit 4 (Week 39); n= 70: number analyzed (Participants) | 70
  Total protein; visit 4 (Week 39); n= 70 | -1.8 (4.13)
  Total protein; visit 5 (Week 52); n= 65: number analyzed (Participants) | 65
  Total protein; visit 5 (Week 52); n= 65 | -2.6 (4.74)
  Total protein; visit 6 (Week 69); n= 62: number analyzed (Participants) | 62
  Total protein; visit 6 (Week 69); n= 62 | -1.4 (4.09)
  Total protein; visit 7 (Week 86); n= 54: number analyzed (Participants) | 54
  Total protein; visit 7 (Week 86); n= 54 | -1.0 (4.44)
  Total protein; visit 8 (Week 104); n= 42: number analyzed (Participants) | 42
  Total protein; visit 8 (Week 104); n= 42 | -1.5 (4.65)
  Total protein; visit 9 (Week 121); n= 39: number analyzed (Participants) | 39
  Total protein; visit 9 (Week 121); n= 39 | -2.1 (4.58)
  Total protein; visit 10 (Week 138); n= 36: number analyzed (Participants) | 36
  Total protein; visit 10 (Week 138); n= 36 | -2.7 (4.90)
  Total protein; visit 11 (Week 156); n= 30: number analyzed (Participants) | 30
  Total protein; visit 11 (Week 156); n= 30 | -3.2 (5.40)
  Total protein; visit 12 (Week 173); n= 23: number analyzed (Participants) | 23
  Total protein; visit 12 (Week 173); n= 23 | -1.1 (4.07)
  Total protein; visit 13 (Week 190); n= 19: number analyzed (Participants) | 19
  Total protein; visit 13 (Week 190); n= 19 | -1.9 (5.57)
  Total protein; visit 14 (Week 208); n= 10: number analyzed (Participants) | 10
  Total protein; visit 14 (Week 208); n= 10 | -3.1 (3.41)
  Total protein; visit 15 (Week 225); n= 5: number analyzed (Participants) | 5
  Total protein; visit 15 (Week 225); n= 5 | -3.4 (2.51)
  Total protein; visit 16 (Week 242); n= 4: number analyzed (Participants) | 4
  Total protein; visit 16 (Week 242); n= 4 | -3.8 (4.99)
  Total protein; visit 17 (Week 260); n= 4: number analyzed (Participants) | 4
  Total protein; visit 17 (Week 260); n= 4 | -2.3 (3.30)
  Total protein; visit 18 (Week 277); n= 2: number analyzed (Participants) | 2
  Total protein; visit 18 (Week 277); n= 2 | -4.5 (2.12)
  Total protein; withdrawal visit; n= 79: number analyzed (Participants) | 79
  Total protein; withdrawal visit; n= 79 | -2.5 (5.27)
  Total protein; follow up visit; n= 60: number analyzed (Participants) | 60
  Total protein; follow up visit; n= 60 | -2.1 (6.12)

16. Primary Outcome: Change From Baseline in Alk. Phosphatase, ALT, AST, Creatine Kinase and LD Levels
Description: Blood samples were collected from participants for evaluation of change from Baseline in clinical chemistry parameters including alk. phosphatase, ALT, AST, creatine kinase and LD. Baseline was defined by and taken directly from the Baseline assessments in the parent study NCT01336621. Change from Baseline was defined as post-Baseline value minus Baseline value. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Time Frame: Baseline and up to 5.8 years
Population: Safety Population
Measure: Mean (Standard Deviation); unit: International unit per liter (IU/L)
Arm/Group | Retigabine IR
Number analyzed (Participants) | 98
International unit per liter (IU/L)
  Alk. phosphatase; visit 1 (Screening); n= 82: number analyzed (Participants) | 82
  Alk. phosphatase; visit 1 (Screening); n= 82 | -2.7 (15.51)
  Alk. phosphatase; visit 2 (Week 13); n= 86: number analyzed (Participants) | 86
  Alk. phosphatase; visit 2 (Week 13); n= 86 | 1.1 (14.02)
  Alk. phosphatase; visit 3 (Week 26); n= 75: number analyzed (Participants) | 75
  Alk. phosphatase; visit 3 (Week 26); n= 75 | 3.5 (15.80)
  Alk. phosphatase; visit 4 (week 39); n= 70: number analyzed (Participants) | 70
  Alk. phosphatase; visit 4 (week 39); n= 70 | 3.9 (15.46)
  Alk. phosphatase; visit 5 (Week 52); n= 65: number analyzed (Participants) | 65
  Alk. phosphatase; visit 5 (Week 52); n= 65 | 1.0 (15.36)
  Alk. phosphatase; visit 6 (Week 69); n= 62: number analyzed (Participants) | 62
  Alk. phosphatase; visit 6 (Week 69); n= 62 | 4.1 (14.22)
  Alk. phosphatase; visit 7 (Week 86); n= 54: number analyzed (Participants) | 54
  Alk. phosphatase; visit 7 (Week 86); n= 54 | 4.0 (16.01)
  Alk. phosphatase; visit 8 (Week 104); n= 42: number analyzed (Participants) | 42
  Alk. phosphatase; visit 8 (Week 104); n= 42 | -0.3 (18.27)
  Alk. phosphatase; visit 9 (Week 121); n= 39: number analyzed (Participants) | 39
  Alk. phosphatase; visit 9 (Week 121); n= 39 | 2.4 (16.33)
  Alk. phosphatase; visit 10 (Week 138); n= 36: number analyzed (Participants) | 36
  Alk. phosphatase; visit 10 (Week 138); n= 36 | 2.2 (21.08)
  Alk. phosphatase; visit 11 (Week 156); n= 30: number analyzed (Participants) | 30
  Alk. phosphatase; visit 11 (Week 156); n= 30 | -1.4 (18.49)
  Alk. phosphatase; visit 12 (Week 173); n= 23: number analyzed (Participants) | 23
  Alk. phosphatase; visit 12 (Week 173); n= 23 | 5.5 (20.76)
  Alk. phosphatase; visit 13 (Week 190); n= 19: number analyzed (Participants) | 19
  Alk. phosphatase; visit 13 (Week 190); n= 19 | 6.3 (23.61)
  Alk. phosphatase; visit 14 (Week 208); n= 10: number analyzed (Participants) | 10
  Alk. phosphatase; visit 14 (Week 208); n= 10 | 6.1 (19.84)
  Alk. phosphatase; visit 15 (Week 225); n= 5: number analyzed (Participants) | 5
  Alk. phosphatase; visit 15 (Week 225); n= 5 | 5.8 (16.95)
  Alk. phosphatase; visit 16 (Week 242); n= 4: number analyzed (Participants) | 4
  Alk. phosphatase; visit 16 (Week 242); n= 4 | 9.5 (15.55)
  Alk. phosphatase; visit 17 (Week 260); n= 4: number analyzed (Participants) | 4
  Alk. phosphatase; visit 17 (Week 260); n= 4 | 7.3 (7.14)
  Alk. phosphatase; visit 18 (Week 277); n= 2: number analyzed (Participants) | 2
  Alk. phosphatase; visit 18 (Week 277); n= 2 | -4.5 (10.61)
  Alk. phosphatase; withdrawal visit; n= 78: number analyzed (Participants) | 78
  Alk. phosphatase; withdrawal visit; n= 78 | 2.5 (19.86)
  Alk. phosphatase; follow up visit; n= 60: number analyzed (Participants) | 60
  Alk. phosphatase; follow up visit; n= 60 | -0.3 (19.59)
  ALT; visit 1 (Screening); n= 83: number analyzed (Participants) | 83
  ALT; visit 1 (Screening); n= 83 | 1.3 (10.90)
  ALT; visit 2 (Week 13); n= 87: number analyzed (Participants) | 87
  ALT; visit 2 (Week 13); n= 87 | 3.4 (23.41)
  ALT; visit 3 (Week 26); n= 76: number analyzed (Participants) | 76
  ALT; visit 3 (Week 26); n= 76 | 1.0 (23.35)
  ALT; visit 4 (Week 39); n= 70: number analyzed (Participants) | 70
  ALT; visit 4 (Week 39); n= 70 | -0.5 (10.22)
  ALT; visit 5 (Week 52); n= 65: number analyzed (Participants) | 65
  ALT; visit 5 (Week 52); n= 65 | -0.4 (8.21)
  ALT; visit 6 (Week 69); n= 62: number analyzed (Participants) | 62
  ALT; visit 6 (Week 69); n= 62 | -0.0 (11.51)
  ALT; visit 7 (Week 86); n= 54: number analyzed (Participants) | 54
  ALT; visit 7 (Week 86); n= 54 | -1.9 (10.02)
  ALT; visit 8 (Week 104); n= 42: number analyzed (Participants) | 42
  ALT; visit 8 (Week 104); n= 42 | -1.5 (8.58)
  ALT; visit 9 (Week 121); n= 39: number analyzed (Participants) | 39
  ALT; visit 9 (Week 121); n= 39 | 0.4 (8.80)
  ALT; visit 10 (Week 138); n= 36: number analyzed (Participants) | 36
  ALT; visit 10 (Week 138); n= 36 | 3.4 (21.74)
  ALT; visit 11 (Week 156); n= 29: number analyzed (Participants) | 29
  ALT; visit 11 (Week 156); n= 29 | -1.1 (8.21)
  ALT; visit 12 (Week 173); n= 23: number analyzed (Participants) | 23
  ALT; visit 12 (Week 173); n= 23 | -1.3 (7.97)
  ALT; visit 13 (Week 190); n= 19: number analyzed (Participants) | 19
  ALT; visit 13 (Week 190); n= 19 | 0.0 (8.10)
  ALT; visit 14 (Week 208); n= 10: number analyzed (Participants) | 10
  ALT; visit 14 (Week 208); n= 10 | 0.7 (7.32)
  ALT; visit 15 (Week 225); n= 5: number analyzed (Participants) | 5
  ALT; visit 15 (Week 225); n= 5 | -2.0 (4.47)
  ALT; visit 16 (Week 242); n= 4: number analyzed (Participants) | 4
  ALT; visit 16 (Week 242); n= 4 | -0.5 (8.54)
  ALT; visit 17 (Week 260); n= 4: number analyzed (Participants) | 4
  ALT; visit 17 (Week 260); n= 4 | 0.0 (6.98)
  ALT; visit 18 (Week 277); n= 2: number analyzed (Participants) | 2
  ALT; visit 18 (Week 277); n= 2 | 3.5 (3.54)
  ALT; withdrawal visit; n= 79: number analyzed (Participants) | 79
  ALT; withdrawal visit; n= 79 | 0.7 (10.17)
  ALT; follow up visit; n= 60: number analyzed (Participants) | 60
  ALT; follow up visit; n= 60 | 0.1 (8.43)
  AST; visit 1 (Screening); n= 82: number analyzed (Participants) | 82
  AST; visit 1 (Screening); n= 82 | 1.7 (7.97)
  AST; visit 2 (Week 13); n= 86: number analyzed (Participants) | 86
  AST; visit 2 (Week 13); n= 86 | 5.1 (31.13)
  AST; visit 3 (Week 26); n= 75: number analyzed (Participants) | 75
  AST; visit 3 (Week 26); n= 75 | 2.9 (23.95)
  AST; visit 4 (Week 39); n= 70: number analyzed (Participants) | 70
  AST; visit 4 (Week 39); n= 70 | 1.3 (8.23)
  AST; visit 5 (Week 52); n= 65: number analyzed (Participants) | 65
  AST; visit 5 (Week 52); n= 65 | 2.5 (6.01)
  AST; visit 6 (Week 69); n= 62: number analyzed (Participants) | 62
  AST; visit 6 (Week 69); n= 62 | 1.5 (7.55)
  AST; visit 7 (Week 86); n= 54: number analyzed (Participants) | 54
  AST; visit 7 (Week 86); n= 54 | 1.7 (8.20)
  AST; visit 8 (Week 104); n= 42: number analyzed (Participants) | 42
  AST; visit 8 (Week 104); n= 42 | 1.5 (7.94)
  AST; visit 9 (Week 121); n= 39: number analyzed (Participants) | 39
  AST; visit 9 (Week 121); n= 39 | 2.6 (7.99)
  AST; visit 10 (Week 138); n= 36: number analyzed (Participants) | 36
  AST; visit 10 (Week 138); n= 36 | 6.4 (17.36)
  AST; visit 11 (Week 156); n= 30: number analyzed (Participants) | 30
  AST; visit 11 (Week 156); n= 30 | 1.4 (7.38)
  AST; visit 12 (Week 173); n= 23: number analyzed (Participants) | 23
  AST; visit 12 (Week 173); n= 23 | 2.7 (4.71)
  AST; visit 13 (Week 190); n= 19: number analyzed (Participants) | 19
  AST; visit 13 (Week 190); n= 19 | 3.3 (5.21)
  AST; visit 14 (Week 208); n= 10: number analyzed (Participants) | 10
  AST; visit 14 (Week 208); n= 10 | 3.5 (6.42)
  AST; visit 15 (Week 225); n= 5: number analyzed (Participants) | 5
  AST; visit 15 (Week 225); n= 5 | 4.2 (2.95)
  AST; visit 16 (Week 242); n= 4: number analyzed (Participants) | 4
  AST; visit 16 (Week 242); n= 4 | 4.3 (4.72)
  AST; visit 17 (Week 260); n= 4: number analyzed (Participants) | 4
  AST; visit 17 (Week 260); n= 4 | 5.5 (3.11)
  AST; visit 18 (Week 277); n= 2: number analyzed (Participants) | 2
  AST; visit 18 (Week 277); n= 2 | 10.0 (9.90)
  AST; withdrawal visit; n= 78: number analyzed (Participants) | 78
  AST; withdrawal visit; n= 78 | 1.8 (7.87)
  AST; follow up visit; n= 60: number analyzed (Participants) | 60
  AST; follow up visit; n= 60 | 1.2 (6.99)
  Creatine kinase; Visit 1 (Screening); n= 82: number analyzed (Participants) | 82
  Creatine kinase; Visit 1 (Screening); n= 82 | 16.4 (132.76)
  Creatine kinase; Visit 2 (Week 13); n= 86: number analyzed (Participants) | 86
  Creatine kinase; Visit 2 (Week 13); n= 86 | 11.3 (78.18)
  Creatine kinase; Visit 3 (Week 26); n= 74: number analyzed (Participants) | 74
  Creatine kinase; Visit 3 (Week 26); n= 74 | 11.7 (59.78)
  Creatine kinase; Visit 4 (Week 39); n= 70: number analyzed (Participants) | 70
  Creatine kinase; Visit 4 (Week 39); n= 70 | 49.4 (397.67)
  Creatine kinase; Visit 5 (Week 52); n= 65: number analyzed (Participants) | 65
  Creatine kinase; Visit 5 (Week 52); n= 65 | 31.3 (136.41)
  Creatine kinase; Visit 6 (Week 69); n= 62: number analyzed (Participants) | 62
  Creatine kinase; Visit 6 (Week 69); n= 62 | 11.1 (55.13)
  Creatine kinase; Visit 7 (Week 86); n= 54: number analyzed (Participants) | 54
  Creatine kinase; Visit 7 (Week 86); n= 54 | 23.6 (92.64)
  Creatine kinase; Visit 8 (Week 104); n= 42: number analyzed (Participants) | 42
  Creatine kinase; Visit 8 (Week 104); n= 42 | 33.2 (110.99)
  Creatine kinase; Visit 9 (Week 121); n= 39: number analyzed (Participants) | 39
  Creatine kinase; Visit 9 (Week 121); n= 39 | 22.5 (77.04)
  Creatine kinase; Visit 10 (Week 138); n= 36: number analyzed (Participants) | 36
  Creatine kinase; Visit 10 (Week 138); n= 36 | 24.8 (83.80)
  Creatine kinase; Visit 11 (Week 156); n= 30: number analyzed (Participants) | 30
  Creatine kinase; Visit 11 (Week 156); n= 30 | 31.9 (86.68)
  Creatine kinase; Visit 12 (Week 173); n= 23: number analyzed (Participants) | 23
  Creatine kinase; Visit 12 (Week 173); n= 23 | 29.1 (97.10)
  Creatine kinase; Visit 13 (Week 190); n= 19: number analyzed (Participants) | 19
  Creatine kinase; Visit 13 (Week 190); n= 19 | 50.2 (125.12)
  Creatine kinase; Visit 14 (Week 208); n= 10: number analyzed (Participants) | 10
  Creatine kinase; Visit 14 (Week 208); n= 10 | -7.9 (101.39)
  Creatine kinase; Visit 15 (Week 225); n= 5: number analyzed (Participants) | 5
  Creatine kinase; Visit 15 (Week 225); n= 5 | 42.6 (99.09)
  Creatine kinase; Visit 16 (Week 242); n= 4: number analyzed (Participants) | 4
  Creatine kinase; Visit 16 (Week 242); n= 4 | 90.3 (127.49)
  Creatine kinase; Visit 17 (Week 260); n= 4: number analyzed (Participants) | 4
  Creatine kinase; Visit 17 (Week 260); n= 4 | 78.8 (110.78)
  Creatine kinase; Visit 18 (Week 277); n= 2: number analyzed (Participants) | 2
  Creatine kinase; Visit 18 (Week 277); n= 2 | -27.5 (102.53)
  Creatine kinase; withdrawal visit; n= 78: number analyzed (Participants) | 78
  Creatine kinase; withdrawal visit; n= 78 | 28.7 (139.96)
  Creatine kinase; follow up visit; n= 60: number analyzed (Participants) | 60
  Creatine kinase; follow up visit; n= 60 | 33.9 (128.19)
  LD; visit 1(Screening); n= 82: number analyzed (Participants) | 82
  LD; visit 1(Screening); n= 82 | 3.7 (23.16)
  LD; visit 2 (Week 13); n= 86: number analyzed (Participants) | 86
  LD; visit 2 (Week 13); n= 86 | 4.3 (32.66)
  LD; visit 3 (Week 26); n= 74: number analyzed (Participants) | 74
  LD; visit 3 (Week 26); n= 74 | 0.0 (27.88)
  LD; visit 4 (Week 39); n= 69: number analyzed (Participants) | 69
  LD; visit 4 (Week 39); n= 69 | 0.4 (28.51)
  LD; visit 5 (Week 52); n= 64: number analyzed (Participants) | 64
  LD; visit 5 (Week 52); n= 64 | 2.1 (28.01)
  LD; visit 6 (Week 69); n= 61: number analyzed (Participants) | 61
  LD; visit 6 (Week 69); n= 61 | -0.1 (25.98)
  LD; visit 7 (Week 86); n= 54: number analyzed (Participants) | 54
  LD; visit 7 (Week 86); n= 54 | 9.2 (30.42)
  LD; visit 8 (Week 104); n= 42 | 4.7 (29.37)
  LD; visit 9 (Week 121); n= 39: number analyzed (Participants) | 39
  LD; visit 9 (Week 121); n= 39 | 18.8 (53.56)
  LD; visit 10 (Week 138); n= 36: number analyzed (Participants) | 36
  LD; visit 10 (Week 138); n= 36 | 33.0 (131.87)
  LD; visit 11 (Week 156); n= 30: number analyzed (Participants) | 30
  LD; visit 11 (Week 156); n= 30 | 13.7 (33.18)
  LD; visit 12 (Week 173); n= 23: number analyzed (Participants) | 23
  LD; visit 12 (Week 173); n= 23 | 4.1 (31.91)
  LD; visit 13 (Week 190); n= 19: number analyzed (Participants) | 19
  LD; visit 13 (Week 190); n= 19 | 30.0 (58.17)
  LD; visit 14 (Week 208); n= 10: number analyzed (Participants) | 10
  LD; visit 14 (Week 208); n= 10 | 25.8 (42.76)
  LD; visit 15 (Week 225); n= 5: number analyzed (Participants) | 5
  LD; visit 15 (Week 225); n= 5 | 34.6 (25.93)
  LD; visit 16 (Week 242); n= 4: number analyzed (Participants) | 4
  LD; visit 16 (Week 242); n= 4 | 25.8 (15.97)
  LD; visit 17 (Week 260); n= 4: number analyzed (Participants) | 4
  LD; visit 17 (Week 260); n= 4 | 20.8 (25.86)
  LD; visit 18 (Week 277); n= 2: number analyzed (Participants) | 2
  LD; visit 18 (Week 277); n= 2 | 52.0 (60.81)
  LD; withdrawal visit; n= 78: number analyzed (Participants) | 78
  LD; withdrawal visit; n= 78 | 7.8 (31.17)
  LD; follow up visit; n= 60: number analyzed (Participants) | 60
  LD; follow up visit; n= 60 | 5.6 (36.94)

17. Primary Outcome: Change From Baseline in Direct Bilirubin, Total Bilirubin and Creatinine
Description: Blood samples were collected from participants for evaluation of change from Baseline in clinical chemistry parameters including direct bilirubin, total bilirubin and creatinine. Baseline was defined by and taken directly from the Baseline assessments in the parent study NCT01336621. Change from Baseline was defined as post-Baseline value minus Baseline value. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Time Frame: Baseline and up to 5.8 years
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Micromole per liter (µmol/L)
Arm/Group | Retigabine IR
Number analyzed (Participants) | 98
Micromole per liter (µmol/L)
  Direct bilirubin; visit 1 (Screening); n= 83: number analyzed (Participants) | 83
  Direct bilirubin; visit 1 (Screening); n= 83 | 0.1 (0.95)
  Direct bilirubin; visit 2 (Week 13); n= 87: number analyzed (Participants) | 87
  Direct bilirubin; visit 2 (Week 13); n= 87 | -0.1 (0.96)
  Direct bilirubin; visit 3 (Week 26); n= 75: number analyzed (Participants) | 75
  Direct bilirubin; visit 3 (Week 26); n= 75 | -0.2 (0.94)
  Direct bilirubin; visit 4 (Week 39); n= 69: number analyzed (Participants) | 69
  Direct bilirubin; visit 4 (Week 39); n= 69 | -0.1 (0.91)
  Direct bilirubin; visit 5 (Week 52); n= 65: number analyzed (Participants) | 65
  Direct bilirubin; visit 5 (Week 52); n= 65 | 0.0 (0.95)
  Direct bilirubin; visit 6 (Week 69); n= 62: number analyzed (Participants) | 62
  Direct bilirubin; visit 6 (Week 69); n= 62 | -0.0 (0.97)
  Direct bilirubin; visit 7 (Week 86); n= 54: number analyzed (Participants) | 54
  Direct bilirubin; visit 7 (Week 86); n= 54 | -0.2 (1.17)
  Direct bilirubin; visit 8 (Week 104); n= 42: number analyzed (Participants) | 42
  Direct bilirubin; visit 8 (Week 104); n= 42 | -0.0 (0.91)
  Direct bilirubin; visit 9 (Week 121); n= 39: number analyzed (Participants) | 39
  Direct bilirubin; visit 9 (Week 121); n= 39 | -0.2 (0.87)
  Direct bilirubin; visit 10 (Week 138); n= 36: number analyzed (Participants) | 36
  Direct bilirubin; visit 10 (Week 138); n= 36 | -0.1 (1.27)
  Direct bilirubin; visit 11 (Week 156); n= 30: number analyzed (Participants) | 30
  Direct bilirubin; visit 11 (Week 156); n= 30 | 0.0 (0.72)
  Direct bilirubin; visit 12 (Week 173); n= 23: number analyzed (Participants) | 23
  Direct bilirubin; visit 12 (Week 173); n= 23 | -0.1 (0.73)
  Direct bilirubin; visit 13 (Week 190); n= 19: number analyzed (Participants) | 19
  Direct bilirubin; visit 13 (Week 190); n= 19 | 0.1 (0.91)
  Direct bilirubin; visit 14 (Week 208); n= 10: number analyzed (Participants) | 10
  Direct bilirubin; visit 14 (Week 208); n= 10 | 0.0 (0.67)
  Direct bilirubin; visit 15 (Week 225); n= 5: number analyzed (Participants) | 5
  Direct bilirubin; visit 15 (Week 225); n= 5 | -0.2 (0.84)
  Direct bilirubin; visit 16 (Week 242); n= 4: number analyzed (Participants) | 4
  Direct bilirubin; visit 16 (Week 242); n= 4 | -0.5 (1.00)
  Direct bilirubin; visit 17 (Week 260); n= 4: number analyzed (Participants) | 4
  Direct bilirubin; visit 17 (Week 260); n= 4 | -0.5 (1.29)
  Direct bilirubin; visit 18 (Week 277); n= 2: number analyzed (Participants) | 2
  Direct bilirubin; visit 18 (Week 277); n= 2 | 0.5 (2.12)
  Direct bilirubin; withdrawal visit; n= 79: number analyzed (Participants) | 79
  Direct bilirubin; withdrawal visit; n= 79 | 0.0 (1.15)
  Direct bilirubin; follow up visit; n= 60: number analyzed (Participants) | 60
  Direct bilirubin; follow up visit; n= 60 | -0.2 (0.98)
  Total bilirubin; visit 1 (Screening); n= 83: number analyzed (Participants) | 83
  Total bilirubin; visit 1 (Screening); n= 83 | 2.5 (3.78)
  Total bilirubin; visit 2 (Week 13); n= 87: number analyzed (Participants) | 87
  Total bilirubin; visit 2 (Week 13); n= 87 | 1.8 (4.28)
  Total bilirubin; visit 3 (Week 26); n= 76: number analyzed (Participants) | 76
  Total bilirubin; visit 3 (Week 26); n= 76 | 1.8 (3.78)
  Total bilirubin; visit 4 (Week 39); n= 70: number analyzed (Participants) | 70
  Total bilirubin; visit 4 (Week 39); n= 70 | 2.1 (4.46)
  Total bilirubin; visit 5 (Week 52); n= 65: number analyzed (Participants) | 65
  Total bilirubin; visit 5 (Week 52); n= 65 | 2.6 (4.26)
  Total bilirubin; visit 6 (Week 69); n= 62: number analyzed (Participants) | 62
  Total bilirubin; visit 6 (Week 69); n= 62 | 1.8 (4.21)
  Total bilirubin; visit 7 (Week 86); n= 54: number analyzed (Participants) | 54
  Total bilirubin; visit 7 (Week 86); n= 54 | 1.4 (4.41)
  Total bilirubin; visit 8 (Week 104); n= 42: number analyzed (Participants) | 42
  Total bilirubin; visit 8 (Week 104); n= 42 | 1.8 (3.28)
  Total bilirubin; visit 9 (Week 121); n= 39: number analyzed (Participants) | 39
  Total bilirubin; visit 9 (Week 121); n= 39 | 1.1 (3.59)
  Total bilirubin; visit 10 (Week 138); n= 36: number analyzed (Participants) | 36
  Total bilirubin; visit 10 (Week 138); n= 36 | 1.6 (6.50)
  Total bilirubin; visit 11 (Week 156); n= 30: number analyzed (Participants) | 30
  Total bilirubin; visit 11 (Week 156); n= 30 | 0.5 (2.99)
  Total bilirubin; visit 12 (Week 173); n= 23: number analyzed (Participants) | 23
  Total bilirubin; visit 12 (Week 173); n= 23 | 0.6 (2.81)
  Total bilirubin; visit 13 (Week 190); n= 19: number analyzed (Participants) | 19
  Total bilirubin; visit 13 (Week 190); n= 19 | 0.2 (4.26)
  Total bilirubin; visit 14 (Week 208); n= 10: number analyzed (Participants) | 10
  Total bilirubin; visit 14 (Week 208); n= 10 | 0.3 (3.27)
  Total bilirubin; visit 15 (Week 225); n= 5: number analyzed (Participants) | 5
  Total bilirubin; visit 15 (Week 225); n= 5 | 0.8 (2.17)
  Total bilirubin; visit 16 (Week 242); n= 4: number analyzed (Participants) | 4
  Total bilirubin; visit 16 (Week 242); n= 4 | 1.3 (1.89)
  Total bilirubin; visit 17 (Week 260); n= 4: number analyzed (Participants) | 4
  Total bilirubin; visit 17 (Week 260); n= 4 | -0.3 (2.63)
  Total bilirubin; visit 18 (Week 277); n= 2: number analyzed (Participants) | 2
  Total bilirubin; visit 18 (Week 277); n= 2 | 1.5 (0.71)
  Total bilirubin; withdrawal visit; n= 79: number analyzed (Participants) | 79
  Total bilirubin; withdrawal visit; n= 79 | 1.2 (3.75)
  Total bilirubin; follow up visit; n= 60: number analyzed (Participants) | 60
  Total bilirubin; follow up visit; n= 60 | -0.8 (3.97)
  Creatinine; visit 1 (Screening); n= 82: number analyzed (Participants) | 82
  Creatinine; visit 1 (Screening); n= 82 | 3.68 (9.813)
  Creatinine; visit 2 (Week 13); n= 86: number analyzed (Participants) | 86
  Creatinine; visit 2 (Week 13); n= 86 | 0.42 (8.033)
  Creatinine; visit 3 (Week 26); n= 74: number analyzed (Participants) | 74
  Creatinine; visit 3 (Week 26); n= 74 | 0.65 (8.879)
  Creatinine; visit 4 (Week 39); n= 70: number analyzed (Participants) | 70
  Creatinine; visit 4 (Week 39); n= 70 | 1.82 (9.716)
  Creatinine; visit 5 (Week 52); n= 65: number analyzed (Participants) | 65
  Creatinine; visit 5 (Week 52); n= 65 | 1.40 (9.394)
  Creatinine; visit 6 (Week 69); n= 62: number analyzed (Participants) | 62
  Creatinine; visit 6 (Week 69); n= 62 | 1.25 (8.980)
  Creatinine; visit 7 (Week 86); n= 54: number analyzed (Participants) | 54
  Creatinine; visit 7 (Week 86); n= 54 | 0.55 (9.053)
  Creatinine; visit 8 (Week 104); n= 42: number analyzed (Participants) | 42
  Creatinine; visit 8 (Week 104); n= 42 | 4.78 (8.921)
  Creatinine; visit 9 (Week 121); n= 39: number analyzed (Participants) | 39
  Creatinine; visit 9 (Week 121); n= 39 | 3.67 (9.581)
  Creatinine; visit 10 (Week 138); n= 36: number analyzed (Participants) | 36
  Creatinine; visit 10 (Week 138); n= 36 | 2.10 (11.317)
  Creatinine; visit 11 (Week 156); n= 30: number analyzed (Participants) | 30
  Creatinine; visit 11 (Week 156); n= 30 | 5.33 (11.211)
  Creatinine; visit 12 (Week 173); n= 23: number analyzed (Participants) | 23
  Creatinine; visit 12 (Week 173); n= 23 | -0.93 (10.097)
  Creatinine; visit 13 (Week 190); n= 19: number analyzed (Participants) | 19
  Creatinine; visit 13 (Week 190); n= 19 | 1.67 (11.314)
  Creatinine; visit 14 (Week 208); n= 10: number analyzed (Participants) | 10
  Creatinine; visit 14 (Week 208); n= 10 | -1.74 (13.636)
  Creatinine; visit 15 (Week 225); n= 5: number analyzed (Participants) | 5
  Creatinine; visit 15 (Week 225); n= 5 | 2.08 (6.680)
  Creatinine; visit 16 (Week 242); n= 4: number analyzed (Participants) | 4
  Creatinine; visit 16 (Week 242); n= 4 | 5.80 (8.844)
  Creatinine; visit 17 (Week 260); n= 4: number analyzed (Participants) | 4
  Creatinine; visit 17 (Week 260); n= 4 | 9.23 (14.076)
  Creatinine; visit 18 (Week 277); n= 2: number analyzed (Participants) | 2
  Creatinine; visit 18 (Week 277); n= 2 | 3.45 (8.697)
  Creatinine; withdrawal visit; n= 78: number analyzed (Participants) | 78
  Creatinine; withdrawal visit; n= 78 | 0.88 (8.920)
  Creatinine; follow up visit; n= 60: number analyzed (Participants) | 60
  Creatinine; follow up visit; n= 60 | 0.16 (9.873)

18. Primary Outcome: Change From Baseline in BUN/Creatinine Ratio
Description: Blood samples were collected from participants for evaluation of change from Baseline in clinical chemistry parameters including BUN/creatinine ratio. Baseline was defined by and taken directly from the Baseline assessments in the parent study NCT01336621. Change from Baseline was defined as post-Baseline value minus Baseline value. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Time Frame: Baseline and up to 5.8 years
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Ratio of BUN to creatinine
Arm/Group | Retigabine IR
Number analyzed (Participants) | 98
Ratio of BUN to creatinine
  Visit 1 (Screening); n= 82: number analyzed (Participants) | 82
  Visit 1 (Screening); n= 82 | 0.3 (20.71)
  Visit 2 (Week 13); n= 86: number analyzed (Participants) | 86
  Visit 2 (Week 13); n= 86 | 3.8 (23.49)
  Visit 3 (Week 26); n= 74: number analyzed (Participants) | 74
  Visit 3 (Week 26); n= 74 | 2.7 (20.38)
  Visit 4 (Week 39); n= 70: number analyzed (Participants) | 70
  Visit 4 (Week 39); n= 70 | 1.0 (23.43)
  Visit 5 (Week 52); n= 65: number analyzed (Participants) | 65
  Visit 5 (Week 52); n= 65 | 1.9 (27.30)
  Visit 6 (Week 69); n= 62: number analyzed (Participants) | 62
  Visit 6 (Week 69); n= 62 | -0.0 (22.69)
  Visit 7 (Week 86); n= 54: number analyzed (Participants) | 54
  Visit 7 (Week 86); n= 54 | 2.5 (24.05)
  Visit 8 (Week 104); n= 42: number analyzed (Participants) | 42
  Visit 8 (Week 104); n= 42 | -2.5 (24.45)
  Visit 9 (Week 121); n= 39: number analyzed (Participants) | 39
  Visit 9 (Week 121); n= 39 | 0.6 (24.67)
  Visit 10 (Week 138); n= 36: number analyzed (Participants) | 36
  Visit 10 (Week 138); n= 36 | 0.2 (27.01)
  Visit 11 (Week 156); n= 30: number analyzed (Participants) | 30
  Visit 11 (Week 156); n= 30 | -6.2 (24.68)
  Visit 12 (Week 173); n= 23: number analyzed (Participants) | 23
  Visit 12 (Week 173); n= 23 | -5.7 (22.82)
  Visit 13 (Week 190); n= 19: number analyzed (Participants) | 19
  Visit 13 (Week 190); n= 19 | 1.1 (22.19)
  Visit 14 (Week 208); n= 10: number analyzed (Participants) | 10
  Visit 14 (Week 208); n= 10 | -0.8 (23.37)
  Visit 15 (Week 225); n= 5: number analyzed (Participants) | 5
  Visit 15 (Week 225); n= 5 | -8.8 (20.22)
  Visit 16 (Week 242); n= 4: number analyzed (Participants) | 4
  Visit 16 (Week 242); n= 4 | 4.0 (18.49)
  Visit 17 (Week 260); n= 4: number analyzed (Participants) | 4
  Visit 17 (Week 260); n= 4 | 2.0 (32.81)
  Visit 18 (Week 277); n= 2: number analyzed (Participants) | 2
  Visit 18 (Week 277); n= 2 | 3.0 (11.31)
  Withdrawal visit; n= 78: number analyzed (Participants) | 78
  Withdrawal visit; n= 78 | 4.2 (23.96)
  Follow up visit; n= 60: number analyzed (Participants) | 60
  Follow up visit; n= 60 | 0.4 (22.68)

19. Primary Outcome: Change From Baseline in Calcium, Chloride, CO2, Glucose, Potassium, Magnesium, Sodium and BUN
Description: Blood samples were collected from participants for evaluation of change from Baseline in clinical chemistry parameters including calcium, chloride, CO2, glucose, potassium, magnesium, sodium and BUN. Baseline was defined by and taken directly from the Baseline assessments in the parent study NCT01336621. Change from Baseline was defined as post-Baseline value minus Baseline value. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Time Frame: Baseline and up to 5.8 years
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Millimoles per liter (mmol/L)
Arm/Group | Retigabine IR
Number analyzed (Participants) | 98
Millimoles per liter (mmol/L)
  Calcium; visit 1 (Screening); n= 82: number analyzed (Participants) | 82
  Calcium; visit 1 (Screening); n= 82 | -0.028 (0.0940)
  Calcium; visit 2 (Week 13); n= 86: number analyzed (Participants) | 86
  Calcium; visit 2 (Week 13); n= 86 | -0.011 (0.1067)
  Calcium; visit 3 (Week 26); n= 74: number analyzed (Participants) | 74
  Calcium; visit 3 (Week 26); n= 74 | -0.026 (0.1061)
  Calcium; visit 4 (Week 39); n= 69: number analyzed (Participants) | 69
  Calcium; visit 4 (Week 39); n= 69 | -0.025 (0.1024)
  Calcium; visit 5 (Week 52); n= 64: number analyzed (Participants) | 64
  Calcium; visit 5 (Week 52); n= 64 | -0.026 (0.1100)
  Calcium; visit 6 (Week 69); n= 61: number analyzed (Participants) | 61
  Calcium; visit 6 (Week 69); n= 61 | -0.019 (0.0942)
  Calcium; visit 7 (Week 86); n= 54: number analyzed (Participants) | 54
  Calcium; visit 7 (Week 86); n= 54 | -0.016 (0.0911)
  Calcium; visit 8 (Week 104); n= 42: number analyzed (Participants) | 42
  Calcium; visit 8 (Week 104); n= 42 | -0.008 (0.0975)
  Calcium; visit 9 (Week 121); n= 39: number analyzed (Participants) | 39
  Calcium; visit 9 (Week 121); n= 39 | -0.024 (0.1096)
  Calcium; visit 10 (Week 138); n= 36: number analyzed (Participants) | 36
  Calcium; visit 10 (Week 138); n= 36 | -0.038 (0.1335)
  Calcium; visit 11 (Week 156); n= 30: number analyzed (Participants) | 30
  Calcium; visit 11 (Week 156); n= 30 | -0.053 (0.1181)
  Calcium; visit 12 (Week 173); n= 23: number analyzed (Participants) | 23
  Calcium; visit 12 (Week 173); n= 23 | -0.059 (0.1031)
  Calcium; visit 13 (Week 190); n= 19: number analyzed (Participants) | 19
  Calcium; visit 13 (Week 190); n= 19 | -0.074 (0.1000)
  Calcium; visit 14 (Week 208); n= 10: number analyzed (Participants) | 10
  Calcium; visit 14 (Week 208); n= 10 | -0.094 (0.0950)
  Calcium; visit 15 (Week 225); n= 5: number analyzed (Participants) | 5
  Calcium; visit 15 (Week 225); n= 5 | -0.108 (0.0858)
  Calcium; visit 16 (Week 242); n= 4: number analyzed (Participants) | 4
  Calcium; visit 16 (Week 242); n= 4 | -0.093 (0.0877)
  Calcium; visit 17 (Week 260); n= 4: number analyzed (Participants) | 4
  Calcium; visit 17 (Week 260); n= 4 | -0.073 (0.0670)
  Calcium; visit 18 (Week 277); n= 2: number analyzed (Participants) | 2
  Calcium; visit 18 (Week 277); n= 2 | -0.125 (0.02122)
  Calcium; withdrawal visit; n= 78: number analyzed (Participants) | 78
  Calcium; withdrawal visit; n= 78 | -0.033 (0.1148)
  Calcium; follow up visit; n= 60: number analyzed (Participants) | 60
  Calcium; follow up visit; n= 60 | -0.050 (0.1059)
  Chloride; visit 1 (Screening); n= 83: number analyzed (Participants) | 83
  Chloride; visit 1 (Screening); n= 83 | 0.5 (2.88)
  Chloride; visit 2 (Week 13); n= 87: number analyzed (Participants) | 87
  Chloride; visit 2 (Week 13); n= 87 | 0.4 (2.73)
  Chloride; visit 3 (Week 26); n=75: number analyzed (Participants) | 75
  Chloride; visit 3 (Week 26); n=75 | 0.1 (2.79)
  Chloride; visit 4 (Week 39); n= 70: number analyzed (Participants) | 70
  Chloride; visit 4 (Week 39); n= 70 | 1.5 (2.80)
  Chloride; visit 5 (Week 52); n= 65: number analyzed (Participants) | 65
  Chloride; visit 5 (Week 52); n= 65 | 1.2 (3.58)
  Chloride; visit 6 (Week 69); n= 62: number analyzed (Participants) | 62
  Chloride; visit 6 (Week 69); n= 62 | 0.4 (2.68)
  Chloride; visit 7 (Week 86); n= 54: number analyzed (Participants) | 54
  Chloride; visit 7 (Week 86); n= 54 | 1.5 (3.34)
  Chloride; visit 8 (Week 104); n= 42: number analyzed (Participants) | 42
  Chloride; visit 8 (Week 104); n= 42 | 1.3 (2.83)
  Chloride; visit 9 (Week 121); n= 39: number analyzed (Participants) | 39
  Chloride; visit 9 (Week 121); n= 39 | 1.4 (3.28)
  Chloride; visit 10 (Week 138); n= 36: number analyzed (Participants) | 36
  Chloride; visit 10 (Week 138); n= 36 | 1.2 (3.35)
  Chloride; visit 11 (Week 156); n= 30: number analyzed (Participants) | 30
  Chloride; visit 11 (Week 156); n= 30 | 2.0 (2.99)
  Chloride; visit 12 (Week 173); n= 23: number analyzed (Participants) | 23
  Chloride; visit 12 (Week 173); n= 23 | 1.6 (2.74)
  Chloride; visit 13 (Week 190); n= 19: number analyzed (Participants) | 19
  Chloride; visit 13 (Week 190); n= 19 | 2.4 (2.09)
  Chloride; visit 14 (Week 208); n= 10: number analyzed (Participants) | 10
  Chloride; visit 14 (Week 208); n= 10 | 1.2 (2.49)
  Chloride; visit 15 (Week 225); n= 5: number analyzed (Participants) | 5
  Chloride; visit 15 (Week 225); n= 5 | 1.2 (3.11)
  Chloride; visit 16 (Week 242); n= 4: number analyzed (Participants) | 4
  Chloride; visit 16 (Week 242); n= 4 | 2.0 (2.00)
  Chloride; visit 17 (Week 260); n= 4: number analyzed (Participants) | 4
  Chloride; visit 17 (Week 260); n= 4 | 3.5 (3.11)
  Chloride; visit 18 (Week 277); n= 2: number analyzed (Participants) | 2
  Chloride; visit 18 (Week 277); n= 2 | -0.5 (0.71)
  Chloride; withdrawal visit; n= 79: number analyzed (Participants) | 79
  Chloride; withdrawal visit; n= 79 | 0.6 (2.89)
  Chloride; follow up visit; n= 60: number analyzed (Participants) | 60
  Chloride; follow up visit; n= 60 | -0.0 (2.79)
  CO2; visit 1 (Screening); n= 82: number analyzed (Participants) | 82
  CO2; visit 1 (Screening); n= 82 | -0.2 (3.07)
  CO2; visit 2 (Week 13); n= 86: number analyzed (Participants) | 86
  CO2; visit 2 (Week 13); n= 86 | 0.3 (2.42)
  CO2; visit 3 (Week 26); n= 74: number analyzed (Participants) | 74
  CO2; visit 3 (Week 26); n= 74 | 0.5 (2.82)
  CO2; visit 4 (Week 39); n= 69: number analyzed (Participants) | 69
  CO2; visit 4 (Week 39); n= 69 | -0.2 (3.03)
  CO2; visit 5 (Week 52); n= 64: number analyzed (Participants) | 64
  CO2; visit 5 (Week 52); n= 64 | -0.2 (2.88)
  CO2; visit 6 (Week 69); n= 61: number analyzed (Participants) | 61
  CO2; visit 6 (Week 69); n= 61 | -0.5 (2.99)
  CO2; visit 7 (Week 86); n= 54: number analyzed (Participants) | 54
  CO2; visit 7 (Week 86); n= 54 | -0.6 (2.71)
  CO2; visit 8 (Week 104); n= 42: number analyzed (Participants) | 42
  CO2; visit 8 (Week 104); n= 42 | -0.6 (2.64)
  CO2; visit 9 (Week 121); n= 39: number analyzed (Participants) | 39
  CO2; visit 9 (Week 121); n= 39 | -1.0 (3.02)
  CO2; visit 10 (Week 138); n= 36: number analyzed (Participants) | 36
  CO2; visit 10 (Week 138); n= 36 | -0.9 (3.42)
  CO2; visit 11 (Week 156); n= 30: number analyzed (Participants) | 30
  CO2; visit 11 (Week 156); n= 30 | -1.0 (2.48)
  CO2; visit 12 (Week 173); n= 23: number analyzed (Participants) | 23
  CO2; visit 12 (Week 173); n= 23 | -0.9 (2.80)
  CO2; visit 13 (Week 190); n= 19: number analyzed (Participants) | 19
  CO2; visit 13 (Week 190); n= 19 | -1.5 (3.39)
  CO2; visit 14 (Week 208); n= 10: number analyzed (Participants) | 10
  CO2; visit 14 (Week 208); n= 10 | -3.6 (4.53)
  CO2; visit 15 (Week 225); n= 5: number analyzed (Participants) | 5
  CO2; visit 15 (Week 225); n= 5 | -2.4 (1.82)
  CO2; visit 16 (Week 242); n= 4: number analyzed (Participants) | 4
  CO2; visit 16 (Week 242); n= 4 | -1.0 (1.41)
  CO2; visit 17 (Week 260); n= 4: number analyzed (Participants) | 4
  CO2; visit 17 (Week 260); n= 4 | -0.5 (0.58)
  CO2; visit 18 (Week 277); n= 2: number analyzed (Participants) | 2
  CO2; visit 18 (Week 277); n= 2 | -0.5 (0.71)
  CO2; withdrawal visit; n= 78: number analyzed (Participants) | 78
  CO2; withdrawal visit; n= 78 | -0.0 (2.33)
  CO2; follow up visit; n= 60: number analyzed (Participants) | 60
  CO2; follow up visit; n= 60 | -0.8 (2.92)
  Glucose; visit 1 (Screening); n= 83: number analyzed (Participants) | 83
  Glucose; visit 1 (Screening); n= 83 | 0.20 (1.303)
  Glucose; visit 2 (Week 13); n= 87: number analyzed (Participants) | 87
  Glucose; visit 2 (Week 13); n= 87 | 0.16 (0.933)
  Glucose; visit 3 (Week 26); n= 75: number analyzed (Participants) | 75
  Glucose; visit 3 (Week 26); n= 75 | 0.17 (0.765)
  Glucose; visit 4 (Week 39); n= 70: number analyzed (Participants) | 70
  Glucose; visit 4 (Week 39); n= 70 | 0.40 (1.259)
  Glucose; visit 5 (Week 52); n= 65: number analyzed (Participants) | 65
  Glucose; visit 5 (Week 52); n= 65 | 0.23 (0.814)
  Glucose; visit 6 (Week 69); n= 62: number analyzed (Participants) | 62
  Glucose; visit 6 (Week 69); n= 62 | 0.25 (1.103)
  Glucose; visit 7 (Week 86); n= 54: number analyzed (Participants) | 54
  Glucose; visit 7 (Week 86); n= 54 | 0.21 (0.985)
  Glucose; visit 8 (Week 104); n= 42: number analyzed (Participants) | 42
  Glucose; visit 8 (Week 104); n= 42 | 0.21 (0.679)
  Glucose; visit 9 (Week 121); n= 39: number analyzed (Participants) | 39
  Glucose; visit 9 (Week 121); n= 39 | 0.31 (1.073)
  Glucose; visit 10 (Week 138); n= 36: number analyzed (Participants) | 36
  Glucose; visit 10 (Week 138); n= 36 | 0.30 (1.007)
  Glucose; visit 11 (Week 156); n= 30: number analyzed (Participants) | 30
  Glucose; visit 11 (Week 156); n= 30 | 0.10 (0.511)
  Glucose; visit 12 (Week 173); n= 23: number analyzed (Participants) | 23
  Glucose; visit 12 (Week 173); n= 23 | -0.03 (0.820)
  Glucose; visit 13 (Week 190); n= 19: number analyzed (Participants) | 19
  Glucose; visit 13 (Week 190); n= 19 | 0.21 (1.446)
  Glucose; visit 14 (Week 208); n= 10: number analyzed (Participants) | 10
  Glucose; visit 14 (Week 208); n= 10 | 0.15 (0.412)
  Glucose; visit 15 (Week 225); n= 5: number analyzed (Participants) | 5
  Glucose; visit 15 (Week 225); n= 5 | 0.38 (0.981)
  Glucose; visit 16 (Week 242); n= 4: number analyzed (Participants) | 4
  Glucose; visit 16 (Week 242); n= 4 | 1.95 (3.313)
  Glucose; visit 17 (Week 260); n= 4: number analyzed (Participants) | 4
  Glucose; visit 17 (Week 260); n= 4 | -0.10 (0.648)
  Glucose; visit 18 (Week 277); n= 2: number analyzed (Participants) | 2
  Glucose; visit 18 (Week 277); n= 2 | -0.30 (0.141)
  Glucose; withdrawal visit; n= 79: number analyzed (Participants) | 79
  Glucose; withdrawal visit; n= 79 | 0.14 (1.035)
  Glucose; follow up visit; n= 60: number analyzed (Participants) | 60
  Glucose; follow up visit; n= 60 | 0.39 (1.162)
  Potassium; visit 1 (Screening); n= 82: number analyzed (Participants) | 82
  Potassium; visit 1 (Screening); n= 82 | -0.04 (0.467)
  Potassium; visit 2 (Week 13); n= 86: number analyzed (Participants) | 86
  Potassium; visit 2 (Week 13); n= 86 | -0.07 (0.403)
  Potassium; visit 3 (Week 26); n= 74: number analyzed (Participants) | 74
  Potassium; visit 3 (Week 26); n= 74 | -0.09 (0.453)
  Potassium; visit 4 (Week 39); n= 69: number analyzed (Participants) | 69
  Potassium; visit 4 (Week 39); n= 69 | -0.11 (0.432)
  Potassium; visit 5 (Week 52); n= 64: number analyzed (Participants) | 64
  Potassium; visit 5 (Week 52); n= 64 | -0.13 (0.430)
  Potassium; visit 6 (Week 69); n= 61: number analyzed (Participants) | 61
  Potassium; visit 6 (Week 69); n= 61 | -0.21 (0.420)
  Potassium; visit 7 (Week 86); n= 54: number analyzed (Participants) | 54
  Potassium; visit 7 (Week 86); n= 54 | -0.13 (0.411)
  Potassium; visit 8 (Week 104); n= 42: number analyzed (Participants) | 42
  Potassium; visit 8 (Week 104); n= 42 | -0.05 (0.433)
  Potassium; visit 9 (Week 121); n= 39: number analyzed (Participants) | 39
  Potassium; visit 9 (Week 121); n= 39 | -0.09 (0.376)
  Potassium; visit 10 (Week 138); n= 36: number analyzed (Participants) | 36
  Potassium; visit 10 (Week 138); n= 36 | -0.07 (0.388)
  Potassium; visit 11 (Week 156); n= 30: number analyzed (Participants) | 30
  Potassium; visit 11 (Week 156); n= 30 | -0.16 (0.390)
  Potassium; visit 12 (Week 173); n= 23: number analyzed (Participants) | 23
  Potassium; visit 12 (Week 173); n= 23 | -0.13 (0.411)
  Potassium; visit 13 (Week 190); n= 19: number analyzed (Participants) | 19
  Potassium; visit 13 (Week 190); n= 19 | -0.02 (0.351)
  Potassium; visit 14 (Week 208); n= 10: number analyzed (Participants) | 10
  Potassium; visit 14 (Week 208); n= 10 | -0.16 (0.430)
  Potassium; visit 15 (Week 225); n= 5: number analyzed (Participants) | 5
  Potassium; visit 15 (Week 225); n= 5 | 0.14 (0.321)
  Potassium; visit 16 (Week 242); n= 4: number analyzed (Participants) | 4
  Potassium; visit 16 (Week 242); n= 4 | 0.30 (0.294)
  Potassium; visit 17 (Week 260); n= 4: number analyzed (Participants) | 4
  Potassium; visit 17 (Week 260); n= 4 | 0.25 (0.351)
  Potassium; visit 18 (Week 277); n= 2: number analyzed (Participants) | 2
  Potassium; visit 18 (Week 277); n= 2 | 0.10 (0.424)
  Potassium; withdrawal visit; n= 78: number analyzed (Participants) | 78
  Potassium; withdrawal visit; n= 78 | -0.04 (0.367)
  Potassium; follow up visit; n= 60: number analyzed (Participants) | 60
  Potassium; follow up visit; n= 60 | -0.20 (0.478)
  Magnesium; visit 1 (Screening); n= 83: number analyzed (Participants) | 83
  Magnesium; visit 1 (Screening); n= 83 | -0.017 (0.0576)
  Magnesium; visit 2 (Week 13); n= 87: number analyzed (Participants) | 87
  Magnesium; visit 2 (Week 13); n= 87 | -0.012 (0.0558)
  Magnesium; visit 3 (Week 26); n= 75: number analyzed (Participants) | 75
  Magnesium; visit 3 (Week 26); n= 75 | -0.007 (0.0619)
  Magnesium; visit 4 (Week 39); n= 70: number analyzed (Participants) | 70
  Magnesium; visit 4 (Week 39); n= 70 | -0.004 (0.0580)
  Magnesium; visit 5 (Week 52); n= 65: number analyzed (Participants) | 65
  Magnesium; visit 5 (Week 52); n= 65 | -0.008 (0.0625)
  Magnesium; visit 6 (Week 69); n= 62: number analyzed (Participants) | 62
  Magnesium; visit 6 (Week 69); n= 62 | -0.012 (0.0599)
  Magnesium; visit 7 (Week 86); n= 54: number analyzed (Participants) | 54
  Magnesium; visit 7 (Week 86); n= 54 | -0.018 (0.0627)
  Magnesium; visit 8 (Week 104); n= 42: number analyzed (Participants) | 42
  Magnesium; visit 8 (Week 104); n= 42 | 0.007 (0.0632)
  Magnesium; visit 9 (Week 121); n= 39: number analyzed (Participants) | 39
  Magnesium; visit 9 (Week 121); n= 39 | -0.011 (0.0763)
  Magnesium; visit 10 (Week 138); n= 36: number analyzed (Participants) | 36
  Magnesium; visit 10 (Week 138); n= 36 | -0.007 (0.0543)
  Magnesium; visit 11 (Week 156); n= 30: number analyzed (Participants) | 30
  Magnesium; visit 11 (Week 156); n= 30 | 0.005 (0.0651)
  Magnesium; visit 12 (Week 173); n= 23: number analyzed (Participants) | 23
  Magnesium; visit 12 (Week 173); n= 23 | -0.003 (0.0688)
  Magnesium; visit 13 (Week 190); n= 19: number analyzed (Participants) | 19
  Magnesium; visit 13 (Week 190); n= 19 | -0.000 (0.0627)
  Magnesium; visit 14 (Week 208); n= 10: number analyzed (Participants) | 10
  Magnesium; visit 14 (Week 208); n= 10 | -0.013 (0.0579)
  Magnesium; visit 15 (Week 225); n= 5: number analyzed (Participants) | 5
  Magnesium; visit 15 (Week 225); n= 5 | 0.000 (0.0474)
  Magnesium; visit 16 (Week 242); n= 4: number analyzed (Participants) | 4
  Magnesium; visit 16 (Week 242); n= 4 | -0.008 (0.1075)
  Magnesium; visit 17 (Week 260); n= 4: number analyzed (Participants) | 4
  Magnesium; visit 17 (Week 260); n= 4 | 0.053 (0.1258)
  Magnesium; visit 18 (Week 277); n= 2: number analyzed (Participants) | 2
  Magnesium; visit 18 (Week 277); n= 2 | 0.070 (0.0424)
  Magnesium; withdrawal visit; n= 79: number analyzed (Participants) | 79
  Magnesium; withdrawal visit; n= 79 | -0.003 (0.0763)
  Magnesium; follow up visit; n= 60: number analyzed (Participants) | 60
  Magnesium; follow up visit; n= 60 | -0.007 (0.0727)
  Sodium; visit 1 (Screening); n= 83: number analyzed (Participants) | 83
  Sodium; visit 1 (Screening); n= 83 | 0.2 (2.88)
  Sodium; visit 2 (Week 13); n= 80: number analyzed (Participants) | 80
  Sodium; visit 2 (Week 13); n= 80 | 0.2 (2.83)
  Sodium; visit 3 (Week 26); n= 69: number analyzed (Participants) | 69
  Sodium; visit 3 (Week 26); n= 69 | -0.2 (2.79)
  Sodium; visit 4 (Week 39); n= 64: number analyzed (Participants) | 64
  Sodium; visit 4 (Week 39); n= 64 | 0.7 (2.37)
  Sodium; visit 5 (Week 52); n= 59: number analyzed (Participants) | 59
  Sodium; visit 5 (Week 52); n= 59 | 0.5 (3.35)
  Sodium; visit 6 (Week 69); n= 58: number analyzed (Participants) | 58
  Sodium; visit 6 (Week 69); n= 58 | -0.2 (2.34)
  Sodium; visit 7 (Week 86); n= 51: number analyzed (Participants) | 51
  Sodium; visit 7 (Week 86); n= 51 | 0.6 (3.03)
  Sodium; visit 8 (Week 104); n= 39: number analyzed (Participants) | 39
  Sodium; visit 8 (Week 104); n= 39 | 0.9 (2.28)
  Sodium; visit 9 (Week 121); n= 36: number analyzed (Participants) | 36
  Sodium; visit 9 (Week 121); n= 36 | 0.7 (2.78)
  Sodium; visit 10 (Week 138); n= 35: number analyzed (Participants) | 35
  Sodium; visit 10 (Week 138); n= 35 | 0.3 (3.06)
  Sodium; visit 11 (Week 156); n= 28: number analyzed (Participants) | 28
  Sodium; visit 11 (Week 156); n= 28 | 0.9 (3.47)
  Sodium; visit 12 (Week 173); n= 21: number analyzed (Participants) | 21
  Sodium; visit 12 (Week 173); n= 21 | 0.7 (3.38)
  Sodium; visit 13 (Week 190); n= 17: number analyzed (Participants) | 17
  Sodium; visit 13 (Week 190); n= 17 | 0.6 (1.73)
  Sodium; visit 14 (Week 208); n= 10: number analyzed (Participants) | 10
  Sodium; visit 14 (Week 208); n= 10 | -1.2 (1.03)
  Sodium; visit 15 (Week 225); n= 5: number analyzed (Participants) | 5
  Sodium; visit 15 (Week 225); n= 5 | -0.4 (1.52)
  Sodium; visit 16 (Week 242); n= 4: number analyzed (Participants) | 4
  Sodium; visit 16 (Week 242); n= 4 | -0.8 (1.89)
  Sodium; visit 17 (Week 260); n= 4: number analyzed (Participants) | 4
  Sodium; visit 17 (Week 260); n= 4 | 0.8 (2.63)
  Sodium; visit 18 (Week 277); n= 2: number analyzed (Participants) | 2
  Sodium; visit 18 (Week 277); n= 2 | -1.0 (0.00)
  Sodium; withdrawal visit; n= 71: number analyzed (Participants) | 71
  Sodium; withdrawal visit; n= 71 | 0.2 (2.85)
  Sodium; follow up visit; n= 53: number analyzed (Participants) | 53
  Sodium; follow up visit; n= 53 | -0.7 (2.45)
  BUN; visit 1 (Screening); n= 83: number analyzed (Participants) | 83
  BUN; visit 1 (Screening); n= 83 | 0.32 (1.317)
  BUN; visit 2 (Week 13); n= 80: number analyzed (Participants) | 80
  BUN; visit 2 (Week 13); n= 80 | 0.44 (1.483)
  BUN; visit 3 (Week 26); n= 69: number analyzed (Participants) | 69
  BUN; visit 3 (Week 26); n= 69 | 0.31 (1.287)
  BUN; visit 4 (Week 39); n= 64: number analyzed (Participants) | 64
  BUN; visit 4 (Week 39); n= 64 | 0.22 (1.322)
  BUN; visit 5 (Week 52); n= 59: number analyzed (Participants) | 59
  BUN; visit 5 (Week 52); n= 59 | 0.37 (1.643)
  BUN; visit 6 (Week 69); n= 58: number analyzed (Participants) | 58
  BUN; visit 6 (Week 69); n= 58 | 0.13 (1.329)
  BUN; visit 7 (Week 86); n= 51: number analyzed (Participants) | 51
  BUN; visit 7 (Week 86); n= 51 | 0.22 (1.467)
  BUN; visit 8 (Week 104); n= 39: number analyzed (Participants) | 39
  BUN; visit 8 (Week 104); n= 39 | 0.22 (1.477)
  BUN; visit 9 (Week 121); n= 36: number analyzed (Participants) | 36
  BUN; visit 9 (Week 121); n= 36 | 0.35 (1.444)
  BUN; visit 10 (Week 138); n= 35: number analyzed (Participants) | 35
  BUN; visit 10 (Week 138); n= 35 | 0.18 (1.578)
  BUN; visit 11 (Week 156); n= 28: number analyzed (Participants) | 28
  BUN; visit 11 (Week 156); n= 28 | -0.06 (1.515)
  BUN; visit 12 (Week 173); n= 21: number analyzed (Participants) | 21
  BUN; visit 12 (Week 173); n= 21 | -0.40 (1.362)
  BUN; visit 13 (Week 190); n= 17: number analyzed (Participants) | 17
  BUN; visit 13 (Week 190); n= 17 | 0.23 (1.088)
  BUN; visit 14 (Week 208); n= 10: number analyzed (Participants) | 10
  BUN; visit 14 (Week 208); n= 10 | -0.11 (1.604)
  BUN; visit 15 (Week 225); n= 5: number analyzed (Participants) | 5
  BUN; visit 15 (Week 225); n= 5 | -0.40 (1.416)
  BUN; visit 16 (Week 242); n= 4: number analyzed (Participants) | 4
  BUN; visit 16 (Week 242); n= 4 | 0.80 (0.707)
  BUN; visit 17 (Week 260); n= 4: number analyzed (Participants) | 4
  BUN; visit 17 (Week 260); n= 4 | 1.10 (2.889)
  BUN; visit 18 (Week 277); n= 2: number analyzed (Participants) | 2
  BUN; visit 18 (Week 277); n= 2 | 0.50 (0.141)
  BUN; withdrawal visit; n= 71: number analyzed (Participants) | 71
  BUN; withdrawal visit; n= 71 | 0.49 (1.450)
  BUN; follow up visit; n= 53: number analyzed (Participants) | 53
  BUN; follow up visit; n= 53 | 0.14 (1.468)

20. Primary Outcome: Change From Baseline in Absolute Basophils, Absolute Eosinophils, Absolute Lymphocytes, Absolute Monocytes, Absolute Total Neutrophils, Platelet Count and WBC Count
Description: Blood samples were collected from participants for evaluation of change from Baseline in clinical hematology parameters including absolute basophils, eosinophils, lymphocytes, monocytes, neutrophils, platelet count and WBC count. Baseline was defined by and taken directly from the Baseline assessments in the parent study NCT01336621. Change from Baseline was defined as post-Baseline value minus Baseline value. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Time Frame: Baseline and up to 5.8 years
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Giga cells per liter (GI/L)
Arm/Group | Retigabine IR
Number analyzed (Participants) | 98
Giga cells per liter (GI/L)
  Basophils; visit 1 (Screening); n= 84: number analyzed (Participants) | 84
  Basophils; visit 1 (Screening); n= 84 | -0.001 (0.0203)
  Basophils; visit 2 (Week 13); n= 85: number analyzed (Participants) | 85
  Basophils; visit 2 (Week 13); n= 85 | -0.005 (0.0159)
  Basophils; visit 3 (Week 26); n= 71: number analyzed (Participants) | 71
  Basophils; visit 3 (Week 26); n= 71 | -0.003 (0.0197)
  Basophils; visit 4 (Week 39); n= 65: number analyzed (Participants) | 65
  Basophils; visit 4 (Week 39); n= 65 | 0.001 (0.0231)
  Basophils; visit 5 (Week 52); n= 60: number analyzed (Participants) | 60
  Basophils; visit 5 (Week 52); n= 60 | 0.002 (0.0170)
  Basophils; visit 6 (Week 69); n= 58: number analyzed (Participants) | 58
  Basophils; visit 6 (Week 69); n= 58 | -0.002 (0.0202)
  Basophils; visit 7 (Week 86); n= 53: number analyzed (Participants) | 53
  Basophils; visit 7 (Week 86); n= 53 | -0.002 (0.0188)
  Basophils; visit 8 (Week 104); n= 36: number analyzed (Participants) | 36
  Basophils; visit 8 (Week 104); n= 36 | 0.003 (0.0165)
  Basophils; visit 9 (Week 121); n= 35: number analyzed (Participants) | 35
  Basophils; visit 9 (Week 121); n= 35 | -0.002 (0.0183)
  Basophils; visit 10 (Week 138); n= 33: number analyzed (Participants) | 33
  Basophils; visit 10 (Week 138); n= 33 | -0.002 (0.0142)
  Basophils; visit 11 (Week 156); n= 29: number analyzed (Participants) | 29
  Basophils; visit 11 (Week 156); n= 29 | -0.001 (0.0151)
  Basophils; visit 12 (Week 173); n= 24: number analyzed (Participants) | 24
  Basophils; visit 12 (Week 173); n= 24 | -0.004 (0.0125)
  Basophils; visit 13 (Week 190); n= 17: number analyzed (Participants) | 17
  Basophils; visit 13 (Week 190); n= 17 | 0.000 (0.0255)
  Basophils; visit 14 (Week 208); n= 10: number analyzed (Participants) | 10
  Basophils; visit 14 (Week 208); n= 10 | -0.004 (0.0165)
  Basophils; visit 15 (Week 225); n= 4: number analyzed (Participants) | 4
  Basophils; visit 15 (Week 225); n= 4 | -0.010 (0.0115)
  Basophils; visit 16 (Week 242); n= 4: number analyzed (Participants) | 4
  Basophils; visit 16 (Week 242); n= 4 | -0.003 (0.0050)
  Basophils; visit 17 (Week 260); n= 4: number analyzed (Participants) | 4
  Basophils; visit 17 (Week 260); n= 4 | -0.005 (0.0129)
  Basophils; visit 18 (Week 277); n= 2: number analyzed (Participants) | 2
  Basophils; visit 18 (Week 277); n= 2 | 0.000 (0.0000)
  Basophils; withdrawal visit; n= 78: number analyzed (Participants) | 78
  Basophils; withdrawal visit; n= 78 | 0.001 (0.0186)
  Basophils; follow up visit; n= 56: number analyzed (Participants) | 56
  Basophils; follow up visit; n= 56 | -0.008 (0.0190)
  Eosinophils; visit 1 (Screening); n= 84: number analyzed (Participants) | 84
  Eosinophils; visit 1 (Screening); n= 84 | -0.011 (0.1103)
  Eosinophils; visit 2 (Week 13); n= 85: number analyzed (Participants) | 85
  Eosinophils; visit 2 (Week 13); n= 85 | -0.018 (0.2505)
  Eosinophils; visit 3 (Week 26); n= 71: number analyzed (Participants) | 71
  Eosinophils; visit 3 (Week 26); n= 71 | -0.029 (0.2191)
  Eosinophils; visit 4 (Week 39); n= 65: number analyzed (Participants) | 65
  Eosinophils; visit 4 (Week 39); n= 65 | -0.050 (0.2523)
  Eosinophils; visit 5 (Week 52); n= 60: number analyzed (Participants) | 60
  Eosinophils; visit 5 (Week 52); n= 60 | -0.065 (0.3016)
  Eosinophils; visit 6 (Week 69); n= 58: number analyzed (Participants) | 58
  Eosinophils; visit 6 (Week 69); n= 58 | -0.025 (0.1586)
  Eosinophils; visit 7 (Week 86); n= 53: number analyzed (Participants) | 53
  Eosinophils; visit 7 (Week 86); n= 53 | -0.016 (0.1585)
  Eosinophils; visit 8 (Week 104); n= 36: number analyzed (Participants) | 36
  Eosinophils; visit 8 (Week 104); n= 36 | -0.020 (0.1992)
  Eosinophils; visit 9 (Week 121); n= 35: number analyzed (Participants) | 35
  Eosinophils; visit 9 (Week 121); n= 35 | -0.015 (0.1721)
  Eosinophils; visit 10 (Week 138); n= 33: number analyzed (Participants) | 33
  Eosinophils; visit 10 (Week 138); n= 33 | -0.052 (0.1918)
  Eosinophils; visit 11 (Week 156); n= 29: number analyzed (Participants) | 29
  Eosinophils; visit 11 (Week 156); n= 29 | -0.046 (0.1846)
  Eosinophils; visit 12 (Week 173); n= 24: number analyzed (Participants) | 24
  Eosinophils; visit 12 (Week 173); n= 24 | -0.065 (0.3068)
  Eosinophils; visit 13 (Week 190); n= 17: number analyzed (Participants) | 17
  Eosinophils; visit 13 (Week 190); n= 17 | -0.104 (0.3376)
  Eosinophils; visit 14 (Week 208); n= 10: number analyzed (Participants) | 10
  Eosinophils; visit 14 (Week 208); n= 10 | -0.158 (0.1591)
  Eosinophils; visit 15 (Week 225); n= 4: number analyzed (Participants) | 4
  Eosinophils; visit 15 (Week 225); n= 4 | -0.140 (0.0589)
  Eosinophils; visit 16 (Week 242); n= 4: number analyzed (Participants) | 4
  Eosinophils; visit 16 (Week 242); n= 4 | -0.070 (0.1131)
  Eosinophils; visit 17 (Week 260); n= 4: number analyzed (Participants) | 4
  Eosinophils; visit 17 (Week 260); n= 4 | -0.055 (0.0850)
  Eosinophils; visit 18 (Week 277); n= 2: number analyzed (Participants) | 2
  Eosinophils; visit 18 (Week 277); n= 2 | 0.005 (0.0636)
  Eosinophils; withdrawal visit; n= 78: number analyzed (Participants) | 78
  Eosinophils; withdrawal visit; n= 78 | -0.056 (0.2713)
  Eosinophils; follow up visit; n= 56: number analyzed (Participants) | 56
  Eosinophils; follow up visit; n= 56 | -0.091 (0.3022)
  Lymphocytes; visit 1 (Screening); n= 84: number analyzed (Participants) | 84
  Lymphocytes; visit 1 (Screening); n= 84 | -0.225 (0.6631)
  Lymphocytes; visit 2 (Week 13); n= 85: number analyzed (Participants) | 85
  Lymphocytes; visit 2 (Week 13); n= 85 | -0.170 (0.5506)
  Lymphocytes; visit 3 (Week 26); n= 71: number analyzed (Participants) | 71
  Lymphocytes; visit 3 (Week 26); n= 71 | -0.133 (0.6123)
  Lymphocytes; visit 4 (Week 39); n= 65: number analyzed (Participants) | 65
  Lymphocytes; visit 4 (Week 39); n= 65 | -0.210 (0.5412)
  Lymphocytes; visit 5 (Week 52); n= 60: number analyzed (Participants) | 60
  Lymphocytes; visit 5 (Week 52); n= 60 | -0.214 (0.6446)
  Lymphocytes; visit 6 (Week 69); n= 58: number analyzed (Participants) | 58
  Lymphocytes; visit 6 (Week 69); n= 58 | -0.178 (0.5194)
  Lymphocytes; visit 7 (Week 86); n= 53: number analyzed (Participants) | 53
  Lymphocytes; visit 7 (Week 86); n= 53 | -0.093 (0.5793)
  Lymphocytes; visit 8 (Week 104); n= 36: number analyzed (Participants) | 36
  Lymphocytes; visit 8 (Week 104); n= 36 | -0.111 (0.5839)
  Lymphocytes; visit 9 (Week 121); n= 35: number analyzed (Participants) | 35
  Lymphocytes; visit 9 (Week 121); n= 35 | 0.008 (0.8295)
  Lymphocytes; visit 10 (Week 138); n= 33: number analyzed (Participants) | 33
  Lymphocytes; visit 10 (Week 138); n= 33 | -0.177 (0.6622)
  Lymphocytes; visit 11 (Week 156); n= 29: number analyzed (Participants) | 29
  Lymphocytes; visit 11 (Week 156); n= 29 | -0.324 (0.6801)
  Lymphocytes; visit 12 (Week 173); n= 24: number analyzed (Participants) | 24
  Lymphocytes; visit 12 (Week 173); n= 24 | -0.226 (0.5720)
  Lymphocytes; visit 13 (Week 190); n= 17: number analyzed (Participants) | 17
  Lymphocytes; visit 13 (Week 190); n= 17 | -0.325 (0.7086)
  Lymphocytes; visit 14 (Week 208); n= 10: number analyzed (Participants) | 10
  Lymphocytes; visit 14 (Week 208); n= 10 | -0.354 (0.6563)
  Lymphocytes; visit 15 (Week 225); n= 4: number analyzed (Participants) | 4
  Lymphocytes; visit 15 (Week 225); n= 4 | -0.990 (0.6633)
  Lymphocytes; visit 16 (Week 242); n= 4: number analyzed (Participants) | 4
  Lymphocytes; visit 16 (Week 242); n= 4 | -0.818 (0.9694)
  Lymphocytes; visit 17 (Week 260); n= 4: number analyzed (Participants) | 4
  Lymphocytes; visit 17 (Week 260); n= 4 | -0.993 (0.7200)
  Lymphocytes; visit 18 (Week 277); n= 2: number analyzed (Participants) | 2
  Lymphocytes; visit 18 (Week 277); n= 2 | -1.465 (0.6718)
  Lymphocytes; withdrawal visit; n= 78: number analyzed (Participants) | 78
  Lymphocytes; withdrawal visit; n= 78 | -0.153 (0.6466)
  Lymphocytes; follow up visit; n= 56: number analyzed (Participants) | 56
  Lymphocytes; follow up visit; n= 56 | -0.081 (0.7105)
  Monocytes; visit 1 (Screening); n= 84: number analyzed (Participants) | 84
  Monocytes; visit 1 (Screening); n= 84 | -0.043 (0.1800)
  Monocytes; visit 2 (Week 13); n= 85: number analyzed (Participants) | 85
  Monocytes; visit 2 (Week 13); n= 85 | -0.009 (0.1603)
  Monocytes; visit 3 (Week 26); n= 71: number analyzed (Participants) | 71
  Monocytes; visit 3 (Week 26); n= 71 | 0.039 (0.2031)
  Monocytes; visit 4 (Week 39); n= 65: number analyzed (Participants) | 65
  Monocytes; visit 4 (Week 39); n= 65 | -0.005 (0.1940)
  Monocytes; visit 5 (Week 52); n= 60: number analyzed (Participants) | 60
  Monocytes; visit 5 (Week 52); n= 60 | -0.006 (0.1876)
  Monocytes; visit 6 (Week 69); n= 58: number analyzed (Participants) | 58
  Monocytes; visit 6 (Week 69); n= 58 | 0.018 (0.1697)
  Monocytes; visit 7 (Week 86); n= 53: number analyzed (Participants) | 53
  Monocytes; visit 7 (Week 86); n= 53 | 0.055 (0.2375)
  Monocytes; visit 8 (Week 104); n= 36: number analyzed (Participants) | 36
  Monocytes; visit 8 (Week 104); n= 36 | -0.032 (0.1911)
  Monocytes; visit 9 (Week 121); n= 35: number analyzed (Participants) | 35
  Monocytes; visit 9 (Week 121); n= 35 | 0.023 (0.1777)
  Monocytes; visit 10 (Week 138); n= 33: number analyzed (Participants) | 33
  Monocytes; visit 10 (Week 138); n= 33 | 0.005 (0.1796)
  Monocytes; visit 11 (Week 156); n= 29: number analyzed (Participants) | 29
  Monocytes; visit 11 (Week 156); n= 29 | -0.028 (0.1982)
  Monocytes; visit 12 (Week 173); n= 24: number analyzed (Participants) | 24
  Monocytes; visit 12 (Week 173); n= 24 | -0.032 (0.1648)
  Monocytes; visit 13 (Week 190); n= 17: number analyzed (Participants) | 17
  Monocytes; visit 13 (Week 190); n= 17 | -0.078 (0.2279)
  Monocytes; visit 14 (Week 208); n= 10: number analyzed (Participants) | 10
  Monocytes; visit 14 (Week 208); n= 10 | -0.090 (0.2821)
  Monocytes; visit 15 (Week 225); n= 4: number analyzed (Participants) | 4
  Monocytes; visit 15 (Week 225); n= 4 | -0.037 (0.0450)
  Monocytes; visit 16 (Week 242); n= 4: number analyzed (Participants) | 4
  Monocytes; visit 16 (Week 242); n= 4 | -0.020 (0.0829)
  Monocytes; visit 17 (Week 260); n= 4: number analyzed (Participants) | 4
  Monocytes; visit 17 (Week 260); n= 4 | 0.025 (0.1173)
  Monocytes; visit 18 (Week 277); n= 2: number analyzed (Participants) | 2
  Monocytes; visit 18 (Week 277); n= 2 | 0.080 (0.0000)
  Monocytes; withdrawal visit; n= 78: number analyzed (Participants) | 78
  Monocytes; withdrawal visit; n= 78 | 0.041 (0.2417)
  Monocytes; follow up visit; n= 56: number analyzed (Participants) | 56
  Monocytes; follow up visit; n= 56 | -0.021 (0.2091)
  Total neutrophils; visit 1 (Screening); n= 84: number analyzed (Participants) | 84
  Total neutrophils; visit 1 (Screening); n= 84 | -0.108 (1.6418)
  Total neutrophils; visit 2 (Week 13); n= 85: number analyzed (Participants) | 85
  Total neutrophils; visit 2 (Week 13); n= 85 | -0.354 (1.4357)
  Total neutrophils; visit 3 (Week 26); n= 71: number analyzed (Participants) | 71
  Total neutrophils; visit 3 (Week 26); n= 71 | -0.175 (1.4304)
  Total neutrophils; visit 4 (Week 39); n= 65: number analyzed (Participants) | 65
  Total neutrophils; visit 4 (Week 39); n= 65 | -0.582 (1.5237)
  Total neutrophils; visit 5 (Week 52); n= 60: number analyzed (Participants) | 60
  Total neutrophils; visit 5 (Week 52); n= 60 | 0.165 (1.9517)
  Total neutrophils; visit 6 (Week 69); n= 58: number analyzed (Participants) | 58
  Total neutrophils; visit 6 (Week 69); n= 58 | -0.159 (1.5356)
  Total neutrophils; visit 7 (Week 86); n= 53: number analyzed (Participants) | 53
  Total neutrophils; visit 7 (Week 86); n= 53 | -0.046 (2.0418)
  Total neutrophils; visit 8 (Week 104); n= 36: number analyzed (Participants) | 36
  Total neutrophils; visit 8 (Week 104); n= 36 | -0.403 (1.5416)
  Total neutrophils; visit 9 (Week 121); n= 35: number analyzed (Participants) | 35
  Total neutrophils; visit 9 (Week 121); n= 35 | 0.519 (1.9016)
  Total neutrophils; visit 10 (Week 138); n= 33: number analyzed (Participants) | 33
  Total neutrophils; visit 10 (Week 138); n= 33 | 0.412 (1.9080)
  Total neutrophils; visit 11 (Week 156); n= 29: number analyzed (Participants) | 29
  Total neutrophils; visit 11 (Week 156); n= 29 | 0.361 (1.5062)
  Total neutrophils; visit 12 (Week 173); n= 24: number analyzed (Participants) | 24
  Total neutrophils; visit 12 (Week 173); n= 24 | 0.144 (1.7867)
  Total neutrophils; visit 13 (Week 190); n= 17: number analyzed (Participants) | 17
  Total neutrophils; visit 13 (Week 190); n= 17 | 0.669 (2.6453)
  Total neutrophils; visit 14 (Week 208); n= 10: number analyzed (Participants) | 10
  Total neutrophils; visit 14 (Week 208); n= 10 | 0.113 (1.7471)
  Total neutrophils; visit 15 (Week 225); n= 4: number analyzed (Participants) | 4
  Total neutrophils; visit 15 (Week 225); n= 4 | -0.825 (1.9404)
  Total neutrophils; visit 16 (Week 242); n= 4: number analyzed (Participants) | 4
  Total neutrophils; visit 16 (Week 242); n= 4 | -1.183 (1.9538)
  Total neutrophils; visit 17 (Week 260); n= 4: number analyzed (Participants) | 4
  Total neutrophils; visit 17 (Week 260); n= 4 | -0.990 (2.1510)
  Total neutrophils; visit 18 (Week 277); n= 2: number analyzed (Participants) | 2
  Total neutrophils; visit 18 (Week 277); n= 2 | -2.210 (2.6446)
  Total neutrophils; withdrawal visit; n= 78: number analyzed (Participants) | 78
  Total neutrophils; withdrawal visit; n= 78 | 0.209 (1.6761)
  Total neutrophils; follow up visit; n= 56: number analyzed (Participants) | 56
  Total neutrophils; follow up visit; n= 56 | 0.095 (1.9626)
  Platelet count; visit 1 (Screening); n= 84: number analyzed (Participants) | 84
  Platelet count; visit 1 (Screening); n= 84 | -1.7 (34.31)
  Platelet count; visit 2 (Week 13); n= 88: number analyzed (Participants) | 88
  Platelet count; visit 2 (Week 13); n= 88 | 3.7 (38.83)
  Platelet count; visit 3 (Week 26); n= 73: number analyzed (Participants) | 73
  Platelet count; visit 3 (Week 26); n= 73 | 5.1 (44.34)
  Platelet count; visit 4 (Week 39); n= 68: number analyzed (Participants) | 68
  Platelet count; visit 4 (Week 39); n= 68 | 2.9 (45.75)
  Platelet count; visit 5 (Week 52); n= 63: number analyzed (Participants) | 63
  Platelet count; visit 5 (Week 52); n= 63 | 4.1 (37.72)
  Platelet count; visit 6 (Week 69); n= 62: number analyzed (Participants) | 62
  Platelet count; visit 6 (Week 69); n= 62 | 6.9 (39.48)
  Platelet count; visit 7 (Week 86); n= 55: number analyzed (Participants) | 55
  Platelet count; visit 7 (Week 86); n= 55 | 1.5 (50.29)
  Platelet count; visit 8 (Week 104); n= 41: number analyzed (Participants) | 41
  Platelet count; visit 8 (Week 104); n= 41 | 4.5 (43.95)
  Platelet count; visit 9 (Week 121); n= 35: number analyzed (Participants) | 35
  Platelet count; visit 9 (Week 121); n= 35 | 8.7 (45.39)
  Platelet count; visit 10 (Week 138); n= 36: number analyzed (Participants) | 36
  Platelet count; visit 10 (Week 138); n= 36 | 6.8 (42.37)
  Platelet count; visit 11 (Week 156); n= 31: number analyzed (Participants) | 31
  Platelet count; visit 11 (Week 156); n= 31 | 1.9 (37.92)
  Platelet count; visit 12 (Week 173); n= 24: number analyzed (Participants) | 24
  Platelet count; visit 12 (Week 173); n= 24 | 9.7 (37.95)
  Platelet count; visit 13 (Week 190); n= 18: number analyzed (Participants) | 18
  Platelet count; visit 13 (Week 190); n= 18 | 7.0 (37.15)
  Platelet count; visit 14 (Week 208); n= 10: number analyzed (Participants) | 10
  Platelet count; visit 14 (Week 208); n= 10 | 18.9 (69.95)
  Platelet count; visit 15 (Week 225); n= 4: number analyzed (Participants) | 4
  Platelet count; visit 15 (Week 225); n= 4 | -31.3 (11.15)
  Platelet count; visit 16 (Week 242); n= 4: number analyzed (Participants) | 4
  Platelet count; visit 16 (Week 242); n= 4 | -9.0 (63.92)
  Platelet count; visit 17 (Week 260); n= 4: number analyzed (Participants) | 4
  Platelet count; visit 17 (Week 260); n= 4 | -10.0 (61.60)
  Platelet count; visit 18 (Week 277); n= 2: number analyzed (Participants) | 2
  Platelet count; visit 18 (Week 277); n= 2 | -19.0 (100.41)
  Platelet count; withdrawal visit; n= 79: number analyzed (Participants) | 79
  Platelet count; withdrawal visit; n= 79 | 8.9 (43.88)
  Platelet count; follow up visit; n= 58: number analyzed (Participants) | 58
  Platelet count; follow up visit; n= 58 | 8.9 (54.58)
  WBC count; visit 1 (Screening); n= 84: number analyzed (Participants) | 84
  WBC count; visit 1 (Screening); n= 84 | 0.30 (6.496)
  WBC count; visit 2 (Week 13); n= 78: number analyzed (Participants) | 78
  WBC count; visit 2 (Week 13); n= 78 | -0.46 (1.512)
  WBC count; visit 3 (Week 26); n= 66: number analyzed (Participants) | 66
  WBC count; visit 3 (Week 26); n= 66 | -0.24 (1.354)
  WBC count; visit 4 (Week 39); n= 59: number analyzed (Participants) | 59
  WBC count; visit 4 (Week 39); n= 59 | -0.84 (1.627)
  WBC count; visit 5 (Week 52); n= 54: number analyzed (Participants) | 54
  WBC count; visit 5 (Week 52); n= 54 | -0.05 (1.989)
  WBC count; visit 6 (Week 69); n= 54: number analyzed (Participants) | 54
  WBC count; visit 6 (Week 69); n= 54 | -0.41 (1.637)
  WBC count; visit 7 (Week 86); n= 50: number analyzed (Participants) | 50
  WBC count; visit 7 (Week 86); n= 50 | -0.12 (2.059)
  WBC count; visit 8 (Week 104); n= 33: number analyzed (Participants) | 33
  WBC count; visit 8 (Week 104); n= 33 | -0.51 (1.666)
  WBC count; visit 9 (Week 121); n= 32: number analyzed (Participants) | 32
  WBC count; visit 9 (Week 121); n= 32 | 0.58 (1.968)
  WBC count; visit 10 (Week 138); n= 32: number analyzed (Participants) | 32
  WBC count; visit 10 (Week 138); n= 32 | 0.22 (2.106)
  WBC count; visit 11 (Week 156); n= 27: number analyzed (Participants) | 27
  WBC count; visit 11 (Week 156); n= 27 | 0.09 (1.805)
  WBC count; visit 12 (Week 173); n= 22: number analyzed (Participants) | 22
  WBC count; visit 12 (Week 173); n= 22 | -0.15 (1.971)
  WBC count; visit 13 (Week 190); n= 15: number analyzed (Participants) | 15
  WBC count; visit 13 (Week 190); n= 15 | 0.43 (2.804)
  WBC count; visit 14 (Week 208); n= 10: number analyzed (Participants) | 10
  WBC count; visit 14 (Week 208); n= 10 | -0.49 (2.247)
  WBC count; visit 15 (Week 225); n= 4: number analyzed (Participants) | 4
  WBC count; visit 15 (Week 225); n= 4 | -2.00 (2.608)
  WBC count; visit 16 (Week 242); n= 4: number analyzed (Participants) | 4
  WBC count; visit 16 (Week 242); n= 4 | -2.10 (2.825)
  WBC count; visit 17 (Week 260); n= 4: number analyzed (Participants) | 4
  WBC count; visit 17 (Week 260); n= 4 | -2.03 (2.941)
  WBC count; visit 18 (Week 277); n= 2: number analyzed (Participants) | 2
  WBC count; visit 18 (Week 277); n= 2 | -3.60 (3.394)
  WBC count; withdrawal visit; n= 70: number analyzed (Participants) | 70
  WBC count; withdrawal visit; n= 70 | 0.13 (1.757)
  WBC count; follow up visit; n= 50: number analyzed (Participants) | 50
  WBC count; follow up visit; n= 50 | -0.05 (1.905)

21. Primary Outcome: Change From Baseline in Hemoglobin and Mean Corpuscle Hemoglobin Concentration (MCHC) Levels
Description: Blood samples were collected from participants for evaluation of change from Baseline in clinical hematology parameters including hemoglobin and MCHC. Baseline was defined by and taken directly from the Baseline assessments in the parent study NCT01336621. Change from Baseline was defined as post-Baseline value minus Baseline value. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Time Frame: Baseline and up to 5.8 years
Population: Safety Population
Measure: Mean (Standard Deviation); unit: G/L
Arm/Group | Retigabine IR
Number analyzed (Participants) | 98
G/L
  Hemoglobin; visit 1 (Screening); n= 85: number analyzed (Participants) | 85
  Hemoglobin; visit 1 (Screening); n= 85 | -3.5 (6.75)
  Hemoglobin; visit 2 (Week 13); n= 89: number analyzed (Participants) | 89
  Hemoglobin; visit 2 (Week 13); n= 89 | -2.4 (7.87)
  Hemoglobin; visit 3 (Week 26); n= 74: number analyzed (Participants) | 74
  Hemoglobin; visit 3 (Week 26); n= 74 | -2.7 (7.59)
  Hemoglobin; visit 4 (Week 39); n= 69: number analyzed (Participants) | 69
  Hemoglobin; visit 4 (Week 39); n= 69 | -2.9 (9.09)
  Hemoglobin; visit 5 (Week 52); n= 64: number analyzed (Participants) | 64
  Hemoglobin; visit 5 (Week 52); n= 64 | -2.9 (9.51)
  Hemoglobin; visit 6 (Week 69); n= 62: number analyzed (Participants) | 62
  Hemoglobin; visit 6 (Week 69); n= 62 | -2.5 (9.83)
  Hemoglobin; visit 7 (Week 86); n= 55: number analyzed (Participants) | 55
  Hemoglobin; visit 7 (Week 86); n= 55 | -0.4 (8.75)
  Hemoglobin; visit 8 (Week 104); n= 41: number analyzed (Participants) | 41
  Hemoglobin; visit 8 (Week 104); n= 41 | -0.7 (8.35)
  Hemoglobin; visit 9 (Week 121); n= 36: number analyzed (Participants) | 36
  Hemoglobin; visit 9 (Week 121); n= 36 | -1.4 (8.68)
  Hemoglobin; visit 10 (Week 138); n= 36: number analyzed (Participants) | 36
  Hemoglobin; visit 10 (Week 138); n= 36 | 0.1 (12.38)
  Hemoglobin; visit 11 (Week 156); n= 31: number analyzed (Participants) | 31
  Hemoglobin; visit 11 (Week 156); n= 31 | -3.4 (9.73)
  Hemoglobin; visit 12 (Week 173); n= 24: number analyzed (Participants) | 24
  Hemoglobin; visit 12 (Week 173); n= 24 | -2.2 (9.46)
  Hemoglobin; visit 13 (Week 190); n= 18: number analyzed (Participants) | 18
  Hemoglobin; visit 13 (Week 190); n= 18 | -4.3 (9.11)
  Hemoglobin; visit 14 (Week 208); n= 10 | -8.0 (10.02)
  Hemoglobin; visit 15 (Week 225); n= 4: number analyzed (Participants) | 4
  Hemoglobin; visit 15 (Week 225); n= 4 | -6.0 (4.76)
  Hemoglobin; visit 16 (Week 242); n= 4: number analyzed (Participants) | 4
  Hemoglobin; visit 16 (Week 242); n= 4 | -9.5 (6.66)
  Hemoglobin; visit 17 (Week 260); n= 4: number analyzed (Participants) | 4
  Hemoglobin; visit 17 (Week 260); n= 4 | -8.0 (6.16)
  Hemoglobin; visit 18 (Week 277); n= 2: number analyzed (Participants) | 2
  Hemoglobin; visit 18 (Week 277); n= 2 | -10.5 (7.78)
  Hemoglobin; withdrawal visit; n= 79: number analyzed (Participants) | 79
  Hemoglobin; withdrawal visit; n= 79 | -1.7 (9.69)
  Hemoglobin; follow up visit; n= 59: number analyzed (Participants) | 59
  Hemoglobin; follow up visit; n= 59 | -2.3 (11.53)
  MCHC; visit 1 (Screening); n= 85: number analyzed (Participants) | 85
  MCHC; visit 1 (Screening); n= 85 | -2.1 (12.61)
  MCHC; visit 2 (Week 13); n= 89: number analyzed (Participants) | 89
  MCHC; visit 2 (Week 13); n= 89 | 1.4 (12.22)
  MCHC; visit 3 (Week 26); n= 74: number analyzed (Participants) | 74
  MCHC; visit 3 (Week 26); n= 74 | -1.1 (11.50)
  MCHC; visit 4 (Week 39); n= 69: number analyzed (Participants) | 69
  MCHC; visit 4 (Week 39); n= 69 | -4.6 (12.75)
  MCHC; visit 5 (Week 52); n= 64: number analyzed (Participants) | 64
  MCHC; visit 5 (Week 52); n= 64 | -5.4 (13.35)
  MCHC; visit 6 (Week 69); n= 62: number analyzed (Participants) | 62
  MCHC; visit 6 (Week 69); n= 62 | -4.8 (11.64)
  MCHC; visit 7 (Week 86); n= 55: number analyzed (Participants) | 55
  MCHC; visit 7 (Week 86); n= 55 | -5.8 (9.79)
  MCHC; visit 8 (Week 104); n= 41 | -9.1 (10.62)
  MCHC; visit 9 (Week 121); n= 36: number analyzed (Participants) | 36
  MCHC; visit 9 (Week 121); n= 36 | -6.9 (11.74)
  MCHC; visit 10 (Week 138); n= 36: number analyzed (Participants) | 36
  MCHC; visit 10 (Week 138); n= 36 | -9.6 (9.87)
  MCHC; visit 11 (Week 156); n= 31: number analyzed (Participants) | 31
  MCHC; visit 11 (Week 156); n= 31 | -10.1 (11.76)
  MCHC; visit 12 (Week 173); n= 24: number analyzed (Participants) | 24
  MCHC; visit 12 (Week 173); n= 24 | -10.7 (9.45)
  MCHC; visit 13 (Week 190); n= 18: number analyzed (Participants) | 18
  MCHC; visit 13 (Week 190); n= 18 | -15.2 (9.24)
  MCHC; visit 14 (Week 208); n= 10: number analyzed (Participants) | 10
  MCHC; visit 14 (Week 208); n= 10 | -21.5 (10.48)
  MCHC; visit 15 (Week 225); n= 4: number analyzed (Participants) | 4
  MCHC; visit 15 (Week 225); n= 4 | -16.3 (7.59)
  MCHC; visit 16 (Week 242); n= 4: number analyzed (Participants) | 4
  MCHC; visit 16 (Week 242); n= 4 | -14.5 (5.51)
  MCHC; visit 17 (Week 260); n= 4: number analyzed (Participants) | 4
  MCHC; visit 17 (Week 260); n= 4 | -16.0 (8.25)
  MCHC; visit 18 (Week 277); n= 2: number analyzed (Participants) | 2
  MCHC; visit 18 (Week 277); n= 2 | -4.5 (9.19)
  MCHC; withdrawal visit; n= 79: number analyzed (Participants) | 79
  MCHC; withdrawal visit; n= 79 | -6.8 (9.61)
  MCHC; follow up visit; n= 59: number analyzed (Participants) | 59
  MCHC; follow up visit; n= 59 | -8.6 (10.18)

22. Primary Outcome: Change From Baseline in Hematocrit Levels
Description: Blood samples were collected from participants for evaluation of change from Baseline in clinical hematology parameters including hematocrit. Baseline was defined by and taken directly from the Baseline assessments in the parent study NCT01336621. Change from Baseline was defined as post-Baseline value minus Baseline value. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Time Frame: Baseline and up to 5.8 years
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Proportion of red blood cells in blood
Arm/Group | Retigabine IR
Number analyzed (Participants) | 98
Proportion of red blood cells in blood
  Visit 1 (Screening); n= 85: number analyzed (Participants) | 85
  Visit 1 (Screening); n= 85 | -0.0080 (0.02259)
  Visit 2 (Week 13); n= 89: number analyzed (Participants) | 89
  Visit 2 (Week 13); n= 89 | -0.0087 (0.02508)
  Visit 3 (Week 26); n= 74: number analyzed (Participants) | 74
  Visit 3 (Week 26); n= 74 | -0.0066 (0.02651)
  Visit 4 (Week 39); n= 69: number analyzed (Participants) | 69
  Visit 4 (Week 39); n= 69 | -0.0030 (0.02861)
  Visit 5 (Week 52); n= 64: number analyzed (Participants) | 64
  Visit 5 (Week 52); n= 64 | -0.0020 (0.02985)
  Visit 6 (Week 69); n= 62: number analyzed (Participants) | 62
  Visit 6 (Week 69); n= 62 | -0.0020 (0.02821)
  Visit 7 (Week 86); n= 55: number analyzed (Participants) | 55
  Visit 7 (Week 86); n= 55 | 0.0063 (0.02627)
  Visit 8 (Week 104); n= 41: number analyzed (Participants) | 41
  Visit 8 (Week 104); n= 41 | 0.0103 (0.02839)
  Visit 9 (Week 121); n= 36: number analyzed (Participants) | 36
  Visit 9 (Week 121); n= 36 | 0.0053 (0.02819)
  Visit 10 (Week 138); n= 36: number analyzed (Participants) | 36
  Visit 10 (Week 138); n= 36 | 0.0129 (0.04091)
  Visit 11 (Week 156); n= 31: number analyzed (Participants) | 31
  Visit 11 (Week 156); n= 31 | 0.0025 (0.02755)
  Visit 12 (Week 173); n= 24: number analyzed (Participants) | 24
  Visit 12 (Week 173); n= 24 | 0.0070 (0.03167)
  Visit 13 (Week 190); n= 18: number analyzed (Participants) | 18
  Visit 13 (Week 190); n= 18 | 0.0061 (0.02857)
  Visit 14 (Week 208); n= 10: number analyzed (Participants) | 10
  Visit 14 (Week 208); n= 10 | 0.0015 (0.03213)
  Visit 15 (Week 225); n= 4: number analyzed (Participants) | 4
  Visit 15 (Week 225); n= 4 | 0.0050 (0.01857)
  Visit 16 (Week 242); n= 4: number analyzed (Participants) | 4
  Visit 16 (Week 242); n= 4 | -0.0097 (0.02017)
  Visit 17 (Week 260); n= 4: number analyzed (Participants) | 4
  Visit 17 (Week 260); n= 4 | -0.0040 (0.00841)
  Visit 18 (Week 277); n= 2: number analyzed (Participants) | 2
  Visit 18 (Week 277); n= 2 | -0.0270 (0.03677)
  Withdrawal visit; n= 79: number analyzed (Participants) | 79
  Withdrawal visit; n= 79 | 0.0034 (0.02926)
  Follow up visit; n= 59: number analyzed (Participants) | 59
  Follow up visit; n= 59 | 0.0039 (0.03501)

23. Primary Outcome: Change From Baseline in Mean Corpuscle Hemoglobin (MCH) Levels
Description: Blood samples were collected from participants for evaluation of change from Baseline in clinical hematology parameters including MCH. Baseline was defined by and taken directly from the Baseline assessments in the parent study NCT01336621. Change from Baseline was defined as post-Baseline value minus Baseline value. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Time Frame: Baseline and up to 5.8 years
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Picograms (Pg)
Arm/Group | Retigabine IR
Number analyzed (Participants) | 98
Picograms (Pg)
  Visit 1 (Screening); n= 85: number analyzed (Participants) | 85
  Visit 1 (Screening); n= 85 | -0.17 (0.910)
  Visit 2 (Week 13); n= 89: number analyzed (Participants) | 89
  Visit 2 (Week 13); n= 89 | -0.33 (1.058)
  Visit 3 (Week 26); n= 74: number analyzed (Participants) | 74
  Visit 3 (Week 26); n= 74 | -0.47 (0.809)
  Visit 4 (Week 39); n= 69: number analyzed (Participants) | 69
  Visit 4 (Week 39); n= 69 | -0.83 (1.238)
  Visit 5 (Week 52); n= 64: number analyzed (Participants) | 64
  Visit 5 (Week 52); n= 64 | -0.77 (1.087)
  Visit 6 (Week 69); n= 62: number analyzed (Participants) | 62
  Visit 6 (Week 69); n= 62 | -0.91 (1.317)
  Visit 7 (Week 86); n= 55: number analyzed (Participants) | 55
  Visit 7 (Week 86); n= 55 | -0.99 (1.227)
  Visit 8 (Week 104); n= 41: number analyzed (Participants) | 41
  Visit 8 (Week 104); n= 41 | -1.17 (1.503)
  Visit 9 (Week 121); n= 36: number analyzed (Participants) | 36
  Visit 9 (Week 121); n= 36 | -1.11 (1.551)
  Visit 10 (Week 138); n= 36: number analyzed (Participants) | 36
  Visit 10 (Week 138); n= 36 | -1.28 (1.282)
  Visit 11 (Week 156); n= 31: number analyzed (Participants) | 31
  Visit 11 (Week 156); n= 31 | -1.44 (1.065)
  Visit 12 (Week 173); n= 24: number analyzed (Participants) | 24
  Visit 12 (Week 173); n= 24 | -1.78 (1.380)
  Visit 13 (Week 190); n= 18: number analyzed (Participants) | 18
  Visit 13 (Week 190); n= 18 | -1.90 (1.251)
  Visit 14 (Week 208); n= 10: number analyzed (Participants) | 10
  Visit 14 (Week 208); n= 10 | -2.19 (1.883)
  Visit 15 (Week 225); n= 4: number analyzed (Participants) | 4
  Visit 15 (Week 225); n= 4 | -2.00 (1.291)
  Visit 16 (Week 242); n= 4: number analyzed (Participants) | 4
  Visit 16 (Week 242); n= 4 | -2.50 (1.669)
  Visit 17 (Week 260); n= 4: number analyzed (Participants) | 4
  Visit 17 (Week 260); n= 4 | -1.83 (1.382)
  Visit 18 (Week 277); n= 2: number analyzed (Participants) | 2
  Visit 18 (Week 277); n= 2 | -2.65 (0.354)
  Withdrawal visit; n= 79: number analyzed (Participants) | 79
  Withdrawal visit; n= 79 | -1.11 (1.305)
  Follow up visit; n= 59: number analyzed (Participants) | 59
  Follow up visit; n= 59 | -1.08 (1.437)

24. Primary Outcome: Change From Baseline in Mean Corpuscle Volume (MCV) and Mean Platelet Volume (MPV) Levels
Description: Blood samples were collected from participants for evaluation of change from Baseline in clinical hematology parameters including MCV and MPV. Baseline was defined by and taken directly from the Baseline assessments in the parent study NCT01336621. Change from Baseline was defined as post-Baseline value minus Baseline value. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Time Frame: Baseline and up to 5.8 years
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Femtoliter (fL)
Arm/Group | Retigabine IR
Number analyzed (Participants) | 98
Femtoliter (fL)
  MCV (Screening); Visit 1; n= 85: number analyzed (Participants) | 85
  MCV (Screening); Visit 1; n= 85 | 0.0 (3.55)
  MCV; Visit 2 (Week 13); n= 89: number analyzed (Participants) | 89
  MCV; Visit 2 (Week 13); n= 89 | -1.5 (3.63)
  MCV; Visit 3 (Week 26); n= 74: number analyzed (Participants) | 74
  MCV; Visit 3 (Week 26); n= 74 | -1.0 (3.32)
  MCV; Visit 4 (Week 39); n= 69: number analyzed (Participants) | 69
  MCV; Visit 4 (Week 39); n= 69 | -1.2 (3.62)
  MCV; Visit 5 (Week 52); n= 64: number analyzed (Participants) | 64
  MCV; Visit 5 (Week 52); n= 64 | -0.8 (3.71)
  MCV; Visit 6 (Week 69); n= 62: number analyzed (Participants) | 62
  MCV; Visit 6 (Week 69); n= 62 | -1.4 (4.29)
  MCV; Visit 7 (Week 86); n= 55: number analyzed (Participants) | 55
  MCV; Visit 7 (Week 86); n= 55 | -1.2 (3.56)
  MCV; Visit 8 (Week 104); n= 41: number analyzed (Participants) | 41
  MCV; Visit 8 (Week 104); n= 41 | -0.9 (4.75)
  MCV; Visit 9 (Week 121); n= 36: number analyzed (Participants) | 36
  MCV; Visit 9 (Week 121); n= 36 | -1.4 (4.00)
  MCV; Visit 10 (Week 138); n= 36: number analyzed (Participants) | 36
  MCV; Visit 10 (Week 138); n= 36 | -1.1 (4.30)
  MCV; Visit 11 (Week 156); n= 31: number analyzed (Participants) | 31
  MCV; Visit 11 (Week 156); n= 31 | -1.5 (4.18)
  MCV; Visit 12 (Week 173); n= 24: number analyzed (Participants) | 24
  MCV; Visit 12 (Week 173); n= 24 | -2.5 (4.64)
  MCV; Visit 13 (Week 190); n= 18: number analyzed (Participants) | 18
  MCV; Visit 13 (Week 190); n= 18 | -1.2 (4.40)
  MCV; Visit 14 (Week 208); n= 10: number analyzed (Participants) | 10
  MCV; Visit 14 (Week 208); n= 10 | -0.9 (4.48)
  MCV; Visit 15 (Week 225); n= 4: number analyzed (Participants) | 4
  MCV; Visit 15 (Week 225); n= 4 | -1.5 (1.73)
  MCV; Visit 16 (Week 242); n= 4: number analyzed (Participants) | 4
  MCV; Visit 16 (Week 242); n= 4 | -4.0 (3.92)
  MCV; Visit 17 (Week 260); n= 4: number analyzed (Participants) | 4
  MCV; Visit 17 (Week 260); n= 4 | -1.3 (2.63)
  MCV; Visit 18 (Week 277); n= 2: number analyzed (Participants) | 2
  MCV; Visit 18 (Week 277); n= 2 | -7.0 (4.24)
  MCV; Withdrawal visit; n= 79: number analyzed (Participants) | 79
  MCV; Withdrawal visit; n= 79 | -1.4 (4.14)
  MCV; Follow up visit; n= 59: number analyzed (Participants) | 59
  MCV; Follow up visit; n= 59 | -0.9 (4.39)
  MPV; visit 1 (Screening); n= 84: number analyzed (Participants) | 84
  MPV; visit 1 (Screening); n= 84 | -0.12 (0.715)
  MPV: visit 2 (Week 13); n= 86: number analyzed (Participants) | 86
  MPV: visit 2 (Week 13); n= 86 | -0.10 (0.756)
  MPV: visit 3 (Week 26); n= 71: number analyzed (Participants) | 71
  MPV: visit 3 (Week 26); n= 71 | -0.08 (0.612)
  MPV; visit 4 (Week 39); n= 67: number analyzed (Participants) | 67
  MPV; visit 4 (Week 39); n= 67 | -0.17 (0.823)
  MPV; visit 5 (Week 52); n= 61: number analyzed (Participants) | 61
  MPV; visit 5 (Week 52); n= 61 | -0.06 (0.746)
  MPV; visit 6 (Week 69); n= 58: number analyzed (Participants) | 58
  MPV; visit 6 (Week 69); n= 58 | -0.03 (0.654)
  MPV; visit 7 (Week 86); n= 53: number analyzed (Participants) | 53
  MPV; visit 7 (Week 86); n= 53 | 0.12 (0.786)
  MPV; visit 8 (Week 104); n= 38: number analyzed (Participants) | 38
  MPV; visit 8 (Week 104); n= 38 | 0.01 (0.902)
  MPV: visit 9 (Week 121); n= 35: number analyzed (Participants) | 35
  MPV: visit 9 (Week 121); n= 35 | 0.13 (0.788)
  MPV; visit 10 (Week 138); n= 34: number analyzed (Participants) | 34
  MPV; visit 10 (Week 138); n= 34 | 0.06 (0.773)
  MPV; visit 11 (Week 156); n= 29: number analyzed (Participants) | 29
  MPV; visit 11 (Week 156); n= 29 | 0.14 (0.728)
  MPV: visit 12 (Week 173); n= 24: number analyzed (Participants) | 24
  MPV: visit 12 (Week 173); n= 24 | 0.04 (0.944)
  MPV; visit 13 (Week 190); n= 17: number analyzed (Participants) | 17
  MPV; visit 13 (Week 190); n= 17 | -0.09 (0.766)
  MPV; visit 14 (Week 208); n= 10: number analyzed (Participants) | 10
  MPV; visit 14 (Week 208); n= 10 | -0.37 (0.455)
  MPV; visit 15 (Week 225); n= 4: number analyzed (Participants) | 4
  MPV; visit 15 (Week 225); n= 4 | -0.33 (1.053)
  MPV; visit 16 (Week 242); n= 4: number analyzed (Participants) | 4
  MPV; visit 16 (Week 242); n= 4 | -0.75 (0.802)
  MPV; visit 17 (Week 260); n= 4: number analyzed (Participants) | 4
  MPV; visit 17 (Week 260); n= 4 | -0.17 (0.670)
  MPV; visit 18 (Week 277); n= 2: number analyzed (Participants) | 2
  MPV; visit 18 (Week 277); n= 2 | -1.15 (0.071)
  MPV; withdrawal visit; n= 78: number analyzed (Participants) | 78
  MPV; withdrawal visit; n= 78 | 0.19 (0.902)
  MPV; follow up visit; n= 57: number analyzed (Participants) | 57
  MPV; follow up visit; n= 57 | 0.12 (0.859)

25. Primary Outcome: Change From Baseline in RBC Count
Description: Blood samples were collected from participants for evaluation of change from Baseline in clinical hematology parameters including RBC count. Baseline was defined by and taken directly from the Baseline assessments in the parent study NCT01336621. Change from Baseline was defined as post-Baseline value minus Baseline value. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Time Frame: Up to 5.8 years
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Tetra cells per liter (TI/L)
Arm/Group | Retigabine IR
Number analyzed (Participants) | 98
Tetra cells per liter (TI/L)
  Visit 1 (Screening); n= 85: number analyzed (Participants) | 85
  Visit 1 (Screening); n= 85 | -0.10 (0.212)
  Visit 2 (Week 13); n= 89: number analyzed (Participants) | 89
  Visit 2 (Week 13); n= 89 | -0.03 (0.255)
  Visit 3 (Week 26); n= 74: number analyzed (Participants) | 74
  Visit 3 (Week 26); n= 74 | -0.03 (0.240)
  Visit 4 (Week 39); n= 69: number analyzed (Participants) | 69
  Visit 4 (Week 39); n= 69 | 0.01 (0.272)
  Visit 5 (Week 52); n= 64: number analyzed (Participants) | 64
  Visit 5 (Week 52); n= 64 | 0.00 (0.311)
  Visit 6 (Week 69); n= 62: number analyzed (Participants) | 62
  Visit 6 (Week 69); n= 62 | 0.04 (0.300)
  Visit 7 (Week 86); n= 55: number analyzed (Participants) | 55
  Visit 7 (Week 86); n= 55 | 0.12 (0.260)
  Visit 8 (Week 104); n= 41: number analyzed (Participants) | 41
  Visit 8 (Week 104); n= 41 | 0.14 (0.280)
  Visit 9 (Week 121); n= 36: number analyzed (Participants) | 36
  Visit 9 (Week 121); n= 36 | 0.11 (0.299)
  Visit 10 (Week 138); n= 36: number analyzed (Participants) | 36
  Visit 10 (Week 138); n= 36 | 0.19 (0.445)
  Visit 11 (Week 156); n= 31: number analyzed (Participants) | 31
  Visit 11 (Week 156); n= 31 | 0.09 (0.344)
  Visit 12 (Week 173); n= 24: number analyzed (Participants) | 24
  Visit 12 (Week 173); n= 24 | 0.18 (0.385)
  Visit 13 (Week 190); n= 18: number analyzed (Participants) | 18
  Visit 13 (Week 190); n= 18 | 0.12 (0.343)
  Visit 14 (Week 208); n= 10: number analyzed (Participants) | 10
  Visit 14 (Week 208); n= 10 | 0.05 (0.366)
  Visit 15 (Week 225); n= 4: number analyzed (Participants) | 4
  Visit 15 (Week 225); n= 4 | 0.13 (0.206)
  Visit 16 (Week 242); n= 4: number analyzed (Participants) | 4
  Visit 16 (Week 242); n= 4 | 0.10 (0.216)
  Visit 17 (Week 260); n= 4: number analyzed (Participants) | 4
  Visit 17 (Week 260); n= 4 | 0.00 (0.082)
  Visit 18 (Week 277); n= 2: number analyzed (Participants) | 2
  Visit 18 (Week 277); n= 2 | 0.05 (0.212)
  Withdrawal visit; n= 79: number analyzed (Participants) | 79
  Withdrawal visit; n= 79 | 0.10 (0.327)
  Follow up visit; n= 59: number analyzed (Participants) | 59
  Follow up visit; n= 59 | 0.07 (0.409)

26. Primary Outcome: Change From Baseline in Percent Basophils, Percent Eosinophils, Percent Lymphocytes, Percent Monocytes, Percent Neutrophils and RBC Distribution Width (RDW) Levels
Description: Blood samples were collected from participants for evaluation of change from Baseline in clinical hematology parameters including percent basophils, eosinophils, lymphocytes, monocytes, neutrophils and RDW. Baseline was defined by and taken directly from the Baseline assessments in the parent study NCT01336621. Change from Baseline was defined as post-Baseline value minus Baseline value. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Time Frame: Baseline and up to 5.8 years
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Percent of blood components
Arm/Group | Retigabine IR
Number analyzed (Participants) | 98
Percent of blood components
  Percent basophils; visit 1 (Screening); n= 84: number analyzed (Participants) | 84
  Percent basophils; visit 1 (Screening); n= 84 | -0.00 (0.312)
  Percent basophils; visit 2 (Week 13); n= 85: number analyzed (Participants) | 85
  Percent basophils; visit 2 (Week 13); n= 85 | -0.06 (0.243)
  Percent basophils; visit 3 (Week 26); n= 71: number analyzed (Participants) | 71
  Percent basophils; visit 3 (Week 26); n= 71 | -0.03 (0.305)
  Percent basophils; visit 4 (Week 39); n= 65: number analyzed (Participants) | 65
  Percent basophils; visit 4 (Week 39); n= 65 | 0.07 (0.393)
  Percent basophils; visit 5 (Week 52); n= 60: number analyzed (Participants) | 60
  Percent basophils; visit 5 (Week 52); n= 60 | 0.04 (0.279)
  Percent basophils; visit 6 (Week 69); n= 58: number analyzed (Participants) | 58
  Percent basophils; visit 6 (Week 69); n= 58 | -0.02 (0.315)
  Percent basophils; visit 7 (Week 86); n= 53: number analyzed (Participants) | 53
  Percent basophils; visit 7 (Week 86); n= 53 | -0.02 (0.302)
  Percent basophils; visit 8 (Week 104); n= 36: number analyzed (Participants) | 36
  Percent basophils; visit 8 (Week 104); n= 36 | 0.11 (0.271)
  Percent basophils; visit 9 (Week 121); n= 35: number analyzed (Participants) | 35
  Percent basophils; visit 9 (Week 121); n= 35 | -0.06 (0.239)
  Percent basophils; visit 10 (Week 138); n= 33: number analyzed (Participants) | 33
  Percent basophils; visit 10 (Week 138); n= 33 | -0.02 (0.255)
  Percent basophils; visit 11 (Week 156); n= 29: number analyzed (Participants) | 29
  Percent basophils; visit 11 (Week 156); n= 29 | -0.00 (0.267)
  Percent basophils; visit 12 (Week 173); n= 24: number analyzed (Participants) | 24
  Percent basophils; visit 12 (Week 173); n= 24 | -0.06 (0.253)
  Percent basophils; visit 13 (Week 190); n= 17: number analyzed (Participants) | 17
  Percent basophils; visit 13 (Week 190); n= 17 | -0.01 (0.339)
  Percent basophils; visit 14 (Week 208); n= 10: number analyzed (Participants) | 10
  Percent basophils; visit 14 (Week 208); n= 10 | -0.03 (0.283)
  Percent basophils; visit 15 (Week 225); n= 4: number analyzed (Participants) | 4
  Percent basophils; visit 15 (Week 225); n= 4 | 0.00 (0.216)
  Percent basophils; visit 16 (Week 242); n= 4: number analyzed (Participants) | 4
  Percent basophils; visit 16 (Week 242); n= 4 | 0.03 (0.126)
  Percent basophils; visit 17 (Week 260); n= 4: number analyzed (Participants) | 4
  Percent basophils; visit 17 (Week 260); n= 4 | 0.03 (0.050)
  Percent basophils; visit 18 (Week 277); n= 2: number analyzed (Participants) | 2
  Percent basophils; visit 18 (Week 277); n= 2 | 0.25 (0.212)
  Percent basophils; withdrawal visit; n= 78: number analyzed (Participants) | 78
  Percent basophils; withdrawal visit; n= 78 | 0.01 (0.291)
  Percent basophils; follow up visit; n= 56: number analyzed (Participants) | 56
  Percent basophils; follow up visit; n= 56 | -0.13 (0.304)
  Percent eosinophils; visit 1 (Screening); n= 84: number analyzed (Participants) | 84
  Percent eosinophils; visit 1 (Screening); n= 84 | -0.06 (1.745)
  Percent eosinophils; visit 2 (Week 13); n= 85: number analyzed (Participants) | 85
  Percent eosinophils; visit 2 (Week 13); n= 85 | -0.00 (3.214)
  Percent eosinophils; visit 3 (Week 26); n= 71: number analyzed (Participants) | 71
  Percent eosinophils; visit 3 (Week 26); n= 71 | -0.29 (2.773)
  Percent eosinophils; visit 4 (Week 39); n= 65: number analyzed (Participants) | 65
  Percent eosinophils; visit 4 (Week 39); n= 65 | -0.44 (3.339)
  Percent eosinophils; visit 5 (Week 52); n= 60: number analyzed (Participants) | 60
  Percent eosinophils; visit 5 (Week 52); n= 60 | -0.77 (4.046)
  Percent eosinophils; visit 6 (Week 69); n= 58: number analyzed (Participants) | 58
  Percent eosinophils; visit 6 (Week 69); n= 58 | -0.26 (2.630)
  Percent eosinophils; visit 7 (Week 86); n= 53: number analyzed (Participants) | 53
  Percent eosinophils; visit 7 (Week 86); n= 53 | -0.30 (2.634)
  Percent eosinophils; visit 8 (Week 104); n= 36: number analyzed (Participants) | 36
  Percent eosinophils; visit 8 (Week 104); n= 36 | -0.04 (3.003)
  Percent eosinophils; visit 9 (Week 121); n= 35: number analyzed (Participants) | 35
  Percent eosinophils; visit 9 (Week 121); n= 35 | -0.47 (2.653)
  Percent eosinophils; visit 10 (Week 138); n= 33: number analyzed (Participants) | 33
  Percent eosinophils; visit 10 (Week 138); n= 33 | -0.92 (2.942)
  Percent eosinophils; visit 11 (Week 156); n= 29: number analyzed (Participants) | 29
  Percent eosinophils; visit 11 (Week 156); n= 29 | -0.79 (2.484)
  Percent eosinophils; visit 12 (Week 173); n= 24: number analyzed (Participants) | 24
  Percent eosinophils; visit 12 (Week 173); n= 24 | -0.70 (5.548)
  Percent eosinophils; visit 13 (Week 190); n= 17: number analyzed (Participants) | 17
  Percent eosinophils; visit 13 (Week 190); n= 17 | -1.38 (5.539)
  Percent eosinophils; visit 14 (Week 208); n= 10: number analyzed (Participants) | 10
  Percent eosinophils; visit 14 (Week 208); n= 10 | -2.49 (2.975)
  Percent eosinophils; visit 15 (Week 225); n= 4: number analyzed (Participants) | 4
  Percent eosinophils; visit 15 (Week 225); n= 4 | -1.53 (1.565)
  Percent eosinophils; visit 16 (Week 242); n= 4: number analyzed (Participants) | 4
  Percent eosinophils; visit 16 (Week 242); n= 4 | -0.43 (1.628)
  Percent eosinophils; visit 17 (Week 260); n= 4: number analyzed (Participants) | 4
  Percent eosinophils; visit 17 (Week 260); n= 4 | 0.00 (1.359)
  Percent eosinophils; visit 18 (Week 277); n= 2: number analyzed (Participants) | 2
  Percent eosinophils; visit 18 (Week 277); n= 2 | 1.65 (0.636)
  Percent eosinophils; withdrawal visit; n= 78: number analyzed (Participants) | 78
  Percent eosinophils; withdrawal visit; n= 78 | -0.83 (3.466)
  Percent eosinophils; follow up visit; n= 56: number analyzed (Participants) | 56
  Percent eosinophils; follow up visit; n= 56 | -1.30 (3.804)
  Percent lymphocytes; visit 1 (Screening); n= 84: number analyzed (Participants) | 84
  Percent lymphocytes; visit 1 (Screening); n= 84 | -2.21 (8.440)
  Percent lymphocytes; visit 2 (Week 13); n= 85: number analyzed (Participants) | 85
  Percent lymphocytes; visit 2 (Week 13); n= 85 | -0.40 (9.550)
  Percent lymphocytes; visit 3 (Week 26); n= 71: number analyzed (Participants) | 71
  Percent lymphocytes; visit 3 (Week 26); n= 71 | -1.14 (10.820)
  Percent lymphocytes; visit 4 (Week 39); n= 65: number analyzed (Participants) | 65
  Percent lymphocytes; visit 4 (Week 39); n= 65 | 0.27 (9.306)
  Percent lymphocytes; visit 5 (Week 52); n= 60: number analyzed (Participants) | 60
  Percent lymphocytes; visit 5 (Week 52); n= 60 | -2.58 (11.216)
  Percent lymphocytes; visit 6 (Week 69); n= 58: number analyzed (Participants) | 58
  Percent lymphocytes; visit 6 (Week 69); n= 58 | -1.26 (8.119)
  Percent lymphocytes; visit 7 (Week 86); n= 53: number analyzed (Participants) | 53
  Percent lymphocytes; visit 7 (Week 86); n= 53 | -0.53 (11.226)
  Percent lymphocytes; visit 8 (Week 104); n= 36: number analyzed (Participants) | 36
  Percent lymphocytes; visit 8 (Week 104); n= 36 | 0.69 (9.013)
  Percent lymphocytes; visit 9 (Week 121); n= 35: number analyzed (Participants) | 35
  Percent lymphocytes; visit 9 (Week 121); n= 35 | -2.27 (11.733)
  Percent lymphocytes; visit 10 (Week 138); n= 33: number analyzed (Participants) | 33
  Percent lymphocytes; visit 10 (Week 138); n= 33 | -3.91 (8.960)
  Percent lymphocytes; visit 11 (Week 156); n= 29: number analyzed (Participants) | 29
  Percent lymphocytes; visit 11 (Week 156); n= 29 | -4.52 (9.015)
  Percent lymphocytes; visit 12 (Week 173); n= 24: number analyzed (Participants) | 24
  Percent lymphocytes; visit 12 (Week 173); n= 24 | -3.19 (9.398)
  Percent lymphocytes; visit 13 (Week 190); n= 17: number analyzed (Participants) | 17
  Percent lymphocytes; visit 13 (Week 190); n= 17 | -4.73 (12.168)
  Percent lymphocytes; visit 14 (Week 208); n= 10: number analyzed (Participants) | 10
  Percent lymphocytes; visit 14 (Week 208); n= 10 | -3.72 (5.911)
  Percent lymphocytes; visit 15 (Week 225); n= 4: number analyzed (Participants) | 4
  Percent lymphocytes; visit 15 (Week 225); n= 4 | -6.58 (3.848)
  Percent lymphocytes; visit 16 (Week 242); n= 4: number analyzed (Participants) | 4
  Percent lymphocytes; visit 16 (Week 242); n= 4 | -3.88 (10.160)
  Percent lymphocytes; visit 17 (Week 260); n= 4: number analyzed (Participants) | 4
  Percent lymphocytes; visit 17 (Week 260); n= 4 | -5.85 (4.886)
  Percent lymphocytes; visit 18 (Week 277); n= 2: number analyzed (Participants) | 2
  Percent lymphocytes; visit 18 (Week 277); n= 2 | -8.10 (3.818)
  Percent lymphocytes; withdrawal visit; n= 78: number analyzed (Participants) | 78
  Percent lymphocytes; withdrawal visit; n= 78 | -2.60 (10.978)
  Percent lymphocytes; follow up visit; n= 56: number analyzed (Participants) | 56
  Percent lymphocytes; follow up visit; n= 56 | -0.81 (12.709)
  Percent monocytes; visit 1 (Screening); n= 84: number analyzed (Participants) | 84
  Percent monocytes; visit 1 (Screening); n= 84 | -0.33 (3.048)
  Percent monocytes; visit 2 (Week 13); n= 85: number analyzed (Participants) | 85
  Percent monocytes; visit 2 (Week 13); n= 85 | 0.27 (2.720)
  Percent monocytes; visit 3 (Week 26); n= 71: number analyzed (Participants) | 71
  Percent monocytes; visit 3 (Week 26); n= 71 | 0.86 (3.274)
  Percent monocytes; visit 4 (Week 39); n= 65: number analyzed (Participants) | 65
  Percent monocytes; visit 4 (Week 39); n= 65 | 0.76 (3.286)
  Percent monocytes; visit 5 (Week 52); n= 60: number analyzed (Participants) | 60
  Percent monocytes; visit 5 (Week 52); n= 60 | -0.01 (3.058)
  Percent monocytes; visit 6 (Week 69); n= 58: number analyzed (Participants) | 58
  Percent monocytes; visit 6 (Week 69); n= 58 | 0.64 (2.834)
  Percent monocytes; visit 7 (Week 86); n= 53: number analyzed (Participants) | 53
  Percent monocytes; visit 7 (Week 86); n= 53 | 0.94 (3.148)
  Percent monocytes; visit 8 (Week 104); n= 36: number analyzed (Participants) | 36
  Percent monocytes; visit 8 (Week 104); n= 36 | 0.04 (3.458)
  Percent monocytes; visit 9 (Week 121); n= 35: number analyzed (Participants) | 35
  Percent monocytes; visit 9 (Week 121); n= 35 | -0.11 (2.895)
  Percent monocytes; visit 10 (Week 138); n= 33: number analyzed (Participants) | 33
  Percent monocytes; visit 10 (Week 138); n= 33 | 0.15 (3.160)
  Percent monocytes; visit 11 (Week 156); n= 29: number analyzed (Participants) | 29
  Percent monocytes; visit 11 (Week 156); n= 29 | -0.27 (3.007)
  Percent monocytes; visit 12 (Week 173); n= 24: number analyzed (Participants) | 24
  Percent monocytes; visit 12 (Week 173); n= 24 | -0.44 (2.687)
  Percent monocytes; visit 13 (Week 190); n= 17: number analyzed (Participants) | 17
  Percent monocytes; visit 13 (Week 190); n= 17 | -1.43 (2.909)
  Percent monocytes; visit 14 (Week 208); n= 10: number analyzed (Participants) | 10
  Percent monocytes; visit 14 (Week 208); n= 10 | -0.71 (5.153)
  Percent monocytes; visit 15 (Week 225); n= 4: number analyzed (Participants) | 4
  Percent monocytes; visit 15 (Week 225); n= 4 | 1.08 (1.090)
  Percent monocytes; visit 16 (Week 242); n= 4: number analyzed (Participants) | 4
  Percent monocytes; visit 16 (Week 242); n= 4 | 1.25 (1.686)
  Percent monocytes; visit 17 (Week 260); n= 4: number analyzed (Participants) | 4
  Percent monocytes; visit 17 (Week 260); n= 4 | 2.03 (2.219)
  Percent monocytes; visit 18 (Week 277); n= 2: number analyzed (Participants) | 2
  Percent monocytes; visit 18 (Week 277); n= 2 | 4.20 (2.687)
  Percent monocytes; withdrawal visit; n= 78: number analyzed (Participants) | 78
  Percent monocytes; withdrawal visit; n= 78 | 0.48 (3.355)
  Percent monocytes; follow up visit; n= 56: number analyzed (Participants) | 56
  Percent monocytes; follow up visit; n= 56 | -0.35 (3.293)
  Percent neutrophils; visit 1 (Screening); n= 84: number analyzed (Participants) | 84
  Percent neutrophils; visit 1 (Screening); n= 84 | 2.60 (11.021)
  Percent neutrophils; visit 2 (Week 13); n= 85: number analyzed (Participants) | 85
  Percent neutrophils; visit 2 (Week 13); n= 85 | 0.19 (11.584)
  Percent neutrophils; visit 3 (Week 26); n= 71: number analyzed (Participants) | 71
  Percent neutrophils; visit 3 (Week 26); n= 71 | 0.60 (12.994)
  Percent neutrophils; visit 4 (Week 39); n= 65: number analyzed (Participants) | 65
  Percent neutrophils; visit 4 (Week 39); n= 65 | -0.66 (11.810)
  Percent neutrophils; visit 5 (Week 52); n= 60: number analyzed (Participants) | 60
  Percent neutrophils; visit 5 (Week 52); n= 60 | 3.31 (14.222)
  Percent neutrophils; visit 6 (Week 69); n= 58: number analyzed (Participants) | 58
  Percent neutrophils; visit 6 (Week 69); n= 58 | 0.90 (10.552)
  Percent neutrophils; visit 7 (Week 86); n= 53: number analyzed (Participants) | 53
  Percent neutrophils; visit 7 (Week 86); n= 53 | -0.09 (14.427)
  Percent neutrophils; visit 8 (Week 104); n= 37: number analyzed (Participants) | 37
  Percent neutrophils; visit 8 (Week 104); n= 37 | -0.81 (11.595)
  Percent neutrophils; visit 9 (Week 121); n= 35: number analyzed (Participants) | 35
  Percent neutrophils; visit 9 (Week 121); n= 35 | 2.91 (14.604)
  Percent neutrophils; visit 10 (Week 138); n= 33: number analyzed (Participants) | 33
  Percent neutrophils; visit 10 (Week 138); n= 33 | 4.70 (12.464)
  Percent neutrophils; visit 11 (Week 156); n= 29: number analyzed (Participants) | 29
  Percent neutrophils; visit 11 (Week 156); n= 29 | 5.58 (10.691)
  Percent neutrophils; visit 12 (Week 173); n= 24: number analyzed (Participants) | 24
  Percent neutrophils; visit 12 (Week 173); n= 24 | 4.39 (13.509)
  Percent neutrophils; visit 13 (Week 190); n= 17: number analyzed (Participants) | 17
  Percent neutrophils; visit 13 (Week 190); n= 17 | 7.55 (16.056)
  Percent neutrophils; visit 14 (Week 208); n= 10: number analyzed (Participants) | 10
  Percent neutrophils; visit 14 (Week 208); n= 10 | 6.95 (7.643)
  Percent neutrophils; visit 15 (Week 225); n= 4: number analyzed (Participants) | 4
  Percent neutrophils; visit 15 (Week 225); n= 4 | 7.03 (5.900)
  Percent neutrophils; visit 16 (Week 242); n= 4: number analyzed (Participants) | 4
  Percent neutrophils; visit 16 (Week 242); n= 4 | 3.03 (10.460)
  Percent neutrophils; visit 17 (Week 260); n= 4: number analyzed (Participants) | 4
  Percent neutrophils; visit 17 (Week 260); n= 4 | 3.80 (3.990)
  Percent neutrophils; visit 18 (Week 277); n= 2: number analyzed (Participants) | 2
  Percent neutrophils; visit 18 (Week 277); n= 2 | 2.00 (7.354)
  Percent neutrophils; withdrawal visit; n= 78: number analyzed (Participants) | 78
  Percent neutrophils; withdrawal visit; n= 78 | 2.94 (13.146)
  Percent neutrophils; follow up visit; n= 56: number analyzed (Participants) | 56
  Percent neutrophils; follow up visit; n= 56 | 2.58 (14.680)
  RDW; visit 1 (Screening); n= 85: number analyzed (Participants) | 85
  RDW; visit 1 (Screening); n= 85 | 0.41 (1.398)
  RDW; visit 2 (Week 13); n= 89: number analyzed (Participants) | 89
  RDW; visit 2 (Week 13); n= 89 | -0.07 (1.532)
  RDW; visit 3 (Week 26); n= 74: number analyzed (Participants) | 74
  RDW; visit 3 (Week 26); n= 74 | 0.05 (0.924)
  RDW; visit 4 (Week 39); n= 69: number analyzed (Participants) | 69
  RDW; visit 4 (Week 39); n= 69 | 0.47 (1.637)
  RDW; visit 5 (Week 52); n= 64: number analyzed (Participants) | 64
  RDW; visit 5 (Week 52); n= 64 | 0.35 (1.598)
  RDW; visit 6 (Week 69); n= 62: number analyzed (Participants) | 62
  RDW; visit 6 (Week 69); n= 62 | 0.05 (1.437)
  RDW; visit 7 (Week 86); n= 55: number analyzed (Participants) | 55
  RDW; visit 7 (Week 86); n= 55 | 0.05 (1.109)
  RDW; visit 8 (Week 104); n= 41: number analyzed (Participants) | 41
  RDW; visit 8 (Week 104); n= 41 | 0.32 (1.386)
  RDW; visit 9 (Week 121); n= 36: number analyzed (Participants) | 36
  RDW; visit 9 (Week 121); n= 36 | -0.19 (1.084)
  RDW; visit 10 (Week 138); n= 36: number analyzed (Participants) | 36
  RDW; visit 10 (Week 138); n= 36 | 0.22 (0.885)
  RDW; visit 11 (Week 156); n= 31: number analyzed (Participants) | 31
  RDW; visit 11 (Week 156); n= 31 | 0.94 (1.760)
  RDW; visit 12 (Week 173); n= 24: number analyzed (Participants) | 24
  RDW; visit 12 (Week 173); n= 24 | 0.41 (1.292)
  RDW; visit 13 (Week 190); n= 18: number analyzed (Participants) | 18
  RDW; visit 13 (Week 190); n= 18 | 0.88 (0.919)
  RDW; visit 14 (Week 208); n= 10: number analyzed (Participants) | 10
  RDW; visit 14 (Week 208); n= 10 | 1.98 (1.605)
  RDW; visit 15 (Week 225); n= 4: number analyzed (Participants) | 4
  RDW; visit 15 (Week 225); n= 4 | 0.28 (0.550)
  RDW; visit 16 (Week 242); n= 4: number analyzed (Participants) | 4
  RDW; visit 16 (Week 242); n= 4 | 3.95 (6.855)
  RDW; visit 17 (Week 260); n= 4: number analyzed (Participants) | 4
  RDW; visit 17 (Week 260); n= 4 | 2.50 (2.202)
  RDW; visit 18 (Week 277); n= 2: number analyzed (Participants) | 2
  RDW; visit 18 (Week 277); n= 2 | 2.05 (0.495)
  RDW; withdrawal visit; n= 79: number analyzed (Participants) | 79
  RDW; withdrawal visit; n= 79 | 0.10 (1.097)
  RDW; follow up visit; n= 59: number analyzed (Participants) | 59
  RDW; follow up visit; n= 59 | 0.27 (1.235)

27. Primary Outcome: Change From Baseline in Urine Albumin Creatinine Ratio
Description: Urine samples were collected from participants for evaluation of change from Baseline in urinalysis parameters including albumin creatinine ratio. Baseline was defined by and taken directly from the Baseline assessments in the parent study NCT01336621. Change from Baseline was defined as post-Baseline value minus Baseline value. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Time Frame: Baseline and up to 5.8 years
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Mg of urine albumin/ mmol of creatinine
Arm/Group | Retigabine IR
Number analyzed (Participants) | 98
Mg of urine albumin/ mmol of creatinine
  Visit 1 (Screening); n= 39: number analyzed (Participants) | 39
  Visit 1 (Screening); n= 39 | -0.57 (3.573)
  Visit 2 (Week 13); n= 72: number analyzed (Participants) | 72
  Visit 2 (Week 13); n= 72 | -0.07 (3.172)
  Visit 3 (Week 26); n= 54: number analyzed (Participants) | 54
  Visit 3 (Week 26); n= 54 | 0.15 (3.678)
  Visit 4 (Week 39); n= 53: number analyzed (Participants) | 53
  Visit 4 (Week 39); n= 53 | -0.64 (3.241)
  Visit 5 (Week 52); n= 52: number analyzed (Participants) | 52
  Visit 5 (Week 52); n= 52 | -0.69 (3.065)
  Visit 6 (Week 69); n= 46: number analyzed (Participants) | 46
  Visit 6 (Week 69); n= 46 | -0.53 (3.489)
  Visit 7 (Week 86); n= 47: number analyzed (Participants) | 47
  Visit 7 (Week 86); n= 47 | 0.07 (6.062)
  Visit 8 (Week 104); n= 32: number analyzed (Participants) | 32
  Visit 8 (Week 104); n= 32 | -0.75 (4.508)
  Visit 9 (Week 121); n= 30: number analyzed (Participants) | 30
  Visit 9 (Week 121); n= 30 | -0.89 (5.421)
  Visit 10 (Week 138); n= 26: number analyzed (Participants) | 26
  Visit 10 (Week 138); n= 26 | -1.05 (4.236)
  Visit 11 (Week 156); n= 22: number analyzed (Participants) | 22
  Visit 11 (Week 156); n= 22 | -0.65 (2.494)
  Visit 12 (Week 173); n= 19: number analyzed (Participants) | 19
  Visit 12 (Week 173); n= 19 | -1.81 (5.060)
  Visit 13 (Week 190); n= 10: number analyzed (Participants) | 10
  Visit 13 (Week 190); n= 10 | -0.59 (1.748)
  Visit 14 (Week 208); n= 8: number analyzed (Participants) | 8
  Visit 14 (Week 208); n= 8 | -1.70 (4.032)
  Visit 15 (Week 225); n= 4: number analyzed (Participants) | 4
  Visit 15 (Week 225); n= 4 | 0.13 (0.981)
  Visit 16 (Week 242); n= 3: number analyzed (Participants) | 3
  Visit 16 (Week 242); n= 3 | -0.33 (0.153)
  Visit 17 (Week 260); n= 3: number analyzed (Participants) | 3
  Visit 17 (Week 260); n= 3 | -0.33 (0.321)
  Visit 18 (Week 277); n= 2: number analyzed (Participants) | 2
  Visit 18 (Week 277); n= 2 | -0.50 (0.990)
  Withdrawal visit; n= 63: number analyzed (Participants) | 63
  Withdrawal visit; n= 63 | -0.35 (3.874)
  Follow up visit; n= 48: number analyzed (Participants) | 48
  Follow up visit; n= 48 | -0.62 (3.515)

28. Primary Outcome: Change From Baseline in Urine Albumin Levels
Description: Urine samples were collected from participants for evaluation of change from Baseline in urinalysis parameters including albumin levels. Baseline was defined by and taken directly from the Baseline assessments in the parent study NCT01336621. Change from Baseline was defined as post-Baseline value minus Baseline value. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Time Frame: Baseline and up to 5.8 years
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Milligrams per liter (mg/L)
Arm/Group | Retigabine IR
Number analyzed (Participants) | 98
Milligrams per liter (mg/L)
  Visit 1 (Screening); n= 39: number analyzed (Participants) | 39
  Visit 1 (Screening); n= 39 | -5.2 (57.64)
  Visit 2 (Week 13); n= 72: number analyzed (Participants) | 72
  Visit 2 (Week 13); n= 72 | -1.8 (48.39)
  Visit 3 (Week 26); n= 54: number analyzed (Participants) | 54
  Visit 3 (Week 26); n= 54 | -17.1 (92.34)
  Visit 4 (Week 39); n= 53: number analyzed (Participants) | 53
  Visit 4 (Week 39); n= 53 | -21.0 (94.25)
  Visit 5 (Week 52); n= 52: number analyzed (Participants) | 52
  Visit 5 (Week 52); n= 52 | -21.6 (94.87)
  Visit 6 (Week 69); n= 46: number analyzed (Participants) | 46
  Visit 6 (Week 69); n= 46 | -15.7 (56.98)
  Visit 7 (Week 86); n= 47: number analyzed (Participants) | 47
  Visit 7 (Week 86); n= 47 | 7.7 (131.03)
  Visit 8 (Week 104); n= 32: number analyzed (Participants) | 32
  Visit 8 (Week 104); n= 32 | -8.1 (59.50)
  Visit 9 (Week 121); n= 30: number analyzed (Participants) | 30
  Visit 9 (Week 121); n= 30 | -14.7 (61.73)
  Visit 10 (Week 138); n= 26: number analyzed (Participants) | 26
  Visit 10 (Week 138); n= 26 | -16.0 (66.79)
  Visit 11 (Week 156); n= 22: number analyzed (Participants) | 22
  Visit 11 (Week 156); n= 22 | -7.4 (35.40)
  Visit 12 (Week 173); n= 19: number analyzed (Participants) | 19
  Visit 12 (Week 173); n= 19 | -27.2 (80.24)
  Visit 13 (Week 190); n= 10: number analyzed (Participants) | 10
  Visit 13 (Week 190); n= 10 | -2.8 (27.95)
  Visit 14 (Week 208); n= 8: number analyzed (Participants) | 8
  Visit 14 (Week 208); n= 8 | -15.9 (45.76)
  Visit 15 (Week 225); n= 4: number analyzed (Participants) | 4
  Visit 15 (Week 225); n= 4 | -1.8 (11.53)
  Visit 16 (Week 242); n= 3: number analyzed (Participants) | 3
  Visit 16 (Week 242); n= 3 | -8.7 (9.61)
  Visit 17 (Week 260); n= 3: number analyzed (Participants) | 3
  Visit 17 (Week 260); n= 3 | -3.3 (12.86)
  Visit 18 (Week 277); n= 2: number analyzed (Participants) | 2
  Visit 18 (Week 277); n= 2 | -7.5 (0.71)
  Withdrawal visit; n= 63: number analyzed (Participants) | 63
  Withdrawal visit; n= 63 | -6.5 (51.69)
  Follow up visit; n= 48: number analyzed (Participants) | 48
  Follow up visit; n= 48 | -19.9 (99.24)

29. Primary Outcome: Change From Baseline in Urine Creatinine Levels
Description: Urine samples were collected from participants for evaluation of change from Baseline in urinalysis parameters including creatinine levels. Baseline was defined by and taken directly from the Baseline assessments in the parent study NCT01336621. Change from Baseline was defined as post-Baseline value minus Baseline value. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Time Frame: Baseline and up to 5.8 years
Population: Safety Population
Measure: Mean (Standard Deviation); unit: µmol/L
Arm/Group | Retigabine IR
Number analyzed (Participants) | 98
µmol/L
  Visit 1 (Screening); n= 52: number analyzed (Participants) | 52
  Visit 1 (Screening); n= 52 | -2019.6 (10153.70)
  Visit 2 (Week 13); n= 89: number analyzed (Participants) | 89
  Visit 2 (Week 13); n= 89 | -1846.2 (8206.65)
  Visit 3 (Week 26); n= 75: number analyzed (Participants) | 75
  Visit 3 (Week 26); n= 75 | -3023.7 (9197.50)
  Visit 4 (Week 39); n= 66: number analyzed (Participants) | 66
  Visit 4 (Week 39); n= 66 | -2849.6 (7810.79)
  Visit 5 (Week 52); n= 63: number analyzed (Participants) | 63
  Visit 5 (Week 52); n= 63 | -1626.5 (10205.13)
  Visit 6 (Week 69); n= 59: number analyzed (Participants) | 59
  Visit 6 (Week 69); n= 59 | -3534.2 (8657.09)
  Visit 7 (Week 86); n= 55: number analyzed (Participants) | 55
  Visit 7 (Week 86); n= 55 | -2664.4 (7900.30)
  Visit 8 (Week 104); n= 42: number analyzed (Participants) | 42
  Visit 8 (Week 104); n= 42 | -2645.1 (8368.43)
  Visit 9 (Week 121); n= 37: number analyzed (Participants) | 37
  Visit 9 (Week 121); n= 37 | -1727.3 (10330.75)
  Visit 10 (Week 138); n= 35: number analyzed (Participants) | 35
  Visit 10 (Week 138); n= 35 | -1712.6 (11352.03)
  Visit 11 (Week 156); n= 30: number analyzed (Participants) | 30
  Visit 11 (Week 156); n= 30 | -1400.0 (13151.92)
  Visit 12 (Week 173); n= 23: number analyzed (Participants) | 23
  Visit 12 (Week 173); n= 23 | -1008.3 (9395.56)
  Visit 13 (Week 190); n= 19: number analyzed (Participants) | 19
  Visit 13 (Week 190); n= 19 | -3604.1 (10215.20)
  Visit 14 (Week 208); n= 10: number analyzed (Participants) | 10
  Visit 14 (Week 208); n= 10 | 3238.3 (12290.24)
  Visit 15 (Week 225); n= 5: number analyzed (Participants) | 5
  Visit 15 (Week 225); n= 5 | -675.0 (16785.90)
  Visit 16 (Week 242); n= 4: number analyzed (Participants) | 4
  Visit 16 (Week 242); n= 4 | -5426.3 (13280.49)
  Visit 17 (Week 260); n= 4: number analyzed (Participants) | 4
  Visit 17 (Week 260); n= 4 | 148.8 (15164.36)
  Visit 18 (Week 277); n= 2: number analyzed (Participants) | 2
  Visit 18 (Week 277); n= 2 | -7337.5 (10850.55)
  Withdrawal visit; n= 80: number analyzed (Participants) | 80
  Withdrawal visit; n= 80 | -3570.3 (8244.65)
  Follow up visit; n= 60: number analyzed (Participants) | 60
  Follow up visit; n= 60 | -515.8 (9359.74)

30. Primary Outcome: Changes From Baseline in American Urological Association Symptom Scale (AUA SS) Score
Description: The effect of retigabine on bladder function was assessed using AUA symptom index. It is a 7-item Likert-scored scale ranging from 0 (no symptom at all) to 5 (almost always symptoms present) with a total possible score of 35. AUA SS score is the sum of the responses to these seven questions. The total score for all questions was classified as mild (0 to 7), moderate (8 to 19), or severe (>19). Baseline was defined by and taken directly from the Baseline assessments in the parent study NCT01336621. Change from Baseline was defined as post-Baseline value minus Baseline value. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Time Frame: Baseline and up to 5.8 years
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Score on AUA SS scale
Arm/Group | Retigabine IR
Number analyzed (Participants) | 98
Score on AUA SS scale
  Visit 3 (Week 26); n= 82: number analyzed (Participants) | 82
  Visit 3 (Week 26); n= 82 | -0.7 (3.50)
  Visit 5 (Week 52); n= 68: number analyzed (Participants) | 68
  Visit 5 (Week 52); n= 68 | -0.9 (4.67)
  Visit 8 (Week 104); n= 42: number analyzed (Participants) | 42
  Visit 8 (Week 104); n= 42 | -1.0 (3.79)
  Visit 11 (Week 156); n= 31: number analyzed (Participants) | 31
  Visit 11 (Week 156); n= 31 | -1.0 (4.18)
  Visit 14 (Week 208); n= 10: number analyzed (Participants) | 10
  Visit 14 (Week 208); n= 10 | -2.3 (5.54)
  Visit 17 (Week 260); n= 4: number analyzed (Participants) | 4
  Visit 17 (Week 260); n= 4 | -6.5 (7.72)
  Withdrawal visit; n= 85: number analyzed (Participants) | 85
  Withdrawal visit; n= 85 | -1.0 (3.99)

31. Primary Outcome: Change From Baseline in Post-Void Residual (PVR) Bladder Ultrasound Urine Volume
Description: The PVR bladder ultrasound was used to assess urinary retention. Baseline was defined by and taken directly from the Baseline assessments in the parent study NCT01336621. Change from Baseline was defined as post-Baseline value minus Baseline value. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Time Frame: Baseline and up to 5.8 years
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Milliliter (mL)
Arm/Group | Retigabine IR
Number analyzed (Participants) | 98
Milliliter (mL)
  Visit 3 (Week 26); n= 77: number analyzed (Participants) | 77
  Visit 3 (Week 26); n= 77 | -6.0 (24.73)
  Visit 5 (Week 52); n= 64: number analyzed (Participants) | 64
  Visit 5 (Week 52); n= 64 | 2.7 (49.20)
  Visit 8 (Week 104); n= 40: number analyzed (Participants) | 40
  Visit 8 (Week 104); n= 40 | 3.9 (49.03)
  Visit 11 (Week 156); n= 25: number analyzed (Participants) | 25
  Visit 11 (Week 156); n= 25 | 2.0 (18.40)
  Visit 14 (Week 208); n= 10: number analyzed (Participants) | 10
  Visit 14 (Week 208); n= 10 | -16.0 (21.33)
  Visit 17 (Week 260); n= 4: number analyzed (Participants) | 4
  Visit 17 (Week 260); n= 4 | -23.3 (25.00)
  Withdrawal visit; n= 67: number analyzed (Participants) | 67
  Withdrawal visit; n= 67 | -7.6 (30.39)

32. Primary Outcome: Number of Participants With Suicidal Ideation or Behavior Assessed by the Columbia Suicide Severity Rating Scale (C-SSRS) Score
Description: Number of participants with suicidal ideation or behavior during treatment were assessed using the C-SSRS score scale. It is a brief questionnaire designed to assess severity and change in suicidality by integrating both behavior and ideation using a semi-structured interview to probe participant responses. Participants are classified with respect to extent of suicidal ideation, extent of suicidal behavior, and with respect to self-injurious behavior.
Time Frame: Up to 5.8 years
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | Retigabine IR
Number analyzed (Participants) | 95
Participants
  Suicidal ideation | 1
  Suicidal behavior | 0
  Self-injurious behavior, no suicidal attempt | 0

33. Primary Outcome: Number of Participants Experiencing New Seizure Types
Description: Number of participants experiencing new seizure type that is seizure not experienced before were summarized. New seizure types were classified into 5 classes including type A (simple partial seizure), type B (complex partial seizure), type C (Partials, evolving to Secondary Generalized Seizures), type D (Generalized, excluding Myoclonic Seizures), type D2 (Myoclonic Seizures) and type E (Unclassified Seizures).
Time Frame: Up to 5.8 years
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | Retigabine IR
Number analyzed (Participants) | 98
Participants
  Type A; Simple Partial Seizures | 5
  Type B; Complex Partial Seizures | 2
  Type C; Partials, evolving to Sec. Gen. Seizures | 0
  Type D; Generalized, excl. Myoclonic Seizures | 0
  Type D2; Myoclonic Seizures | 0
  Type E; Unclassified seizures | 0

34. Primary Outcome: Number of Participants Experiencing Worsening of Seizures
Description: Worsening of seizures was defined as an increase in seizure frequency or the occurrence of a new, more severe seizure type, or status epilepticus occurring in a participant without a history of status epilepticus. An increase in seizure frequency was defined as doubling of the 28-day seizure frequency compared to the 28-day Baseline seizure frequency established in the parent study. Number of participants experiencing worsening of seizure during study period are presented.
Time Frame: Up to 5.8 years
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | Retigabine IR
Number analyzed (Participants) | 98
Participants | 1

35. Primary Outcome: Duration of Retigabine Exposure
Description: Duration of exposure was calculated from the first dose through the last dose during study including the Taper Phase and presented using median and full range.
Time Frame: Up to 5.8 years
Population: Safety Population
Measure: Median (Full Range); unit: Weeks
Arm/Group | Retigabine IR
Number analyzed (Participants) | 98
Weeks | 103.7 [0.5 to 284]

36. Primary Outcome: Number of Participants With Resolution of Abnormal Eye Pigmentation After Discontinuation of Retigabine
Description: The ophthalmologist/retina specialist determined the presence or absence of retinal and non-retinal ocular abnormalities. Retinal abnormalities included abnormalities in the macula and/or the peripheral retina and non-retinal ocular pigmentary abnormality.
Time Frame: Up to 2.6 years
Population: All SFUCP Subjects
Measure: Number; unit: Participants
Groups:
- Retigabine IR in SFUCP: Participants who withdrew from the Open-Label Treatment Phase and who had retinal pigmentation or unexplained vision loss, pigmentation of non-retinal ocular tissue or abnormal discoloration of nails, lips, skin or mucosa were followed-up in SFUCP following discontinuation of their retigabine, which is the final reporting phase of the study. During SFUCP, participants underwent six monthly comprehensive eye examinations and/or dermatological assessments. Participants were followed-up until the discoloration /pigmentation either resolves or stabilizes, as defined by no change over two consecutive six monthly assessments over at least 12 months after discontinuation of RTG IR.
Arm/Group | Retigabine IR in SFUCP
Number analyzed (Participants) | 9
Participants
  Retinal pigmentary abnormality | 1
  Non-retinal ocular pigmentary abnormality | 1

37. Primary Outcome: Number of Participants With Resolution of Dermatologist Confirmed Abnormal Discoloration After Discontinuation of Retigabine
Description: Participants who enter the SFUCP who had an on-treatment finding(s) of abnormal discoloration of skin, lips, nails or mucosa confirmed by a dermatologist entered the SFUCP and underwent assessments performed by a dermatologist at 6-monthly intervals. The assessment of the participant's skin included assessment of the skin around the eyes and the eyelids, lips, nails, and mucosa.
Time Frame: Up to 2.6 years
Population: All SFUCP Subjects
Measure: Number; unit: Participants
Arm/Group | Retigabine IR in SFUCP
Number analyzed (Participants) | 9
Participants | 2

38. Primary Outcome: Time From Discontinuation of Retigabine to Resolution of Abnormal Eye Pigmentation
Description: Retinal pigmentary abnormality was determined by either an ophthalmologist or retina specialist. Retinal pigmentary abnormality included abnormality of macula, peripheral retina and unspecified location. If a participant had pigmentary abnormality of macula and pigmentary abnormality of the peripheral retina both should be resolved in order for retinal pigmentary abnormality to be considered resolved. If a participant had non-retinal ocular pigmentary abnormality in more than one location (conjunctiva, sclera, cornea, iris or lens), all should be resolved for non-retinal pigmentary abnormality to be considered resolved.
Time Frame: Up to 2.6 years
Population: All SFUCP Subjects
Measure: Median (Full Range); unit: Days
Arm/Group | Retigabine IR in SFUCP
Number analyzed (Participants) | 1
Days
  Retinal Pigmentary Abnormality | 157.0 [157 to 157]
  Non-Retinal Ocular Pigmentary Abnormality | 119.0 [119 to 119]

39. Primary Outcome: Time From Discontinuation of Retigabine to Resolution of All Dermatologist-confirmed Abnormal Discoloration
Description: Assessments were at approximately 6-monthly intervals (timed relative to the participants previous dermatology assessment) until the abnormal discoloration either resolved or stabilized (as defined by no changes over 2 consecutive 6-monthly assessments performed by the dermatologist over at least 12 months after discontinuation of retigabine). The assessment of the participant's skin included assessment of the skin around the eyes and the eyelids, lips, nails, and mucosa. Only participants with resolution of the specified tissue are included in this analysis.
Time Frame: Up to 2.6 years
Population: All SFUCP Subjects
Measure: Median (Full Range); unit: Days
Arm/Group | Retigabine IR in SFUCP
Number analyzed (Participants) | 9
Days
  All; n= 2: number analyzed (Participants) | 2
  All; n= 2 | 582.0 [253 to 911]
  Skin; n= 1: number analyzed (Participants) | 1
  Skin; n= 1 | 192.0 [192 to 192]
  Lips; n= 0: number analyzed (Participants) | 0
  Nails; n= 1: number analyzed (Participants) | 1
  Nails; n= 1 | 253.0 [253 to 253]
  Mucosa; n= 3: number analyzed (Participants) | 3
  Mucosa; n= 3 | 701.0 [192 to 911]

40. Secondary Outcome: Number of Participants Experiencing a 0 to <25, 25 to <50, 50 to <75 and 75 to 100 Percent Reduction in 28 Day POS Frequency From Baseline
Description: The seizure frequency was recorded in daily seizure calendar by participants during the treatment period. Baseline assessments in this OLE study are defined by and taken directly from the Baseline assessments in the parent study NCT01336621.
Time Frame: Baseline and up to 5.8 years
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | Retigabine IR
Number analyzed (Participants) | 98
Participants
  0 to <25 percent reduction | 7
  25 to <50 percent reduction | 13
  50 to <75 percent reduction | 26
  75 to 100 percent reduction | 42

41. Secondary Outcome: Percent Change From Baseline in 28-day Partial-onset Seizure Frequency
Description: The seizure frequency was recorded in daily seizure calendar by participants during the treatment period. Percent change from Baseline in 28-day partial onset seizure frequency was presented as mean and standard deviation (SD). Baseline assessments in this OLE study are defined by and taken directly from the Baseline assessments in the parent study NCT01336621. Percent change from Baseline was calculated as post-Baseline value minus Baseline value divided by Baseline value into 100.
Time Frame: Baseline and up to 5.8 years
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Retigabine IR
Number analyzed (Participants) | 98
Percent change | -56.9 (52.46)

42. Secondary Outcome: Number of Participants Experiencing an Increase in 28-day Partial-onset Seizure Frequency From Baseline
Description: as for outcome 40
Time Frame: Baseline and up to 5.8 years
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | Retigabine IR
Number analyzed (Participants) | 98
Participants | 10

43. Secondary Outcome: Number of Participants Who Remained Seizure-free
Description: The seizure frequency was recorded in daily seizure calendar by participants during the treatment period. Number of participants who were treated retigabine for at least 6 months and who remained seizure free for any 6 continuous months as well as number of participants who were treated with retigabine for at least 12 months and who remained seizure free for any 12 continuous months are presented.
Time Frame: Up to 5.8 years
Population: Safety population
Measure: Number; unit: Participants
Arm/Group | Retigabine IR
Number analyzed (Participants) | 98
Participants
  Seizure free for 6 months; n= 85: number analyzed (Participants) | 85
  Seizure free for 6 months; n= 85 | 27
  Seizure free for 12 months; n= 71: number analyzed (Participants) | 71
  Seizure free for 12 months; n= 71 | 13

ADVERSE EVENTS:
Time Frame: Treatment emergent Serious adverse events (TESAEs) and non-serious adverse events (TEAEs) were collected from the start of the study treatment until the end-of study treatment (Up to 5.8 years).
Description: AEs and SAEs were collected in 'Safety Population' for retigabine IR arm and in 'All SFUCP subjects Population' for Retigabine IR in SFUCP arm. The MedDRA version for the Primary Reporting Phase is 19.1. However the SFUCP phase uses version 20.1.
Groups:
- Retigabine IR in SFUCP: Participants who withdrew from the Open-Label Treatment Phase and who had retinal pigmentation or unexplained vision loss, pigmentation of non-retinal ocular tissue or abnormal discoloration of nails, lips, skin or mucosa were followed-up in SFUCP following discontinuation of their retigabine, which was the final reporting phase of the study. During SFUCP, participants underwent six monthly comprehensive eye examinations and/or dermatological assessments. Participants were followed-up until the discoloration /pigmentation either resolves or stabilizes, as defined by no change over two consecutive six monthly assessments over at least 12 months after discontinuation of RTG IR .
Arm/Group | Retigabine IR | Retigabine IR in SFUCP
All-Cause Mortality (participants affected / at risk) | 0/98 | 0/9
Serious Adverse Events (participants affected / at risk) | 4/98 | 1/9
Other Adverse Events (participants affected / at risk) | 38/98 | 3/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Retigabine IR (N=98) | Retigabine IR in SFUCP (N=9)
Cerebrovascular disorder (Nervous system disorders) | 1 (2) | 0
Generalised tonic-clonic seizure (Nervous system disorders) | 1 (1) | 0
Seizure (Nervous system disorders) | 1 (1) | 0
Agitation (Psychiatric disorders) | 1 (1) | 0
Epileptic psychosis (Psychiatric disorders) | 1 (1) | 0
Scar (Injury, poisoning and procedural complications) | 1 (1) | 0
Hemoglobin decreased (Investigations) | 1 (1) | 0
Malignant melanoma stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Retigabine IR (N=98) | Retigabine IR in SFUCP (N=9)
Dizziness (Nervous system disorders) | 14 (18) | 0
Headache (Nervous system disorders) | 10 (23) | 0
Asthenia (General disorders) | 11 (20) | 0
Weight increased (Investigations) | 7 (7) | 0
Bacteriuria (Infections and infestations) | 6 (7) | 0
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 0
Nail pigmentation (Skin and subcutaneous tissue disorders) | 6 (6) | 0
Breast fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Iridocyclitis (Eye disorders) | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 1
Oral mucosal discolouration (Gastrointestinal disorders) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Amenorrhoea (Reproductive system and breast disorders) | 0 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
17 parts. withdrew due to AE, however only 16 had a TEAE leading to withdrawal of RTG. 1 part. with a TEAE of seizure, withdrew due to lack of efficacy. 2 further parts. withdrew due to AE but had no TEAEs which led to withdrawal of RTG.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.